#### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | : | Reporting and Analysis Plan for 206898: An Open Label,<br>Phase 1 Study to Evaluate the PK, Safety, Tolerability and<br>Acceptability of Long Acting Injections of the HIV Integrase<br>Inhibitor, Cabotegravir (CAB; GSK1265744) in HIV<br>Uninfected Chinese Men |
|---|---|---|
| <b>Compound Number</b> | : | GSK1265744 |
| <b>Effective Date</b> | : | 22-APR-2019 |

#### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 206898.
- This RAP is intended to describe the safety, tolerability, and pharmacokinetic (PK) analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

#### **Author's Name and Functional Area:**

| PPD | | 22-APR-2019 |
|----------------|-------------|-------------|
| Senior Biostat | 22-AFR-2019 | |
| PPD | | |
| Pharmacokine | 22-APR-2019 | |
| | , , | |

#### Approved by:

| PPD | | 22-APR-2019 |
|---------------|--------------|-------------|
| Statistics Le | 22-AFK-2019 | |
| PPD | | 22-APR-2019 |
| Manager Sta | 22-A1 K-2019 | |

Copyright 2019 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

## **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| 1. | REPO | RTING 8 | ANALYSIS PLAN SYNOPSIS | 5 |
| 2. | SUMM | IARY OF | KEY PROTOCOL INFORMATION | 8 |
| ۷. | 2.1. | | es to the Protocol Defined Statistical Analysis Plan | |
| | 2.2. | | Objective(s) and Endpoint(s) | |
| | 2.2. | | Design | |
| | 2.3.<br>2.4. | • | cal Hypotheses | |
| | ۷.4. | Statistic | ai i iypotileses | 10 |
| 3. | PLANI | NED ANA | ALYSES | 11 |
| | 3.1. | Interim . | Analyses | 11 |
| | 3.2. | Final Ar | nalyses | 11 |
| 4 | ΔΝΔΙΥ | YSIS PO | PULATIONS | 12 |
| →. | 4.1. | | l Deviations | |
| | 4.1. | FIOLOGO | Deviations | 13 |
| 5. | | | IONS FOR DATA ANALYSES AND DATA HANDLING | |
| | CONV | 'ENTION | S | 14 |
| 6. | STUD | Y POPUI | LATION ANALYSES | 15 |
| Ο. | 6.1. | | w of Planned Analyses | |
| | 0.1. | 6.1.1. | Disposition | |
| | | 6.1.2. | Demographics | |
| | | 6.1.3. | Medical History | |
| | | 6.1.4. | Prior and Concomitant Medications | |
| | | 6.1.5. | Protocol Deviation | |
| 7. | PRIMA | ARY STA | TISTICAL ANALYSES | 17 |
| | 7.1. | Safety A | Analyses of CAB LA | 17 |
| | | 7.1.1. | Injection Site Reaction | 17 |
| | | 7.1.2. | Adverse Events | |
| | | 7.1.3. | Clinical Laboratory Tests | 19 |
| | | 7.1.4. | Vital Sign Assessments | 19 |
| | | 7.1.5. | Death | 20 |
| | 7.2. | Tolerab | ility Analyses of CAB LA | 21 |
| | 7.3. | | Pharmacokinetic Analyses | |
| | | 7.3.1. | Overview of Planned Primary Pharmacokinetic Analyses | 22 |
| | | 7.3.2. | Primary Drug Concentration Measures | 22 |
| | | 7.3.3. | Primary Pharmacokinetic Parameters | |
| | | | 7.3.3.1. Deriving Primary Pharmacokinetic Parameters | |
| | | | 7.3.3.2. Statistical Analysis of Primary Pharmacokinetic | |
| | | | Parameters | 24 |
| 8. | SECO | NDARY | STATISTICAL ANALYSES | 25 |
| | 8.1. | | ary Pharmacokinetic Analyses | |
| | - | 8.1.1. | Overview of Planned Secondary Pharmacokinetic | _3 |
| | | | Analyses | 25 |
| | | 8.1.2. | Secondary Drug Concentration Measures | |
| | | 8.1.3. | Secondary Pharmacokinetic Parameters | |

| | | | 8.1.3.1. | Deriving Secondary Pharmacokinetic Parameters | 25 |
|---|---|---|---|---|---|
| | 8.2. | Safaty ar | nd Tolorabi | lity Analyses of Oral CAB | |
| | 8.3. | Accentat | ility of CAF | B LA | 20<br>27 |
| | 8.4. | | | t Relationships for Safety and Tolerability | 21 |
| | 0. 1. | Paramete | ers | | 28 |
| | 8.5. | | | lyses | |
| | | 8.5.1. | | Exposure to CAB | |
| | | 8.5.2. | Possible s | uicidality-related Adverse Events | 29 |
| | | 8.5.3. | | ms | |
| | | 8.5.4. | | | |
| | | 8.5.5. | | cular Events | |
| | | 8.5.6. | Liver Ever | nts | 30 |
| 9. | REFE | RENCES. | | | 32 |
| 10. | APPE | NDICES | | | 33 |
| | 10.1. | | | ol Deviation Management and Definitions for Per | |
| | | 10.1.1. | Exclusions | s from Per Protocol Population | 34 |
| | 10.2. | | | Events | |
| | | | | Pefined Time & Events | |
| | 10.3. | | | ment Windows | |
| | 40.4 | | | ent Windows | |
| | 10.4. | | • | Phase and State | |
| | | 10.4.1. | | PhasesStates | |
| | | 10.4.2. | | Treatment States for AE Data | |
| | 10.5. | Annendiy | | isplay Standards & Handling Conventions | |
| | 10.0. | 10.5.1. | | atment & Sub-group Display Descriptors | |
| | | 10.5.2. | | Definition & Derivations | |
| | | | 10.5.2.1. | | |
| | | | 10.5.2.2. | | |
| | | | | Data | 41 |
| | | | | Process & Standards | |
| | 10.6. | | | d and Transformed Data | |
| | | 10.6.1. | | | |
| | | 10.6.2. | | ulation | |
| | 10.7 | 10.6.3. | | ura Withdrawala & Handling of Missing Data | |
| | 10.7. | 10.7.1. | | ure Withdrawals & Handling of Missing Data | |
| | | 10.7.1. | | of Missing Data | |
| | | 10.7.2. | 10.7.2.1. | | |
| | | | 10.7.2.1. | 3 | |
| | | | 10.7.2.3. | Handling of Missing Data for Statistical | |
| | 10.8. | Annandi | , Q. \/aluaa | Analysisof Potential Clinical Importance | |
| | 10.6. | 10.8.1. | | / Values | |
| | | 10.8.1. | | y values | |
| | | 10.8.3. | | S | |
| | 10.9 | | • | nter Studies | |

| | 10.9.1. Methods for | or Handling Centres | 50 |
|---|---|---|---|
| 10.10. | Appendix 10: Exami | nation of Covariates, Subgroups & Other Strata | 51 |
| | 10.10.1. Handling o | of Covariates, Subgroups & Other Strata | 51 |
| 10.11. | Appendix 11: Multipl | e Comparisons & Multiplicity | 52 |
| | 10.11.1. Handling o | f Multiple Comparisons & Multiplicity | 52 |
| 10.12. | Appendix 12: Model | Checking and Diagnostics for Statistical | |
| | Analyses | | <u>53</u> |
| | 10.12.1. Statistical | Analysis Assumptions | <u>53</u> |
| 10.13. | Appendix 13: Abbrev | viations & Trade Marks | 54 |
| | 10.13.1. Abbreviation | ons | 54 |
| | 10.13.2. Trademark | 'S | 55 |
| 10.14. | Appendix 14: List of | Data Displays | 56 |
| | 10.14.1. Data Displa | ay Numbering | 56 |
| | 10.14.2. Mock Exar | nple Shell Referencing | 56 |
| | 10.14.3. Deliverable | e [Priority] | 56 |
| | 10.14.4. Study Pop | ulation Tables | 57 |
| | 10.14.5. Safety Tab | les | 58 |
| | 10.14.6. Tolerability | <sup>,</sup> Tables | 61 |
| | 10.14.7. Acceptabil | ity Tables | 61 |
| | | kinetic Tables | |
| | 10.14.9. Pharmacol | kinetic Figures | 64 |
| | | js | |
| | 10.14.11. Non-ICH L | istings | 70 |
| 10.15. | Appendix 15: Examp | ole Mock Shells for Data Displays | 71 |
| 10.16. | Appendix 16: Advers | se Events of Special Interest Used for Data | |
| | Summaries | | 72 |

## 1. REPORTING & ANALYSIS PLAN SYNOPSIS

| Overview | Key Elements of the RAP |
|---|---|
| Purpose | <ul> <li>The purpose of this reporting and analysis plan (RAP) is to describe any<br/>planned analyses and output to be included in the clinical study report for<br/>Protocol 206898.</li> </ul> |
| Protocol | This RAP is based on the Protocol Amendment 1 (Dated: 06JUN2018) of study Protocol 206898 (GSK Document No.: 2016N293702_01] and eCRF Version (2.00, Dated: 26SEP2018). |
| Primary<br>Objective | Evaluate the safety and tolerability of the injectable agent, cabotegravir (GSK1265744) long acting (CAB LA) injectable (600 mg dose administered every 4 weeks for 2 doses followed by every 8 weeks for 3 doses) through Week 5-41 in HIV-1 uninfected Chinese men. |
| | <ul> <li>Evaluate the plasma pharmacokinetics of CAB following repeat oral<br/>administration (Day 1 to Week 4) and CAB LA IM injections throughout the<br/>Injection Phase (Weeks 5-41).</li> </ul> |
| Primary<br>Endpoint | <ul> <li>Safety and tolerability parameters, including adverse events, clinical laboratory<br/>tests, study withdrawals due to AEs, vital signs assessments, and evaluation of<br/>injection site reactions (ISRs), for injection phase (Week 5-41).</li> </ul> |
| | <ul> <li>Plasma CAB AUC(0-τ), Cmax, Cτ, tmax, λz, t½, CL/F, and Vz/F following daily<br/>oral administration of CAB through Day 1 to Week 4.</li> </ul> |
| | • Plasma CAB AUC(0- $\tau$ ), Cmax, C $\tau$ , and tmax following IM injections of CAB LA once every 8 weeks through Weeks 5-41. |
| Secondary<br>Objective | Evaluate the plasma pharmacokinetics of CAB LA throughout the Injection and Long-term Follow-up Phases (Week 5 to Week 89). |
| | Evaluate the safety and tolerability of oral CAB in HIV uninfected Chinese men during the oral lead-in Phase (Day 1 to Week 4) |
| | Evaluate the acceptability of CAB LA injections through 41 weeks. |
| | Explore concentration-effect relationships for various safety and tolerability parameters if relevant. |
| Secondary<br>Endpoint | <ul> <li>Plasma CAB AUC(0-τ), Cmax, Cτ, tmax, λz, t½, CL/F, and Vz/F through Weeks 5-89.</li> </ul> |
| | <ul> <li>Safety and tolerability parameters, including adverse events, study withdrawals due to AEs, vital signs assessments, and clinical laboratory assessments, for oral lead-in phase (Day 1 to Week 4).</li> </ul> |
| | <ul> <li>Injection discontinuation rate, the number and severity of ISRs and additional<br/>acceptability measures.</li> </ul> |
| | Evaluation of relationships between significant safety and tolerability |

| Overview | Key Elements of the RAP |
|---|---|
| | parameters and CAB PK may be explored. |
| Study<br>Design | <ul> <li>This will be an open label, non-randomized, single arm study. Participants will<br/>receive daily oral CAB (30mg tablets) for 4 weeks during the Oral Phase of the<br/>study and intramuscular (IM) injections of 600 mg of CAB LA at Week 5, Week<br/>9, Week 17, Week 25 and Week 33.</li> </ul> |
| | Starting at 8 weeks post last injection, participants will be seen once every 12 weeks for 48 weeks during the follow-up phase. |
| | <ul> <li>Subjects who volunteer to participate in the intensive PK assessment will have<br/>serial blood sampling for measurement of plasma CAB concentrations following<br/>oral administration over a 24 h window starting on Day 27 and ending on Day<br/>28</li> </ul> |
| | PK samples at trough for Oral Phase will be collected for all subjects prior to dose within 20 to 28 hours following oral administration the day prior; Intensive oral PK samples will be collected from approximately 16 participants. |
| | PK Samples for Injection Phase will be collected prior to CAB LA injections at Week 5, 9, 17, 25, and 33 with the exception of 1-week post injection samples at Weeks 6, 10, 18, 26, 34, 37 (4-week post injection sample) and Week 41 |
| | Long-term follow up PK samples will be collected at Week 53, 65, 77, and 89. |
| Planned<br>Analyses | The primary safety analysis and PK analyses including both oral phase and injection phase through Weeks 5 to 41 will be performed after all ongoing participants complete the Week 41 visit or withdraw from the study treatment, whichever comes first. |
| | The end of study analysis will be performed after all ongoing participants complete the Week 89 visit or withdraw from the study treatment, whichever comes first. |
| Analysis<br>Populations | The All Subjects Screened Population will include all subjects who consent to participate in the clinical study. Subjects in this population will be used for disposition summary |
| | The Safety Population will include all subjects who receive at least one dose of the study treatment. Subjects in this population will be used for all demographic and safety summaries or listings, as well as for the analysis of acceptability of CAB LA. |
| | Safety Injection Population will include all subjects received at least one CAB LA injection. Subjects in this population will be used to evaluate the safety and tolerability of CAB LA injection in primary analysis. |
| | Oral PK Population: subjects in the 'Safety population' for whom an intensive oral pharmacokinetic sample was obtained and analysed. PK samples that may be affected by protocol deviations will be reviewed by the study team to determine whether or not the sample will be excluded. This population will be used for reporting of Oral PK data. |

| Overview | Key Elements of the RAP |
|---|---|
| | • Injection (Week 41) PK Population: subjects in the 'Safety population' for whom an injection pharmacokinetic sample was obtained and analysed during Weeks 5 to 41. PK samples that may be affected by protocol deviations will be reviewed by the study team to determine whether or not the sample will be excluded. This population will be used for reporting of Injection PK data from Weeks 5 to 41. |
| | <ul> <li>Injection (Week 89) PK Population: subjects in the 'Safety population' for whom<br/>an injection pharmacokinetic sample was obtained and analysed during Weeks<br/>5 to 89. PK samples that may be affected by protocol deviations will be<br/>reviewed by the study team to determine whether or not the sample will be<br/>excluded. This population will be used for reporting of Injection PK data from<br/>Weeks 5 to 89.</li> </ul> |
| Hypothesis | No formal statistical hypotheses will be evaluated. |
| Primary<br>Analyses | To assess safety of CAB LA, the number and the percent of participants experiencing each safety endpoint will be tabulated including adverse events, clinical laboratory tests, study withdrawals due to AEs, and vital signs assessments. |
| | To assess tolerability of CAB LA, the proportion of participants who terminate from receiving injections prior to the full course due to AE, intolerability of injection, frequency of injections, or burden of procedures related to injections out of those participants that received at least one injection. |
| | To assess the plasma pharmacokinetics of CAB following repeat oral administration (Day 1 to Week 4) and CAB LA IM injections throughout the Injection Phase (Week 5 to Week 41). |
| Secondary<br>Analyses | To assess the plasma pharmacokinetics of CAB LA throughout the Injection and Long-term Follow-up Phases (Week 5 to Week 89). |
| | To assess the safety and tolerability of oral CAB, each safety and tolerability endpoint will be tabulated including adverse events, study withdrawals due to AEs, vital signs assessments and clinical laboratory assessments. |
| | To assess the acceptability of the CAB LA, injection discontinuation rate, the number and severity of ISRs, and the proportion (with 95% CI for the CAB LA arm) of participants who would consider using CAB LA for HIV prevention in the future will be tabulated among all enrolled participants (including those who terminated product use during the trial. |
| | Overall treatment satisfaction score and answers to each individual question on<br>HIV-PrevTSQc will be summarized to evaluate tolerability |

#### 2. SUMMARY OF KEY PROTOCOL INFORMATION

## 2.1. Changes to the Protocol Defined Statistical Analysis Plan

The current adverse events of special interest (AESIs) included in the protocol are seizures and seizure like events, diarrhea, hypertriglyceridemia/hypercholesterolemia, decline in renal function, proximal renal tubule dysfunctions and proteinuria.

We are modifying the study AESIs to align them with the rest of the Cabotegravir programme, now that the AESIs related to CAB have now been fully developed.

The RAP AESIs will differ from the AESIs defined in the protocol. AESIs of hepatoxicity, hypersensitivity reactions, injection site reactions, impact on creatinine, and neuropsychiatric events have been added to the list of AESIs for the RAP.

The events of diarrhea, hypertriglyceridemia/hypercholesterolemia, have been removed for the list of AESIs in the RAP.

Seizures and seizure like events, Decline in renal function, proximal renal tubule dysfunctions, proteinuria, which were defined in the protocol, will be kept as the AESIs for the study.

## 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| Evaluate the safety and tolerability of the injectable agent, cabotegravir (GSK1265744) long acting (CAB LA) injectable (600 mg dose administered every 4 weeks for 2 doses followed by every 8 weeks for 3 doses) through Week 5-41 in HIV-1 uninfected Chinese men. | Safety and tolerability parameters, including adverse events, clinical laboratory tests, study withdrawals due to AEs, vital signs assessments, and evaluation of injection site reactions (ISRs). |
| Evaluate the plasma pharmacokinetics of CAB following repeat oral administration (Day 1 to Week 4) and CAB LA IM injections throughout the Injection Phase (Week 5 to Week 41). | Plasma CAB AUC(0-τ), Cmax, Cτ, tmax, λz, t½, CL/F, and Vz/F at Week 4 following daily oral administration of CAB. Plasma CAB AUC(0-τ), Cmax, Cτ, and tmax at Week 41 following IM injections of CAB LA. |
| Secondary Objectives | Secondary Endpoints |
| Evaluate the plasma pharmacokinetics of CAB LA throughout the Injection and Longterm Follow-up Phases (Week 5 to Week 89) | Plasma CAB AUC(0- $\tau$ ), Cmax, C $\tau$ , tmax, $\lambda z$ , t½, CL/F, and Vz/F |
| Evaluate the safety and tolerability of oral CAB in HIV uninfected Chinese men during the oral lead-in Phase (Day 1 to Week 4) | Safety and tolerability parameters, including adverse events, study withdrawals due to AEs, vital signs assessments and clinical laboratory |

| Objectives | Endpoints |
|---|---|
| | assessments. |
| Evaluate the acceptability of CAB LA injections through 41 weeks. | Injection discontinuation rate, the number and severity of ISRs and additional acceptability measures. |
| Explore concentration-effect relationships for various safety and tolerability parameters if relevant. | Evaluation of relationships between significant safety and tolerability parameters and CAB PK may be explored. |

## 2.3. Study Design



This study is an open label (OL) Phase 1, multi-site, study to evaluate the PK, safety, tolerability, and acceptability of CAB LA in adult male participants. Eligible participants will receive oral CAB tablets as well as open label CAB LA.

| Design Features | Oral lead-in phase is from Day 1 to week 4; injection phase is from week 5 to week 41; and follow-up phase is from week 41 to week 89 |
|---|---|
| Dosing | Oral CAB tablet is 30mg and dose level=1 tablet; CAB Sterile Suspension for Injection Vial is 200mg/mL and dose level = 600mg (3mL) Participants will receive daily oral CAB (30mg tablets) for 4 weeks during the Oral Phase of the study and IM injections of 600 mg of CAB LA at Week 5, Week 9, Week 17, Week 25 and |
| | Week 33. |

| Overview of Study Design and Key Features | |
|---|---|
| Treatment Assignment | Eligible participants will receive oral CAB tablets in the first four |
| | weeks, and will received CAB LA injections since Week 5 |
| | following planned schedules. |
| Interim Analysis | No interim analysis is planned in this study. |

## 2.4. Statistical Hypotheses

No formal statistical hypotheses will be evaluated. The study is designed to evaluate the PK, safety, tolerability, and acceptability of the injectable agent, CAB LA (600 mg dose administered at 8-week intervals after 2 initial doses 4 weeks apart) in HIV-uninfected men in China where at least 60% of the men are of a population who have sex with men. Where appropriate, an estimation approach will be taken, and point estimates and confidence intervals will be constructed.

#### 3. PLANNED ANALYSES

#### 3.1. Interim Analyses

No formal interim analysis is planned in the study.

However, two preliminary PK analyses during the study will be performed in an informal manner. One will be after all planned participants complete the oral phase, and the other one will be after 50% of planned participants complete Week 17 visit. Safety data will be provided after all planned participants complete the oral phase as well. Study team will review preliminary safety and PK data.

## 3.2. Final Analyses

The primary safety analysis and PK analyses including both oral phase and injection phase through Weeks 5 to 41 will be performed after all ongoing participants complete the Week 41 visit and datasets have been authorized. Other secondary analyses as mentioned, where appropriate, will also be performed. The end of study analysis will be performed after all ongoing participants complete the Week 89 visit. All planned primary and secondary analyses will be included in the second formal analyses.

The planned analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have completed the specific study visit (i.e. week 41 or week 89) as defined in the protocol.
- 2. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.

## 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All Subjects<br>Screened | Comprise of all subjects who consent to participate in the clinical study. | Disposition summary |
| Safety | Comprise of all subjects who receive at least one dose of the study treatment. | <ul> <li>All demographic</li> <li>General safety analyses</li> <li>Safety analysis for the oral phase</li> <li>Analysis of acceptability of CAB LA</li> </ul> |
| Safety Injection | Comprise of all subjects received at least one CAB LA injection | <ul> <li>Safety and tolerability<br/>analyses of CAB LA in<br/>primary and extended<br/>analyses</li> </ul> |
| Oral | Will consist of all subjects in the 'Safety | Oral PK Concentration |
| Pharmacokinetic<br>(PK) | population' for whom an intensive oral pharmacokinetic sample was obtained and analysed. PK samples that may be affected by protocol deviations will be reviewed by the study team to determine whether or not the sample will be excluded. | Oral PK Parameters |
| Injection (Week 41) Pharmacokinetic (PK) | Will consist of all subjects in the 'Safety population' for whom an injection pharmacokinetic sample was obtained and analysed during Weeks 5 to 41. PK samples that may be affected by protocol deviations will be reviewed by the study team to determine whether or not the sample will be excluded. | <ul> <li>Injection PK Concentration</li> <li>Injection PK Parameters</li> </ul> |
| Injection (Week 89) Pharmacokinetic (PK) | Will consist of all subjects in the 'Safety population' for whom an injection pharmacokinetic sample was obtained and analysed during Weeks 5 to 89. PK samples that may be affected by protocol deviations will be reviewed by the study team to determine whether or not the sample will be excluded. | <ul> <li>Injection PK<br/>Concentration</li> <li>Injection PK<br/>Parameters</li> </ul> |

## NOTES:

Please refer to Appendix 14: List of Data Displays which details the population to be used for each display being generated.

#### 4.1. Protocol Deviations

- Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.
- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.
  - O Data will be reviewed prior to freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
  - This dataset will be the basis for the summaries and listings of protocol deviations.
- A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Table 1 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 1 Overview of Appendices

| Section | Component |
|---|---|
| 10.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population |
| 10.2 | Appendix 2: Time & Events |
| 10.3 | Appendix 3: Assessment Windows |
| 10.4 | Appendix 4: Treatment States and Phases |
| 10.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 10.6 | Appendix 6: Derived and Transformed Data |
| 10.7 | Appendix 7: Premature Withdrawals & Handling of Missing Data |
| 10.8 | Appendix 8: Values of Potential Clinical Importance |
| 10.9 | Appendix 9: Multicenter Studies |
| 10.10 | Appendix 10: Examination of Covariates, Subgroups & Other Strata |
| 10.11 | Appendix 11: Multiple Comparisons & Multiplicity |
| 10.12 | Appendix 12: Model Checking and Diagnostics for Statistical Analyses. |
| 10.13 | Appendix 13: Abbreviations & Trade Marks |
| 10.14 | Appendix 14: List of Data Displays |

#### 6. STUDY POPULATION ANALYSES

## 6.1. Overview of Planned Analyses

The study population analyses will be based on the safety population, unless otherwise specified. All summary data and statistics are calculated from available data, unless otherwise specified.

Table 2 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 14: List of Data Displays.

Table 2 Overview of Planned Study Population Analyses

| Display Type | Data | Displays Gene | rated |
|---|---|---|---|
| | Table | Figure | Listing |
| Disposition | | | |
| Retention Rate and Reasons for Withdrawals | Υ | | Υ |
| Demography and Baseline Characteristics | | | |
| General Demographics Characteristics | Υ | | Υ |
| Medical History and Concomitant Medications | | | |
| Medical History | Υ | | Υ |
| Prior Medications | Υ | | Y |
| Concomitant Medications | Υ | | Υ |
| Protocol Deviations | | | |
| Deviation of Inclusion/Exclusion Criteria | Υ | | Y |
| Important Protocol Deviations | Y | | Y |

#### NOTES:

Y = Yes display generated.

### 6.1.1. Disposition

The reasons of screening failure will be summarized based on the screened population. The number and percentage of each reason will be tabulated.

A summary of subject disposition by phase will be provided, including the number and percentage of subjects entering oral/injection phase, the number and percentage of subjects completing oral/injection phase and the number and percentage of subjects withdrawing from oral/injection phase.

Subject disposition data will be presented in a listing.

#### 6.1.2. Demographics

General demographics including age, self-identified gender when entering the study, and ethnicity will be summarized.

A subject's age is calculated using the year part of informed consent form (ICF) – year of birth collected in CRF.

## 6.1.3. Medical History

Summaries of medical history will be presented by GSK pre-specified body system categories as collected in the eCRF. Number and percentage of subjects in each category will be tabulated.

#### 6.1.4. Prior and Concomitant Medications

Medications will be coded to therapeutic drug classes and generic drug names using the GSKDRUG 1.4 or later. Medications initiated prior to the Day 1 of the study will be counted as prior medications. Concomitant medications are defined as medications that are taken on or after the Day 1. Medications initiated prior to the Day 1 and continued after the Day 1 will be counted as both prior and concomitant medications.

Summaries showing the number and percentage of subjects who take prior or concomitant medications will be presented by therapeutic drug class and generic drug name.

#### 6.1.5. Protocol Deviation

Important protocol deviations (PD) will be summarized PD category and subcategory, and will also be presented in a listing. A separate summary table and a listing will be provided for subjects with deviation of the inclusion/exclusion criteria in the safety population

#### 7. PRIMARY STATISTICAL ANALYSES

## 7.1. Safety Analyses of CAB LA

Four study phases are defined for this study: screening phase, oral phase, injection phase and follow-up phase (see Appendix 4 for the definition of each phase).

The primary safety analysis will be conducted after all ongoing participants complete the Week 41 visit and datasets have been authorized. All data from injected participants collected from Week 5 to Week 41 (i.e., in the injection phase) will be analysed. Analysis endpoints will include Grade 2 or higher clinical and laboratory events that occur from the initial injection to 8 weeks after the last injection among participants who receive at least one injection.

The extended safety analysis will be conducted after all ongoing participants complete the Week 89 visit and datasets have been authorized. All data from injected participants collected from Week 5 to Week 89 (i.e., in the injection phase and the follow-up phase) will be analysed. Analysis endpoints are the same as in the primary safety analysis.

To assess safety, the number and the percent of participants experiencing each safety endpoint will be tabulated. Each participant will contribute once in each category (i.e., only for the highest severity AE) for the evaluation of safety.

## 7.1.1. Injection Site Reaction

The number and percentage of participants experiencing each type of injection site reaction sign or symptom will be tabulated by severity from the safety injection population. For a given sign or symptom, each participant's ISR will be counted once under the maximum severity for all injection visits. Overall summary of ISR and summary of ISR by needle length will both be provided. ISR related details, such as cardiovascular activity, strength training exercise, will be listed only.

Table 3 provides an overview of the planned ISR analyses, with full details of data displays being presented in Appendix 14: List of Data Displays.

Table 3 Overview of Planned ISR Analyses

| Display Type | Data Displays Generated | | | | | | |
|---|---|---|---|---|---|---|---|
| | S | tats Analysis | 3 | Sum | mary | Individual | |
| | T | F | L | T | F | F | L |
| ISR Analyses | | | | | | | |
| All ISR Symptoms | | | | Υ | | | Υ |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

#### 7.1.2. Adverse Events

Adverse events will be tabulated using MedDRA (v20.0 or above) system organ class (SOC) and preferred terms (PT), or preferred terms alone, by study phase. The number and percentage of participants experiencing each specific AEs (Grade 2 or higher, All AEs, SAEs, AEs leading to permanent treatment discontinuation or study withdrawal) will be tabulated. Number of subjects in the safety population who entered the study phase will be used as denominator in the calculation of percentages.

Drug-related AEs, SAEs, and Grade 2-4 AEs will also be tabulated. Any AE is assumed to be study treatment-related if relationship is marked 'YES' on CRF or value is missing. In addition, a summary table will be created for AEs by maximum severity by study phase. Common AEs are defined as AEs occurring in >=5% subjects during the study (based on preferred term). Common AEs, common non-serious AEs, common Grade 2-4 AEs, and common drug-related Grade 2-4 AEs will be tabulated.

All AE tables will be presented in a decreasing frequency order of SOC or PT unless otherwise specified.

Table 4 provides an overview of the planned AE analyses, with full details of data displays being presented in Appendix 14: List of Data Displays.

| | | Data Displays Generated | | | | | |
|---|---|---|---|---|---|---|---|
| Display Type | | Stats Analys | sis | Sum | mary | Individual | |
| | T | F | L | T | F | F | L |
| AE Analyses | | | | | | | |
| All AEs | | | | Y | | | Υ |
| Grade 2 or higher AEs | | | | Y | | | Υ |
| SAEs | | | | Υ | | | Υ |
| AE leading to treatment | | | | Y | | | Υ |
| discontinuation or study | | | | | | | |
| withdrawal | | | | | | | |
| Drug-related AEs | | | | Υ | | | |
| Drug-related SAEs | | | | Y | | | |
| Drug-related Grade 2 or | | | | Υ | | | |
| higher AEs | | | | | | | |
| Common AEs | | | | Y | | | |
| Common non-serious AEs | | | | Υ | | | |

Table 4 Overview of Planned AE Analyses

#### NOTES:

Common Grade 2-4 AEs Common drug-related Grade 2-4 AEs

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

#### 7.1.3. Clinical Laboratory Tests

All clinical laboratory tests will be graded according to the Appendix 7 from the study protocol. Grade 2 or higher laboratory events will be tabulated by number and percentage of subjects with the event by study phase.

Change from baseline in hematology, fasting chemistry, fasting lipid profile, and coagulation profile will be summarized by visit. For the definition of baseline, refer to Section 10.5.2. Urinalysis and urine chemistry results will be summarized by visit as either categorical values or as continuous values, depending on the type of the parameter.

For each lab test, shift from baseline table will be provided based on toxicity grade, both by visit and for the shift to maximum toxicity grade in each study phase. Data collected at unscheduled visits will not be included in the by-visit summary, but will be used in the calculation of maximum grade in each study phase. Subjects having both high and low values will be counted in both High and Low categories for the summary by study phase.

All lab data, as well as lab data for subjects with Grade 2 or higher abnormalities, will be listed. Abnormal data will be listed with an indicator, which is low/high relative to normal range. All laboratory results from local labs, if any, will be listed only

Table 5 provides an overview of the planned lab test analyses, with full details of data displays being presented in Appendix 14: List of Data Displays.

| | | Abso | olute | | Change from Baseline | | | |
|---|---|---|---|---|---|---|---|---|
| Display Type | Summary | | Indiv | ridual | Sum | mary | Individual | |
| | T | F | F | L | T | F | F | L |
| Laboratory Test Analys | ses | | | | | | | |
| Grade 2 or high | Υ | | | | | | | |
| laboratory events | | | | | | | | |
| Clinical Chemistry | | | | Υ | Υ | | | |
| Hematology | | | | Υ | Υ | | | |
| Fasting Lipid Profile | | | | Υ | Υ | | | |
| Coagulation Profile | | | | Υ | Υ | | | |
| Urinalysis and Urine | Υ | | | Υ | Υ | | | |
| Chemistry | | | | | | | | |
| Other lab data | | | | Υ | | | | |
| including local lab | | | | | | | | |

Table 5 Overview of Planned Lab Test Analyses

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

#### 7.1.4. Vital Sign Assessments

Change from baseline in vital signs, including temperature, systolic and diastolic blood pressure, and pulse rate and respiratory rate will be summarized by study visit. For the

definition of baseline, refer to Section 10.5.2. Shift from baseline table (with respect to clinical concern range) will also be provided.

All vital signs, as well as vital signs for subjects with abnormalities of potential clinical importance, will be listed with an indicator, which is low/high relative to clinical concern range.

Table 6 provides an overview of the planned vital sign analyses, with full details of data displays being presented in Appendix 14: List of Data Displays.

Table 6 Overview of Planned Vital Sign Analyses

| Display Type | | Abso | olute | | Change from Baseline | | | |
|---|---|---|---|---|---|---|---|---|
| | Summary | | Individual | | Summary | | Individual | |
| | T F | | F | L | Т | F | F | L |
| Vital Signs | | | | | | | | |
| Vital signs | | | | Υ | Υ | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

#### 7.1.5. Death

Both primary and secondary causes, if any, will be listed for each deceased participant.

Table 7 provides an overview of the planned death analyses, with full details of data displays being presented in Appendix 14: List of Data Displays.

Table 7 Overview of Planned Death Analyses

| Display Type | Data Displays Generated | | | | | | |
|---|---|---|---|---|---|---|---|
| | S | tats Analysis | 3 | Sum | mary | Individual | |
| | T | ΓF | | T F | | F | L |
| Death Analysis | | | | | | | |
| Death | | | | | | | Υ |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

## 7.2. Tolerability Analyses of CAB LA

The tolerability analyses will be based on the safety injection population, unless otherwise specified. All summary data and statistics are calculated from available data, unless otherwise specified.

To assess tolerability of CAB LA, the proportion (with 95% confidence interval) of participants who terminate from receiving injections prior to the full course due to AE, intolerability of injection, frequency of injections, or burden of procedures related to injections will be calculated out of those participants that received at least one injection.

A questionnaire will also be used to assess participant tolerability and satisfaction to the treatment. For each question, the responses will be summarized by the proportion of participants reporting the response out of all those that answered the question. An overall treatment satisfaction score will be calculated for each participant.

Total score is defined as the sum of the scores for individual questions. If less than or equal to 50% of the questions for an individual participant are missing, the missing total scores will be estimated using the average of the existing questions multiplied by twelve; if more than 50% of the questions for an individual participant are missing, the total score will not be estimated and will be considered as missing. When calculating total scores,



Table 8 provides an overview of the planned tolerability analyses, with further details of data displays being presented in Appendix 14: List of Data Displays.

Table 8 Overview of Planned Tolerability Analyses

| | | Data Displays Generated | | | | | |
|---|---|---|---|---|---|---|---|
| Display Type | S | tats Analysis | 3 | Sum | mary | Individual | |
| | Τ | F | L | Т | F | F | L |
| CAB LA Discontinuation | | | | | | | |
| Injection | | | | Υ | | | Υ |
| Discontinuation Rate | | | | | | | |
| Treatment Satisfaction | n Questio | nnaire | | | | | |
| Each question in the | | | | Υ | | | Υ |
| questionnaire | | | | | | | |
| Treatment total | | | | Y | | | Υ |
| satisfaction score | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data

## 7.3. Primary Pharmacokinetic Analyses

### 7.3.1. Overview of Planned Primary Pharmacokinetic Analyses

The primary pharmacokinetic (PK) analyses will be based on the Oral PK and Injection (Week 41) PK populations, unless otherwise specified.

Table 9 provides an overview of the planned efficacy analyses, with full details of data displays being presented in Appendix 14: List of Data Displays.

Table 9 Overview of Planned Primary Pharmacokinetic Analyses

| Display Type | Untransformed | | | | | | Log-1 | ransf | ormed | i | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stats Analysis | Summary Individual | | | Stats Analysis | | | Summary | | Individual | | |
| | T F L | Т | F | F | L | Т | F | L | Т | F | F | L |
| Oral/Injection | | | | | | | | | | | | |
| PK Concentrations | | Υ | <b>Y</b> [1] | <b>Y</b> [1] | Υ | | | | | | | |
| Plasma PK Parameters | Υ | Υ | | | Υ | | | Υ | Υ | | | |

#### NOTES:

- T = Table, F = Figure, L = Listings, Y = Display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

#### 7.3.2. Primary Drug Concentration Measures

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 10.5.3 Reporting Process & Standards).

<sup>[1]</sup> Linear and Semi-Logarithmic plots will be created on the same display.

### 7.3.3. Primary Pharmacokinetic Parameters

#### 7.3.3.1. Deriving Primary Pharmacokinetic Parameters

- Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 10.5.3 Reporting Process & Standards).
- The pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using Phoenix WinNonlin Version 6.4 or higher.
- All calculations of non-compartmental parameters will be based on actual sampling times, and all concentrations will be included in the estimation of PK parameters regardless of whether samples are collected within the specified time window or not.
- Pharmacokinetic parameters described in Table 10 will be determined from the plasma concentration-time data, as data permits.

 Table 10
 Derived Primary Pharmacokinetic Parameters

| Parameter | Parameter Description |
|---|---|
| AUC(0-τ) | Area under the concentration-time curve over the dosing interval will be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. |
| Cmax | Maximum observed concentration, determined directly from the concentration-time data. |
| tmax | Time to reach Cmax, determined directly from the concentration-time data. |
| Сτ | Observed concentration at the end of the dosing interval, determined directly from the concentration-time data. |
| t½ | Terminal absorption elimination half-life will be calculated as: $t\frac{1}{2} = \ln 2 / \lambda z$ |
| λz | Terminal absorption elimination rate constant |
| CL/F | Clearance (adjusted for bioavailability, F) will be calculated as: CL/F = Dose / AUC(0-τ) |
| Vz/F | Volume of distribution (adjusted for bioavailability, F) will be calculated as: $Vz/F = CL / \lambda z$ |

#### NOTES:

- Additional parameters may be included as required.
- λz, CL/F, Vss and t½ will be determined for the Oral PK population only in the primary analysis; these parameters will be further explored for the Injection (Week 89) PK population (Section 8.1.3.1).

#### 7.3.3.2. Statistical Analysis of Primary Pharmacokinetic Parameters

The following pharmacokinetic statistical analyses will only be performed, if sufficient data is available (i.e. if subjects have well defined plasma profiles).

### **Pharmacokinetic Statistical Analyses**

#### Endpoint(s)

• Plasma primary PK endpoints include  $C\tau$ , as data permit

#### **Model Specification**

#### Assessment of Accumulation (Injection Phase only):

To determine accumulation of plasma CAB following treatment with CAB LA, the log-transformed Cτ values for CAB will be analyzed using a mixed effects model (ANOVA) as appropriate to the study design, fitting fixed effect terms for visit and treating subject as a random effect. Point estimates and 90% confidence intervals (CIs) for the differences of interest (i.e. accumulation of CAB based on AUC(0-τ): Week 34 / Week 6) will be constructed using the residual variance.

#### Attainment of Steady state (Injection Phase only):

• If data permit, a statistical analysis of steady-state trough concentrations (Cτ) will be performed after log-transformation of Cτ on Weeks 17, 25, 33, and 41 to evaluate whether steady state was achieved using the Helmert transformation approach. A mixed effect model (ANOVA) will be fitted by visit (as a categorical covariate) as a fixed effect term and subject as a random effect term. The comparison will begin with Week 17 vs. the average of Weeks 25 through Week 41. If the p-value for Week 17 vs. the average of Week 25 through Week 41 comparison is ≤0.05 (i.e. steady state not achieved at Week 17), then the comparison will continue with Week 25 vs. Week 33 through Week 41.

#### **Model Checking & Diagnostics**

Refer to Appendix 12: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- Statistical analysis of accumulation of plasma CAB following treatment with CAB LA will be presented in tabular format with geometric mean ratios between Week 34 and Week 6, and 90% CIs for the ratios of  $C\tau$  for CAB.
- In steady-state analysis, the ratio of Geometric LS means and its 95% CI will be presented for the comparison(s).

## 8. SECONDARY STATISTICAL ANALYSES

## 8.1. Secondary Pharmacokinetic Analyses

## 8.1.1. Overview of Planned Secondary Pharmacokinetic Analyses

The secondary pharmacokinetic (PK) analyses will be based on the Injection (Week 89) PK population, unless otherwise specified.

Table 11 provides an overview of the planned analyses, with full details being presented in Appendix 14: List of Data Displays.

Table 11 Overview of Planned Secondary Pharmacokinetic Analyses

| Display Type | | Untransformed | | | | Log-Transformed | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stat | Stats Analysis S | | Summary | | Indiv | idual | Stat | s Ana | lysis | Sum | mary | Indiv | idual |
| | Т | F | L | Т | F | F | L | Т | F | L | Т | F | F | L |
| Oral/Injection | Oral/Injection | | | | | | | | | | | | | |
| PK Concentrations | | | | Υ | <b>Y</b> [1] | Υ[1] | Υ | | | | | | | |
| Plasma PK Parameters | Υ | | | Υ | | | Υ | | | Υ | Υ | | | |

#### NOTES:

- T = Table, F = Figure, L = Listings, Y = Display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

#### 8.1.2. Secondary Drug Concentration Measures

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 10.5.3 Reporting Process & Standards).

## 8.1.3. Secondary Pharmacokinetic Parameters

#### 8.1.3.1. Deriving Secondary Pharmacokinetic Parameters

- Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 10.5.3 Reporting Process & Standards).
- The pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using Phoenix WinNonlin Version 6.4 or higher.
- All calculations of non-compartmental parameters will be based on actual sampling times, and all concentrations will be included in the estimation of PK parameters regardless of whether samples are collected within the specified time window or not.
- Pharmacokinetic parameters described in Table 12 will be determined from the plasma concentration-time data, as data permits.

<sup>[1]</sup> Linear and Semi-Logarithmic plots will be created on the same display.

Table 12 Derived Secondary Pharmacokinetic Parameters

| Parameter | Parameter Description |
|---|---|
| AUC(0-τ) | Area under the concentration-time curve over the dosing interval will be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. |
| Cmax | Maximum observed concentration, determined directly from the concentration-time data. |
| tmax | Time to reach Cmax, determined directly from the concentration-time data. |
| Сτ | Observed concentration at the end of the dosing interval, determined directly from the concentration-time data. |
| t½ | Terminal absorption elimination half-life will be calculated as: $t\frac{1}{2} = \ln 2 \ / \ \lambda z$ |
| λz | Terminal absorption elimination rate constant |
| CL/F | Clearance (adjusted for bioavailability, F) will be calculated as: |
| | $CL/F = Dose / AUC(0-\tau)$ |
| Vz/F | Volume of distribution (adjusted for bioavailability, F) will be calculated as: Vz/F = CL / λz |

#### NOTES:

Additional parameters may be included as required.

## 8.2. Safety and Tolerability Analyses of Oral CAB

The safety and tolerability analyses of oral CAB will include Grade 2 or higher clinical and laboratory events occurred during the oral phase. Analysis time frame is from the first date of taking oral CAB tablet to the date right before the first CAB LA injection. For subjects who withdraw treatment from the oral phase, the analysis will include all safety and tolerability assessments from the first date of taking oral CAB tablet up to the date of last study visit.

Safety endpoints including adverse events, laboratory test, vital signs, and death will be analysed. The same analysis approaches will be conducted as in the primary analysis, but with different time frame.

Table 13 provides an overview of the planned analyses, with full details of data displays being presented in Appendix 14: List of Data Displays.

Table 13 Overview of Planned AE, LB, VS, and Death Analyses

| | | | Data I | Displays Ge | nerated | | |
|---|---|---|---|---|---|---|---|
| Display Type | | tats Analysis | ) | | mary | Indivi | dual |
| | Т | F | L | Т | F | F | L |
| AE Analyses | | | | | | | |
| All AEs | | | | Υ | | | Υ |
| Grade 2 or higher AEs | | | | Υ | | | Υ |
| SAEs | | | | Υ | | | Υ |
| AE leading to | | | | Υ | | | Υ |
| treatment | | | | | | | |
| discontinuation or | | | | | | | |
| study withdrawal | | | | | | | |
| Drug-related AEs | | | | Υ | | | |
| Drug-related SAEs | | | | Υ | | | |
| Drug-related Grade 2 | | | | Υ | | | |
| or higher AEs | | | | | | | |
| Common AEs | | | | Y | | | |
| Common non-serious | | | | Υ | | | |
| AEs | | | | | | | |
| Common Grade 2-4 | | | | Υ | | | |
| AEs | | | | | | | |
| Common drug-related | | | | Υ | | | |
| Grade 2-4 AEs | | | | | | | |
| Laboratory Tests | | | | | | | |
| Grade 2 or higher | | | | Υ | | | |
| laboratory events | | | | | | | |
| Clinical Chemistry | | | | Υ | | | Υ |
| Hematology | | | | Y | | | Υ |
| Fasting Lipid Profile | | | | Υ | | | Υ |
| Urinalysis | | | | Υ | | | Υ |
| Coagulation Profile | | | · | Υ | | | Υ |
| Other lab data | | | | | | | Υ |
| including local lab | | | | | | | |
| Vital Sign Analysis | | | | | | | |
| Vital Signs | | | | Υ | | | Υ |
| Death Analysis | | | | | | | |
| Death | | | | | | | Υ |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

## 8.3. Acceptability of CAB LA

The secondary acceptability analyses will be based on safety population, unless otherwise specified. All summary data and statistics are calculated from available data, unless otherwise specified.

To assess acceptability of the CAB LA, the proportion (with 95% confidence interval) of participants who would consider using CAB LA for HIV prevention in the future will be calculated among all subjects in the safety population (including those who terminated product use during the trial). Participants will be asked if they would consider using CAB LA for HIV prevention in the future at their Week 41 visit or at their withdrawal visit, whichever occurs first. Patients who are lost to follow up or with missing responses will be presented as such in a separate category.

Table 14 provides an overview of the planned acceptability analyses, with further details of data displays being presented in Appendix 14: List of Data Displays.

Table 14 Overview of Planned Acceptability Analyses

| | Data Displays Generated | | | | | | |
|---|---|---|---|---|---|---|---|
| Display Type | S | tats Analysis | 3 | Sum | mary | Individual | |
| | T | F | L | T | F | F | L |
| Acceptability of the C | ability of the CAB LA | | | | | | |
| participants who would consider using | | | | Y | | | Υ |
| CAB LA | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

# 8.4. Concentration-effect Relationships for Safety and Tolerability Parameters

Evaluation of relationships between significant safety and tolerability parameters and CAB PK may be explored.

## 8.5. General Safety Analyses

This section will describe safety analyses that are not mentioned in Section 7.1 or Section 8.2, but usually are performed as safety assessment.

## 8.5.1. Extent of Exposure to CAB

Duration of exposure to CAB and cumulative dose (see Section 10.6.2 for the definition) will be summarized for the oral phase and the injection phase separately. Overall exposure to the study drug and to the study (for safety evaluation) will also be calculated and summarized. Exposure data will also be listed.

Table 15 provides an overview of the planned analyses, with full details of data displays being presented in Appendix 14: List of Data Displays.

Table 15 Overview of Planned Analyses for Extent of Exposure

| | Data Displays Generated | | | | | | |
|---|---|---|---|---|---|---|---|
| Display Type | S | tats Analysis | 3 | Sum | mary | Individual | |
| | T F L | | | T F | | F | L |
| Extent of Exposure | | | | | | | |
| Extent of exposure | | | | Υ | | | Υ |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

## 8.5.2. Possible suicidality-related Adverse Events

Possible suicidality-related will be listed.

Table 16 provides an overview of the planned analyses, with full details of data displays being presented in Appendix 14: List of Data Displays.

Table 16 Overview of Analyses for possible suicidality-related AEs

| | Data Displays Generated | | | | | | |
|---|---|---|---|---|---|---|---|
| Display Type | S | tats Analysis | S | Sum | mary | Individual | |
| | T F L | | | T | F | F | L |
| AE Analyses | | | | | | | |
| Possible Suicidality- | | | | | | | Υ |
| Related Adverse Event | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

#### 8.5.3. Social Harms

Details of social harms collected on the eCRF will be listed for each participant.

Table 17 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 14: List of Data Displays.

Table 17 Overview of Planned Study Population Analyses

| Display Type | Data Displays Generated | | |
|------------------|-------------------------|--------|---------|
| | Table | Figure | Listing |
| Social Harms | | | |
| All Social Harms | | | Y |

#### NOTES:

• Y = Yes display generated.

#### 8.5.4. ECG

ECG test will be performed at Screening only. Details collected on the eCRF will be listed for each subject. Baseline ECG findings (normal, abnormal – not clinically significant, or abnormal – clinically significant) will be summarized by number and percentage of subjects and presented as part of the 'Demographic Characteristics' table.

Table 18 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 14: List of Data Displays.

Table 18 Overview of Planned Study Population Analyses

| Display Type | Data Displays Generated | | |
|----------------------------|-------------------------|--------|---------|
| | Table | Figure | Listing |
| ECG | | | |
| ECG Parameters and Results | Y | | Υ |

#### NOTES:

Y = Yes display generated.

#### 8.5.5. Cardiovascular Events

Any cardiovascular events will be listed only.

Table 19 provides an overview of the planned cardiovascular event analyses, with full details of data displays being presented in Appendix 14: List of Data Displays.

Table 19 Overview of Planned Cardiovascular Event Analyses

| | Data Displays Generated | | | | | | |
|---|---|---|---|---|---|---|---|
| Display Type | S | tats Analysis | 3 | Sum | mary | Individual | |
| | T F L | | T F | | F | L | |
| CV Event Analyses | | | | | | | |
| All CV events | | | | | | | Υ |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

#### 8.5.6. Liver Events

Number and percentage of subjects with liver events will be tabulated by study phase. Number and percentage of subjects with clinical significant hepatobiliary laboratory abnormalities during the study will also be tabulated. Full information of liver events will be listed.

Table 20 provides an overview of the planned liver event analyses, with full details of data displays being presented in Appendix 14: List of Data Displays.

 Table 20
 Overview of Planned Liver Event Analyses

| | Data Displays Generated | | | | | | |
|---|---|---|---|---|---|---|---|
| Display Type | 9 | Stats Analysis | S | Sum | mary | Individual | |
| | T | F | L | T | F | F | L |
| Liver Event Analyses | | | | | | | |
| All liver events | | | | Υ | | | Υ |
| Hepatobiliary | | | | Υ | | | |
| laboratory | | | | | | | |
| abnormalities | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

#### 9. REFERENCES

Dube MP, Stein JH, Aberg JA, Fichtenbaum CJ, Gerber JG, Tashima KT et al. Guidelines for the evaluation and management of dyslipidemia in human immunodeficiency virus (HIV)-infected adults receiving antiretroviral therapy: recommendations of the HIV Medical Association of the Infectious Disease Society of America and the Adult AIDS Clinical Trials Group. *Clin Infect Dis* 2003; 37(5):613-27.

GlaxoSmithKline Document Number 2016N293702\_00 (Original – 20-JUL-2017): An Open Label, Phase 1 Study to Evaluate the PK, Safety, Tolerability and Acceptability of Long Acting Injections of the HIV Integrase Inhibitor, Cabotegravir (CAB; GSK1265744) in HIV Uninfected Chinese Men (20-JUL-2017)

GlaxoSmithKline Document Number 2016N293702\_01 (Original – 20-JUL-2017): An Open Label, Phase 1 Study to Evaluate the PK, Safety, Tolerability and Acceptability of Long Acting Injections of the HIV Integrase Inhibitor, Cabotegravir (CAB; GSK1265744) in HIV Uninfected Chinese Men (06-JUN-2018)

Levey AS, Stevens LA, Schmid CH, Zhang YL, Castro AF, Feldman HI, et.al. A new equation to estimate glomerular filtration rate. Ann Int Med. 2009; 150: 604-12.

## 10. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 4 | : Analysis Populations |
| Section 10.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol |
| | Population |
| RAP Section 5 | : General Considerations for Data Analyses & Data Handling Conventions |
| Section 10.2 | Appendix 2: Time and Events |
| Section 10.3 | Appendix 3: Assessment Windows |
| Section 10.4 | Appendix 4: Treatment States & Phases |
| Section 10.5 | Appendix 5: Data Display Standards & Handling Conventions |
| | <ul> <li>Study Treatment &amp; Sub-group Display Descriptors</li> </ul> |
| | Baseline Definitions & Derivations |
| | Reporting Process & Standards |
| Section 10.6 | Appendix 6: Derived and Transformed Data |
| | General, Study Population & Safety |
| Section 10.7 | Appendix 7: Premature Withdrawals & Handling of Missing Data |
| | Premature Withdrawals |
| | Handling of Missing Data |
| Section 10.8 | Appendix 8: Values of Potential Clinical Importance |
| Section 10.9 | Appendix 9: Multicentre Studies |
| Section 10.10 | Appendix 10: Examination of Covariates and Subgroups & Other Strata |
| Section 10.11 | Appendix 11: Multiple Comparisons and Multiplicity |
| Section 10.12 | Appendix 12: Model Checking and Diagnostics for Statistical Analyses |
| Other RAP App | endices |
| Section 10.13 | Appendix 13: Abbreviations & Trade Marks |
| Section 10.14 | Appendix 14: List of Data Displays |

# 10.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

Protocol waivers or exemptions are not allowed with the exception of immediate safety concerns that may arise after the oral administration of CAB.

Deviations from inclusion and exclusion criteria are not allowed because they can potentially jeopardize the scientific integrity of the study, regulatory acceptability or participant safety. Therefore, adherence to the criteria as specified in the protocol is essential

#### 10.1.1. Exclusions from Per Protocol Population

Not applicable. Per protocol population is not defined in this study.

## 10.2. Appendix 2: Time & Events

## 10.2.1. Protocol Defined Time & Events

## Table 21 Schedule of Activities<sup>q</sup>

| | e, | Oral<br>Phase <sup>m</sup> | | Injection Phase | | | | | | | | | | | | | Follow- |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Clinical Assessments | Screening <sup>a</sup> | | | | | | | | | | | | | | | | up |
| | ree | | | | | | | | | | | | | | | | Phase<br>& Final |
| | Sc | | | | | | | | | | | | | | | | Visit |
| | | | 4 | 5) | | | | | | | | | | | | | |
| | | | (Week 4) | (Week 5)<br>n 1 | (Week 6) | | | | | | | | | | | 5, 77 | |
| | | | We | We<br>1 | We | 2 | | $\omega$ | | 4 | | 5 | | | | , 65, | |
| | | | 28 ( | 5 (<br>ion | 15 ( | ion | 10 | 17<br>ion | 18 | . 25<br>ion | 26 | 33<br>ion | 34 | 37 | 41 | 53 | 8 |
| | | Day 1 | Day 2 | Day 35 (W<br>Injection 1 | Day 42 | Week 9<br>Injection | Week 10 | Week 17<br>Injection | Week 18 | Week 25<br>Injection | Week 26 | Week 33<br>Injection | Week 34 | Week 37 | Week 41 | Week 53, | Week |
| | | Ds | Ŋį | Dê<br>Inj | Ďį | W<br>Inj | W | W | $\otimes$ | W<br>Inj | W | W<br>Inj | ≱ | $\otimes$ | $\otimes$ | $\otimes$ | $\geqslant$ |
| Written informed consent | X | | | | | | | | | | | | | | | | |
| Inclusion/Exclusion criteria <sup>b</sup> | X | | | | | | | | | | | | | | | | |
| Demographic information | X | | | | | | | | | | | | | | | | |
| Full physical exam/medical | X | | | | | | | | | | | | | | | | X |
| history <sup>c</sup> | Λ | | | | | | | | | | | | | | | | Λ |
| Brief physical exam | | X | X | X | X | X | X | X | X | X | X | X | X | | X | | |
| Height/weight/BMI <sup>d</sup> | X | | | | | | | | | | | | | | | | X |
| Medication/drug/alcohol history | X | | | | | | | | | | | | | | | | |
| HIV counseling | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Offer condoms and lubricant | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Dispense oral study medication | | X | | | | | | | | | | | | | | | |
| (with counseling) <sup>e</sup> | | | | | | | | | | | | | | | | | |
| Drug accountability (pill counts) | | X | X | | | | | | | | | | | | | | |

| Clinical Assessments | Screening <sup>a</sup> | | ral<br>use <sup>m</sup> | | Injection Phase | | | | | | | | | Foll<br>u<br>Pha | p<br>ase | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Scr | | | | | | | | | | | | | | | | |
| | | | (Week 4) | Day 35 (Week 5)<br>Injection 1 | Day 42 (Week 6) | | | | | | | | | | | 5, 77 | |
| | | | 8 (W | 5 (Wo | 2 (W | 9<br>on 2 | 10 | 17<br>on 3 | 18 | 25<br>on 4 | 26 | 33<br>on 5 | 34 | 37 | 41 | 53, 6 | 68 |
| | | Day 1 | Day 28 | Day 35 (W<br>Injection 1 | )ay 4 | Week 9<br>Injection | Week 10 | Week 17<br>Injection | Week 18 | Week 25<br>Injection | Week 26 | Week 33<br>Injection | Week 34 | Week 37 | Week 41 | Week 53, 65, | Week |
| CAB LA Injection (with counseling) | | Ι | I | X | П | X | | X | | X | | X | | | | | |
| HIV-PrevTSQc <sup>f</sup> | | | | | | | X | | | | | | | | | | |
| ISR AE Diary <sup>g</sup> | | | | X | | X | | X | | X | | X | | | | | |
| AE | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| SAE review (SAE will be collected from the signing of ICF) | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant medication check | | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Vital signs <sup>h</sup> | X | X | | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Qualitative HIV RNA by NAAT <sup>i</sup> | X | | | | | | | | | | | | | | | | |
| HIV PoC test <sup>j</sup> | X | X | | X | | X | | X | | X | | X | | | X | X | X |
| ECG <sup>k</sup> | X | | | | | | | | | | | | | | | | |
| HbsAg and HbsAb, HCV | X | | | | | | | | | | | | | | | | |
| Antibody | | | | | | | | | | | | | | | | | |
| Hematology/Chemistry testing | X | X | X | X | X | X | | X | | X | | X | | | X | | X |
| Urinalysis | X | | | | | | | | | | | | | | X | | |
| Urine screen for Chlamydia and gonorrhea | X | | | | | | | | | | | | | | | | |
| Liver Chemistry Tests <sup>1</sup> | | | | | | | | | | | | | | | | X | |
| | $\mathfrak{S}_a$ | | ral | | | | | Inje | ction | Phase | | | | | | | ow- |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Clinical Assessments | Screening <sup>a</sup> | Phase <sup>m</sup> | | | | | | | | up<br>Phase<br>& Final | | | | | | | |
| | Sc | | | | | | | | | | | | | | | | sit |
| | | Day 1 | Day 28 (Week 4) | Day 35 (Week 5)<br>Injection 1 | Day 42 (Week 6) | Week 9<br>Injection 2 | Week 10 | Week 17<br>Injection 3 | Week 18 | Week 25<br>Injection 4 | Week 26 | Week 33<br>Injection 5 | Week 34 | Week 37 | Week 41 | Week 53, 65, 77 | Week 89 |
| Fasting lipid profile | | X | | | | | | | | | | | | | X | | |
| Coagulation testing | X | | | | | | | | | | | | | | X | | |
| TRUST for Syphilis screen | X | | | | | | | | | | | | | | | | |
| Plasma for CAB concentration <sup>m,n,o</sup> | | | Xm | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Plasma storage sample <sup>p</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |

AE: Adverse events, BMI: Body mass index, CAB: Cabotegravir, CAB LA: Cabotegravir long-acting, ECG: Electrocardiogram, HbsAg: Hepatitis B surface antigen, HIV: Human Immunodeficiency Virus, HCV: Hepatitis C Virus, ISR: Injection site reactions, SAE: Serious adverse event, HIV-PrevTSQc: HIV-Prevention Treatment Satisfaction Questionnaire (change): TRUST: Toluidine Red Unheated Serum Test, RNA: Ribonucleic acid.

- a. Screening (including drug screen) is to be performed within 30 days of the first dose in the Oral Phase of the study. See Appendix 2 from the study protocol
- b. Inclusion/exclusion criteria will be fully assessed at the Screening visit. Changes between the screening visit and the Day 1 visit should be assessed to ensure eligibility, including additional assessments performed at Day 1.
- c. A full physical exam will be performed at Week 89.
- d. Weight will be collected at Screening and at Week 89. Height and BMI will be collected at Screening only.
- e. Oral phase consists of 28 days with a 7 day washout period between Day 28 (last oral dose) and Day 35 (first injection visit).
- f. HIV-PrevTSQc: HIV-Prevention Treatment Satisfaction Questionnaire (change) will be given at Week 10 only (after 2<sup>nd</sup> injection).
- g. ISR AE 7 Day Post Injection Diary will be distributed at the injection visit at Week 5, 9, 17, 25 and 33 and returned to the clinic at weeks 6, 10, 18, 26, and 34. For participants having ISR on the last day of week 5, 9, 17, 25 and 33, additional ISR AE Weeks 2 12 Post Injection Diary will be distributed at weeks 6,10, 18, and 26,34. Participants will be asked to bring the diary to each clinic visit.
- h. Vital sign measurements will be performed following 5 minutes of rest.
- i. Qualitative HIV Nucleic Acid Amplification Testing (NAAT) will be performed at Screening. See Appendix 9 from the study protocol for the HIV testing algorithm at screening, Day 1 and during the course of the study.

- j. HIV PoC (Point of care) test will be performed at each time point during the course of the study and must be reviewed prior to IM dosing. See Appendix 9 from the study protocol for the HIV testing algorithm at screening, Day 1 and during the course of the study.
- k. ECGs will be performed following 5 minutes of rest in a semi-supine position.
- I. Liver Chemistry Tests include Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), Bilirubin total and direct.
- m. Oral Pharmacokinetic (PK) sampling at trough will be collected for all subjects prior to dose within 20 to 28 hours following oral administration the day prior. Intensive oral PK sampling will be collected from approximately16 participants as shown in Table 20.
- n. PK sampling for Injection phase: All PK samples will be collected prior to CAB LA injections at Week 5, 9, 17, 25, and 33 with the exception of 1-week post injection samples at Weeks 6, 10, 18, 26, 34, 37 (2-week post injection sample) and Week 41
- o. Long-term follow up PK samples: PK sampling during follow up will occur at, Week 53, 65, 77, and 89.
- p. Additional testing is required for participants who have a reactive or positive HIV test after enrolment. Stored plasma from the visit previous to the positive test should be tested for HIV using the 4th generation HIV test to best estimate time of infection. HIV acquisition must be confirmed by either western blot, HIV ½ Multispot or the Geenius HIV Confirmation ½ Assay, and HIV RNA.
- q. Visit may occur in a window ±3 Day

Table 22 Schedule of Intensive Oral PK (Approximately 16 Participants) a,b

| | Day 25 | Day 26 | Day 27 | | | | | | Day 28 | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | Oral dose<br>administered<br>(e.g. 8AM) | | 1-<br>hour post<br>dose (e.g.<br>9AM) | post dose<br>(e.g. | post dose<br>(e.g. | post dose<br>(e.g.<br>12AM) | post<br>dose | hour post | Oral dose<br>administered<br>(e.g. after 8 AM) |
| Plasma for CAB concentration | | | X | X | X | X | X | X | X | |

- **a.** PK sampling may occur  $\pm$  15min
- **b.** Central lab tests for the intensive oral PK subjects refer to Table 21.

# 10.3. Appendix 3: Assessment Windows

### 10.3.1. Assessment Windows

The nominal visit information collected on CRF will be used in the analysis. Analysis visit based on the time window will not be defined in this study.

### 10.4. Appendix 4: Study Phase and State

### 10.4.1. Treatment Phases

Assessments and events will be classified according to the time of occurrence relative to the start date of study treatment.

| Treatment Phase | Definition |
|---|---|
| Screening Phase | Date < Date of first Oral CAB |
| Oral Phase | Date of First Oral CAB <= Date <= Date of First CAB LA Injection -1 day; for subjects who discontinued before receiving CAB LA Injection, the end date of the oral phase is the date of last study visit. |
| Injection Phase | Date of First CAB LA Injection <= Date <= 8 weeks after Last CAB LA Injection |
| Follow-up Phase | Date > 8 weeks after Last CAB LA Injection |

### 10.4.2. Treatment States

Assessments and events will be classified according to time of occurrence relative to the start date of the study treatment.

### 10.4.2.1. Treatment States for AE Data

| Treatment State | Definition |
|---|---|
| Screening Phase | AE Start Date < Date of First Oral CAB |
| On-Oral CAB- | Day 1 ≤ AE Start Date ≤ Date of First CAB LA Injection – 1; |
| Treatment | for subjects who withdraw from oral CAB treatment, Day 1 ≤ AE Start Date ≤ Withdrawal date + 7 days |
| On-CAB LA-<br>treatment | Date of First CAB LA Injection ≤ AE Start Date ≤ Date of Week 41 Visit; for subjects who withdraw from CAB LA injection, Date of First CAB LA Injection ≤ AE Start Date ≤ Date of Last CAB LA Injection + 8 Weeks |
| Post-Treatment | AE Start Date > Date of Last CAB LA Injection + 8 weeks |
| Onset Time Since<br>1st Dose (Days) | If Date of First Oral CAB (or CAB LA injection) >AE Onset Date, duration = AE Onset Date - Treatment Start Date |
| | If Date of First Oral CAB (or CAB LA injection) ≤ AE Onset Date, duration = AE Onset Date - Treatment Start Date +1 |
| | Missing otherwise. |
| AE Duration (Days) | AE Resolution Date – AE Onset Date + 1 |
| Drug-related | If relationship is marked 'YES' on CRF OR value is missing |

# 10.5. Appendix 5: Data Display Standards & Handling Conventions

### 10.5.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | |
|---|---|---|---|
| | Study Group Data Displays for Reporting | | |
| Code | Description | Description | Order [1] |
| Α | CAB PO 30 mg QD | CAB 30 mg | 1 |
| В | CAB LA IM 600 mg Q8W | CAB LA 600 mg | 2 |

#### NOTES:

#### 10.5.2. Baseline Definition & Derivations

#### 10.5.2.1. Baseline Definitions

The baseline or pre-dose assessment is the last available assessment prior to the time of the first dose unless it is specified otherwise.

### 10.5.2.2. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|---|---|
| Change from Baseline | = Post-Dose Visit Value – Baseline |
| % Change from Baseline | = 100 x [(Post-Dose Visit Value – Baseline) / Baseline] |
| Maximum Change from Baseline | = Calculate the change from baseline at each given timepoint and determine the maximum change |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 10.5.2.1 Baseline Definitions will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.
- The baseline definition will be footnoted on all change from baseline displays.

### 10.5.3. Reporting Process & Standards

### Reporting Process

#### Software

 The currently supported versions of SAS software 9.2 or higher and Phoenix WinNonlin will be used.

### **Analysis Datasets**

- Analysis datasets will be created according to CDISC standards SDTMIG v3.2 & ADaMIG v1.0
- For creation of ADaM datasets (ADCM/ADAE), the same version of dictionary datasets will be implemented for conversion from SI to SDTM.

<sup>1.</sup> Order represents treatments being presented in TFL, as appropriate.

### **Reporting Process**

#### **Generation of RTF Files**

RTF files will be generated for the TLFs. But only compiled PDF file will be used in the delivery.

### **Reporting Standards**

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - 4.03 to 4.23: General Principles
  - 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the actual treatment the subject received unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses :
  - Nominal visits collected on the eCRF will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in Pharmacokinetic listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.
  - Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings but omitted from figures, summaries and statistical analyses.

### **Unscheduled Visits**

Summary Statistics

- Unscheduled visits will not be included in summary tables.
- Unscheduled visits will not be included in figures.
- All unscheduled visits will be included in listings.

| | | | | O4 41 41 |
|----|--------|--------|---------|------------|
| 11 | Decrin | tiva 🦠 | iimmarv | Statistics |

| Continuous Data | Refer to IDSL Statistical Principle 6.06.1 |
|---|---|
| Categorical Data | N, n, frequency, % |
| Reporting of Pharm | armacokinetic Concentration Data |
| Descriptive | Refer to IDSL Statistical Principle 6.06.1 |

Assign zero to NQ values (Refer to GUI\_51487 for further details)

### **Reporting Standards**

### **Reporting of Pharmacokinetic Parameters**

- Reporting for PK tables, figures and listings:
  - Planned time relative to dosing will be used in mean concentration-time figures and summaries, and actual times will be used for individual concentration-time figures.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
  - Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in all PK figures, summaries and listings.

| | <u> </u> |
|---|---|
| Descriptive | N, n, geometric mean, 95% CI of geometric mean, standard deviation (SD) |
| Summary Statistics | of logged data and [between and or within] geometric coefficient of variation |
| (Log Transformed) | (CV <sub>b</sub> (%)) will be reported. |
| | $CV_b$ (%) = $\sqrt{(exp(SD^2) - 1) * 100}$ |
| | (SD = SD of log transformed data) |
| Parameters Not | tmax, first point, last point, and number of points used in the determination of |
| Being Log | λz. |
| Transformed | |
| Summary Tables | The following PK parameters will not be summarised: first point, last point, and number of points used in the determination of λz |
| Listings | Additionally, include the first point, last point and number of points used in |
| | the determination of lambda_z for listings. |
| Granhical Displays | |

### Graphical Displays

Refer to IDSL Statistical Principals 7.01 to 7.13.

### 10.6. Appendix 6: Derived and Transformed Data

### 10.6.1. **General**

### **Multiple Measurements at One Time Point**

- If there are two values within a time window the value closest to the target day for that window will be used. If values are the same distance from the target then the mean will be taken.
- Subjects having both High and Low values for Normal Ranges at any post-baseline visits for safety parameters will be counted in both the High and Low categories of "Any visit postbaseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

### **Study Day**

- Calculated as the number of days from Day 1 Visit:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < Date of Day 1 Visit → Study Day = Ref Date -Date of Day 1 Visit
  - Ref Date ≥ Date of Day 1 Visit → Study Day = Ref Date –Date of Day 1 Visit + 1

### 10.6.2. Study Population

### **Demographics**

### Age

- As the month and date of birth will not be collected in the study, the age will be calculated as Year of ICF – Year of Birth;
- Birth date will be presented in listings as 'YYYY'.

#### **Body Mass Index (BMI)**

• Calculated as Weight (kg) / [Height (m)<sup>2</sup>]

### **Extent of Exposure**

- Duration of exposure to study drug will be calculated based on the formula:
  - The duration of exposure for oral phase is defined as the number of days starting from the first oral dose to the last oral dose.
  - Duration of exposure for injection phase is defined as the number of injections (1, 2, 3, 4 or 5)
  - Overall exposure to CAB is defined as number of days from the first oral dose to 8 weeks following the participant's last injection. If a participant does not enter the injection phase, the overall CAB exposure for the study will be defined as the number of days from the first oral dose to the last oral dose.
  - Overall exposure to the study (for safety evaluation) is defined as number of days from the first dose to last visit (including unscheduled visit) in days.
- The cumulative dose will be based on the formula:
  - Cumulative dose in oral phase is defined as (number of tablets dispensed number of tablets returned) \* 30 mg

### **Extent of Exposure**

Cumulative dose in injection phase is defined as number of injections \* 600 mg

### 10.6.3. Safety

### **Adverse Events**

### **Adverse Events of Special Interest**

- Seizures and seizure like events
- Decline in Renal Function
- Proximal Renal Tubule Dysfunctions
- Proteinuria
- Hepatoxicity
- Hypersensitivity Reactions
- Injection Site Reactions
- Impact on Creatinine
- Neuropsychiatirc Events

The adverse events of special interest that were used for data summaries are provided in Section 10.16

### **Laboratory Parameters**

- HIV-1 RNA: For summaries and analyses which use HIV-1 RNA level as a continuous measure, the logarithm to base 10 of the value will be used.
- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - $\circ$  Example 1: 2 Significant Digits = '< x' becomes x 0.01
  - Example 2: 1 Significant Digit = '> x' becomes x + 0.1
  - Example 3: 0 Significant Digits = '< x' becomes x 1

# 10.7. Appendix 7: Premature Withdrawals & Handling of Missing Data

### 10.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | Subject study completion (i.e. as specified in the protocol) was defined as completing all phases of the study including week 89. |
| | <ul> <li>If participants prematurely discontinue the oral phase of the study, additional replacement participants may be recruited at the discretion of the Sponsor. Participants who enter the injection phase of the study will not be replaced</li> <li>All available data from subjects who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

### 10.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument:</li> <li>These data will be indicated using a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table. </li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to<br/>be missing data and should be displayed as such.</li> </ul> |
| | <ul> <li>Missing endpoints which are not covered in the following rule will not be imputed,<br/>unless otherwise specified.</li> </ul> |
| Outliers | Any subjects excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

### 10.7.2.1. Handling of Missing Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| Adverse<br>Events | <ul> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> <li>Partial missing start or end dates will be imputed using the convention specified in Section 10.7.2.2 Handling of Partial Dates</li> </ul> |

## 10.7.2.2. Handling of Partial Dates

| Element | Reporting Detail |
|---|---|
| Concomitant | Partial dates for any concomitant medications recorded in the CRF will be |

| Element | Reporting Detail |
|---|---|
| Medications | <ul> <li>imputed using the following convention:</li> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> <li>The recorded partial date will be displayed in listings.</li> </ul> |
| Adverse<br>Events | <ul> <li>Any partial dates for adverse events will be raised to data management. If the full date cannot be ascertained, the following assumptions will be made: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month.</li> <li>However, if these results in a date prior to Week 1 Day 1 and the event could possibly have occurred during treatment from the partial information, then the Week 1 Day 1 date will be assumed to be the start date. The AE will then be considered to start on-treatment (worst case).</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

## 10.7.2.3. Handling of Missing Data for Statistical Analysis

| Element | Reporting Detail |
|---------|-----------------------------------------------------------------|
| N/A | No statistical analysis is planned, unless otherwise specified. |

# 10.8. Appendix 8: Values of Potential Clinical Importance

### 10.8.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| | | Male | | 0.54 |
| Hematocrit | Ratio of 1 | Female | | 0.54 |
| | | $\Delta$ from BL | ↓0.075 | |
| | g/L | Male | | 180 |
| Hemoglobin | | Female | | 180 |
| | | $\Delta$ from BL | <b>↓25</b> | |
| Lymphocytes | x109/ L | | 8.0 | |
| Neutrophil Count | x109/ L | | 1.5 | |
| Platelet Count | x109/ L | | 100 | 550 |
| While Blood Cell Count (WBC) | x10 <sup>9</sup> / L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | g/L | | 30 | |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | umol/L | $\Delta$ from BL | | ↑ 44.2 |
| Glucose | mmol/L | | 3 | 9 |
| Phosphorus | mmol/L | | 0.8 | 1.6 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |
| Total CO2 | mmol/L | | 18 | 32 |

| Liver Function | | | |
|--------------------|--------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | µmol/L | High | ≥ 1.5xULN |
| | µmol/L | | 1.5xULN T. Bilirubin |
| T. Bilirubin + ALT | | High | + |
| | U/L | | ≥ 2x ULN ALT |

### 10.8.2. ECG

| ECG Parameter | Units | Clinical Concern Range | |
|---|---|---|---|
| | | Lower | Upper |
| Absolute | | | |
| | | > 450 [1] | |
| Abaqluta OTa Intonval | mana | > 450 [1] | ≤ 479 <sup>[1]</sup> |
| Absolute QTc Interval | msec | ≥ 480 [1] | ≤ 499 <sup>[1]</sup> |
| | | ≥ 500 <sup>[1]</sup> | |
| Absolute PR Interval | msec | < 110 <sup>[1]</sup> | > 220 [1] |
| Absolute QRS Interval | msec | < 75 [1] | > 110 [1] |
| Change from Baseline | | | |
| | msec | > 60 [1] | |
| Increase from Baseline QTc | msec | > 30 [1] | ≤ 59 <sup>[1]</sup> |
| | msec | ≥ 60 <sup>[1]</sup> | |

**NOTES:** [Remove footnotes for RAP development]

- 1. Represent standard ECG values of PCI for HV studies
- 2. Represent further subdivisions of ECG values for analysis whereby the RAP team needs to decide whether these need to be generated in addition to standard ECG values being flagged. IF not required, then delete.

### 10.8.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |

| Vital Sign Parameter | Units Clinical Concern Range | | | | |
|---|---|---|---|---|---|
| (Change from Baseline) | | Decrease | | Increase | |
| | | Lower | Upper | Lower | Upper |
| Systolic Blood Pressure | mmHg | ≥ 20 | ≥ 40 | ≥ 20 | ≥ 40 |
| Diastolic Blood Pressure | mmHg | ≥ 10 | ≥ 20 | ≥ 10 | ≥ 20 |
| Heart Rate | bpm | ≥ 15 | ≥ 30 | ≥ 15 | ≥ 30 |

**NOTES:** [Remove footnotes for RAP development]

Represent further subdivisions of BP & HR for analysis whereby the RAP team needs to decide whether these need to be generated in addition to standard absolute BP & HR values being flagged. IF not required, then delete.

## 10.9. Appendix 9: Multicenter Studies

### 10.9.1. Methods for Handling Centres

• In this multicentre study, enrolment will be presented by investigative site.

# 10.10. Appendix 10: Examination of Covariates, Subgroups & Other Strata

### 10.10.1. Handling of Covariates, Subgroups & Other Strata

- Demographic covariates that may be used in descriptive summaries and statistical analyses, some of which may also be used for subgroup analyses.
- Additional covariates of clinical interest may also be considered.

## 10.11. Appendix 11: Multiple Comparisons & Multiplicity

### 10.11.1. Handling of Multiple Comparisons & Multiplicity

Not applicable.

# 10.12. Appendix 12: Model Checking and Diagnostics for Statistical Analyses

### 10.12.1. Statistical Analysis Assumptions

| Endpoint(s) | • | PK endpoint $C_{\tau}$ |
|-------------|---|------------------------|
| Analysis | • | ANOVA (primary) |

- Model assumptions will be applied, but appropriate adjustments maybe made based on the data.
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.

## 10.13. Appendix 13: Abbreviations & Trade Marks

### 10.13.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AUC(0-τ) | Area under the concentration-time curve (AUC) over the dosing interval |
| Сτ | The observed concentration at the end of the dosing interval |
| CAB | Cabotegravir |
| CAB LA | Cabotegravir Long Acting |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CL/F | The apparent clearance (adjusted for bioavailability, F) |
| Cmax | Maximum observed concentration |
| CSR | Clinical Study Report |
| CTMS | Clinical Trial Management System |
| $CV_b$ | Coefficient of Variation (Between) |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| GSK | GlaxoSmithKline |
| HIV | Human Immunodeficiency Virus |
| ICH | International Conference on Harmonisation |
| IDSL | Integrated Data Standards Library |
| IM | Intramuscular |
| IP | Investigational Product |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mg | Milligrams |
| PCI | Potential Clinical Importance |
| PK | Pharmacokinetic |
| PrEP | Pre-exposure prophylaxis |
| QC | Quality Control |
| RAP | Reporting & Analysis Plan |
| SAC | Statistical Analysis Complete |
| SAS | Statistical Analysis Software |
| SD | Standard deviation |
| SDTM | Study Data Tabulation Model |
| SOP | Standard Operation Procedure |
| t½ | Terminal phase half-life |
| tmax | Time to first occurrence of Cmax |
| TFL | Tables, Figures & Listings |
| Vz/F | The volume of distribution associated with the terminal phase (adjusted |
| | for bioavailability, F) |
| λz | Terminal-phase rate constant |

## 10.13.2. Trademarks

| Trademarks of the GlaxoSmithKline |
|-----------------------------------|
| Group of Companies |

NONE

# Trademarks not owned by the GlaxoSmithKline Group of Companies

Phoenix WinNonlin

SAS

### 10.14. Appendix 14: List of Data Displays

### 10.14.1. Data Display Numbering

The following numbering will be applied for RAP generated display according to ICH standards:

| Section | Tables | Figures |
|------------------|-------------|---------|
| Study Population | 1.1 to 1.10 | NA |
| Safety | 2.1 to 2.32 | NA |
| Pharmacokinetic | 3.1 to 3.11 | 3.1-3.8 |
| Section | Listings | |
| ICH Listings | 1-51 | |

### 10.14.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required an example mock-up displays provided in Appendix 15: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |

### NOTES:

 Non-Standard displays are indicated in the 'IDSL / TST ID / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

### 10.14.3. Deliverable [Priority]

| Delivery [Priority] [1] | Description |
|-------------------------|--------------------------------------------------|
| W41 SAC [1] | Primary Statistical Analysis Complete at Week 41 |
| SAC [1] | Final Statistical Analysis Complete at Week 89 |

#### NOTES:

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort.

# 10.14.4. Study Population Tables

| Study Pop | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| Study Po | Study Population, Disposition and Demographics | | | | |
| 1.1 | Screened | SP1 | Summary of Study Population | | W41 SAC [1],<br>SAC [1] |
| 1.2 | Screened | ES6 | Summary of Screen Status and Reasons for Screen Failures | | W41 SAC [1],<br>SAC [1] |
| 1.3 | Screened | ES1 | Summary of Subject Disposition for the Subject Conclusion Record | | W41 SAC [1], SAC [1] |
| 1.4 | Safety | SD1 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment | | W41 SAC [1], SAC [1] |
| 1.5 | Safety | DM1 | Summary of Demographic Characteristics | | W41 SAC [1], SAC [1] |
| Medical H | listory and Cond | omitant Medications | | | |
| 1.6 | Safety | MH4 | Summary of Medical Conditions | | W41 SAC [1], SAC [1] |
| 1.7 | Safety | CM1 | Summary of Prior Medications | | W41 SAC [1], SAC [1] |
| 1.8 | Safety | CM1 | Summary of Concomitant Medications | | W41 SAC [1], SAC [1] |
| Protocol | Protocol Deviations | | | | |
| 1.9 | Safety | IE1 | Summary of Inclusion/Exclusion Criteria Deviations | | W41 SAC [1], SAC [1] |
| 1.10 | Safety | DV1A | Summary of Important Protocol Deviations | | W41 SAC [1], SAC [1] |

# 10.14.5. Safety Tables

| | | | Safety: Tables | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| Exposure | • | • | | | |
| 2.1 | Safety | EX1 | Summary of Extent of Exposure | | W41 SAC [1],<br>SAC [1] |
| Injection S | Site Reactions | | | , | |
| 2.2 | Safety<br>Injection | | Summary of Injection Site Reaction | | W41 SAC [1],<br>SAC [1] |
| Adverse E | vents | • | | | |
| 2.3 | Safety | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term | | W41 SAC [1], SAC [1] |
| 2.4 | Safety | AE5B | Summary of All Adverse Events by Maximum Grade by System Organ Class and Preferred Term | | W41 SAC [1], SAC [1] |
| 2.5 | Safety | AE3 | Summary of All Grade 2 or Higher Adverse Events by Overall Frequency | | W41 SAC [1], SAC [1] |
| 2.6 | Safety | AE3 | Summary of Serious Adverse Events | | W41 SAC [1], SAC [1] |
| 2.7 | Safety | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term (Number of Subjects and Occurrences) | | W41 SAC [1], SAC [1] |
| 2.8 | Safety | AE3 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Drug or Withdrawal from Study | | W41 SAC [1], SAC [1] |
| 2.9 | Safety | AE1 | Summary of Drug-Related Adverse Events | | W41 SAC [1], SAC [1] |
| 2.10 | Safety | AE1 | Summary of Drug-Related Serious Adverse Events | | W41 SAC [1], SAC [1] |

| | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| 2.11 | Safety | AE3 | Summary of Drug-related Grade 2 or Higher Adverse Events | | W41 SAC [1], SAC [1] |
| 2.12 | Safety | AE3 | Summary of Common (>=5%) Adverse Events by Overall Frequency | | W41 SAC [1], SAC [1] |
| 2.13 | Safety | AE15 | Summary of Common (>=5%) Non-Serious Adverse<br>Events by System Organ Class and Preferred Term<br>(Number of Subjects and Occurrences) | | W41 SAC [1], SAC [1] |
| 2.14 | Safety | AE3 | Summary of Common (>=5%) Grade 2-4 Adverse Events by Overall Frequency | | W41 SAC [1], SAC [1] |
| 2.15 | Safety | AE3 | Summary of Common (>=5%) Drug-Related Grade 2-4<br>Adverse Events by Overall Frequency | | W41 SAC [1], SAC [1] |
| Laborator | y Tests | | | | |
| 2.16 | Safety | | Summary of Grade 2 or Higher Laboratory Tests | | W41 SAC [1], SAC [1] |
| 2.17 | Safety | ES11 | Summary of Characteristics of Adverse Events of Special Interest | | W41 SAC [1], SAC [1] |
| 2.18 | Safety | LB1 | Summary of Change from Baseline in Hematology and Coagulation Data | | W41 SAC [1], SAC [1] |
| 2.19 | Safety | LB1 | Summary of Change from Baseline in Chemistry Data and Fasting Lipid Profile | | W41 SAC [1], SAC [1] |
| 2.20 | Safety | UR3 | Summary of Urinalysis and Urine Chemistry Results | | W41 SAC [1], SAC [1] |
| 2.21 | Safety | LB18 | Summary of Hematology and Coagulation Grade Shifts from Baseline Grade | | W41 SAC [1], SAC [1] |
| 2.22 | Safety | LB18 | Summary of Chemistry and Fasting Lipid Profile Grade Shifts from Baseline Grade | | W41 SAC [1], SAC [1] |

| | Safety: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| 2.23 | Safety | LB18 | Summary of Urinalysis Grade Shifts from Baseline Grade | | W41 SAC [1], SAC [1] |
| Vital Signs | | | | | |
| 2.24 | Safety | VS1 | Summary of Change from Baseline in Vital Signs | | W41 SAC [1], SAC [1] |
| 2.25 | Safety | VS8 | Summary of Vital Sign Shifts from Baseline with Respect to Clinical Concern Range | | W41 SAC [1], SAC [1] |
| Liver Event | Liver Events | | | | |
| 2.26 | Safety | LIVER1 | Summary of Liver Events Reporting | | W41 SAC [1], SAC [1] |
| 2.27 | Safety | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities | | W41 SAC [1], SAC [1] |

# 10.14.6. Tolerability Tables

| | Tolerability: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Tolerability | Tolerability of CAB Injection | | | | |
| 2.28 | Safety<br>Injection | | Summary of HIV-Prevention Treatment Satisfaction Scores | | W41 SAC [1],<br>SAC [1] |

## 10.14.7. Acceptability Tables

| | Acceptability: Tables | | |
|---|---|---|---|
| NO I PODILIZION I I I I I I I I I I I I I I I I I I | | | Deliverable<br>[Priority] |
| | Acceptability of the CAB Injection | | |
| 2.29 | Safety | Summary of Acceptability of the CAB LA | W41 SAC [1],<br>SAC [1] |

### 10.14.8. Pharmacokinetic Tables

| Pharma | Pharmacokinetic : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Oral Pha | ase | | | | |
| 3.1 | Oral PK | PKCT1 | Summary of CAB Plasma Pharmacokinetic Concentration-<br>Time Data – Oral Phase | | SAC [1] |
| 3.2 | Oral PK | PKPT4 | Summary of Derived CAB Plasma Pharmacokinetic Parameters (Non-Transformed) – Oral Phase | Parameters with units | SAC [1] |
| 3.3 | Oral PK | PKPT4 | Summary of Derived CAB Plasma Pharmacokinetic Parameters (Log-Transformed) – Oral Phase | Parameters with units | SAC [1] |
| Injection | n Phase (up to Week | ( 41) | | | |
| 3.4 | Injection<br>(Week 41) PK | PKCT1 | Summary of CAB Plasma Pharmacokinetic Concentration-<br>Time Data – Injection Phase (up to Week 41) | | W41 SAC [1],<br>SAC [1] |
| 3.5 | Injection<br>(Week 41) PK | PKPT4 | Summary of Derived CAB Plasma Pharmacokinetic<br>Parameters (Non-Transformed) – Injection Phase (up to<br>Week 41) | Parameters with units | W41 SAC [1],<br>SAC [1] |
| 3.6 | Injection<br>(Week 41) PK | PKPT4 | Summary of Derived CAB Plasma Pharmacokinetic<br>Parameters (Log-Transformed) – Injection Phase (up to<br>Week 41) | Parameters with units | W41 SAC [1]<br>SAC [1] |
| 3.7 | Injection<br>(Week 41) PK | PKPT3 | Statistical Analysis of CAB Plasma Accumulation – Injection Phase (up to Week 41) | Cτ only for Injection<br>Phase at Week 41. | W41 SAC [1],<br>SAC [1] |
| 3.8 | Injection<br>(Week 41) PK | PKPT3 | Statistical Analysis of CAB Plasma Steady-state Pre-dose Concentrations – Injection Phase (up to Week 41) | Cτ only for Injection<br>Phase at Week 41. | W41 SAC [1],<br>SAC [1] |

| Pharma | Pharmacokinetic : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Injection | n Phase (up to Week | 89) | | | |
| 3.9 | Injection<br>(Week 89) PK | PKCT1 | Summary of CAB Plasma Pharmacokinetic Concentration-<br>Time Data – Injection Phase (up to Week 89) | | SAC [1] |
| 3.10 | Injection<br>(Week 89) PK | PKPT4 | Summary of Derived CAB Plasma Pharmacokinetic<br>Parameters (Non-Transformed) – Injection Phase (up to<br>Week 89) | Parameters with units | SAC [1] |
| 3.11 | Injection<br>(Week 89) PK | PKPT4 | Summary of Derived CAB Plasma Pharmacokinetic<br>Parameters (Log-Transformed) – Injection Phase (up to<br>Week 89) | Parameters with units | SAC [1] |

# 10.14.9. Pharmacokinetic Figures

| Pharm | Pharmacokinetic : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| Oral Pl | hase | | | | • |
| 3.1 | Oral PK | PKCF1P | Individual CAB Plasma Concentration-Time Plots (Linear and Semi-Logarithmic) – Oral Phase | | SAC [1] |
| 3.2 | Oral PK | PKCF4 | Mean (±SD) CAB Plasma Concentration-Time Plots (Linear and Semi-Logarithmic) – Oral Phase | | SAC [1] |
| Injection | on Phase (up to Wee | k 41) | | | |
| 3.3 | Injection<br>(Week 41) PK | PKCF1P | Individual CAB Plasma Concentration-Time Plots (Linear and Semi-Logarithmic) – Injection Phase (up to Week 41) | | W41 SAC [1],<br>SAC [1] |
| 3.4 | Injection<br>(Week 41) PK | PKCF4 | Mean (±SD) CAB Plasma Concentration-Time Plots (Linear and Semi-Logarithmic) – Injection Phase (up to Week 41) | | W41 SAC [1],<br>SAC [1] |
| 3.5 | Injection<br>(Week 41) PK | PK26 | Individual CAB Plasma Pre-dose Concentration versus Week (Linear and Semi-Logarithmic) – Injection Phase (up to Week 41) | | W41 SAC [1],<br>SAC [1] |
| 3.6 | Injection<br>(Week 41) PK | PK27 | Median (range) CAB Plasma Pre-dose Concentration versus Week (Linear and Semi log) – Injection Phase (up to Week 41) | | W41 SAC [1],<br>SAC [1] |
| Injection | on Phase (up to Wee | k 89) | | | • |
| 3.7 | Injection<br>(Week 89) PK | PKCF1P | Individual CAB Plasma Concentration-Time Plots (Linear and Semi-Logarithmic) – Injection Phase (up to Week 89) | | SAC [1] |
| 3.8 | Injection<br>(Week 89) PK | PKCF4 | Mean (±SD) CAB Plasma Concentration-Time Plots (Linear and Semi-Logarithmic) – Injection Phase (up to Week 89) | | SAC [1] |

# 10.14.10. ICH Listings

| ICH: List | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Study P | opulation, Disposit | ion and Demogra | phics | | |
| 1 | Screened | SP3 | Listing of Subjects Excluded from Any Population | | W41 SAC [1], SAC [1] |
| 2 | Screened | ES7 | Listing of Reasons for Screen Failure | | W41 SAC [1], SAC [1] |
| 3 | Safety | ES2 | Listing of Reasons for Withdrawal | | W41 SAC [1], SAC [1] |
| 4 | Safety | SD2 | Listing of Study Drug Discontinuation Record | | W41 SAC [1], SAC [1] |
| 5 | Safety | DM2 | Listing of Demographic Characteristics | | W41 SAC [1], SAC [1] |
| 6 | Safety | EX3 | Listing of Exposure Data – Oral Dose | | W41 SAC [1], SAC [1] |
| 7 | Safety | | Listing of Exposure Data – Injection | | W41 SAC [1], SAC [1] |
| Medical | History and Conco | mitant Medication | on | | • |
| 8 | Safety | MH2 | Listing of Medical Conditions | | W41 SAC [1], SAC [1] |
| 9 | Safety | CM5 | Listing of Prior Medications | | W41 SAC [1], SAC [1] |
| 10 | Safety | CM5 | Listing of Concomitant Medications | | W41 SAC [1], SAC [1] |

| ICH: Listi | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Protocol | l Deviations | | | | |
| 11 | Safety | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | W41 SAC [1], SAC [1] |
| 12 | Safety | DV2 | Listing of Important Protocol<br>Deviations | | W41 SAC [1], SAC [1] |
| Injection | Site Reaction | | | | <u> </u> |
| 13 | Safety Injection | | Listing of Injection Site Reaction –<br>Daily Diary Card 1 | | W41 SAC [1],<br>SAC [1] |
| 14 | Safety Injection | | Listing of Injection Site Reaction –<br>Daily Diary Card 2 | | W41 SAC [1],<br>SAC [1] |
| Adverse | Events | | | | - |
| 15 | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | | W41 SAC [1],<br>SAC [1] |
| 16 | Safety | AE8 | Listing of All Adverse Events | | W41 SAC [1], SAC [1] |
| 17 | Safety | AE8CPA | Listing of Serious Adverse Events (Fatal and Non-Fatal) | | W41 SAC [1], SAC [1] |
| 18 | Safety | AE8 | Listing of Grader 2 or Higher Adverse Events | | W41 SAC [1], SAC [1] |
| 19 | Safety | AE8 | Listing of All Adverse Events Leading to Premature Discontinuation of Study Drug or Withdrawal from Study | | W41 SAC [1], SAC [1] |
| 20 | Safety | AE8 | Listing of Adverse Events of Special Interest | | W41 SAC [1], SAC [1] |

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 21 | Safety | | Listing of Possible Suicidality-Rated Adverse Events | | W41 SAC [1], SAC [1] |
| 22 | Safety | AE2 | Listing of Relationship Between<br>System Organ Classes and Verbatim<br>Text | | W41 SAC [1], SAC [1] |
| 23 | Safety | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | | W41 SAC [1], SAC [1] |
| Deaths | | | | | <u>.</u> |
| 24 | Safety | | Listing of Death | | W41 SAC [1], SAC [1] |
| Laborato | ry Tests | | | | |
| 25 | Safety | LB5 | Listing of Chemistry Data and Fasting Lipid Profile | | W41 SAC [1], SAC [1] |
| 26 | Safety | LB5 | Listing of Hematology and Coagulation Data | | W41 SAC [1], SAC [1] |
| 27 | Safety | UR2a | Listing of Urinalysis and Urine<br>Chemistry Data | | W41 SAC [1], SAC [1] |
| 28 | Safety | LB5 | Listing of Laboratory Data for Subjects with Grade 2 or Higher Abnormalities | | W41 SAC [1], SAC [1] |
| 29 | Safety | LB14 | Listing of HIV Tests | | W41 SAC [1], SAC [1] |
| 30 | Safety | LB5 | Listing of Local Lab Data | | W41 SAC [1], SAC [1] |

| ICH: Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Vital Sign | /ital Sign | | | | |
| 31 | Safety | VS4 | Listing of Vital Signs | | W41 SAC [1], SAC [1] |
| 32 | Safety | VS4 | Listing of Vital Signs for Subjects with<br>Any Value of Potential Clinical<br>Importance | | W41 SAC [1], SAC [1] |
| ECG's | | | | | |
| 33 | Safety | | Listing of ECG Results | | W41 SAC [1], SAC [1] |
| Social Harn | Social Harm | | | | |
| 34 | Safety | | Listing of Social Harm | | W41 SAC [1], SAC [1] |
| Cardiovasc | ular Event | | | | • |
| 35 | Safety | | Listing of Cardiovascular Event | | W41 SAC [1], SAC [1] |
| Liver Event | Liver Event | | | | |
| 36 | Safety | | Listing of Liver Event | | W41 SAC [1], SAC [1] |
| Tolerability | Tolerability of CAB Injection | | | | |
| 37 | Safety Injection | | Listing of HIV-Prevention Treatment Satisfaction Questionnaire | | W41 SAC [1], SAC [1] |

| ICH: Listi | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Acceptab | ility of the CAB Inject | ion | | | |
| 38 | Safety | | Listing of Acceptability of the CAB LA | | W41 SAC [1],<br>SAC [1] |
| Pharmace | okinetic | | | | |
| 39 | Oral PK | PKCL1P | Listing of CAB Plasma Pharmacokinetic Concentration-Time Data – Oral Phase | Please list all the concentration data including unscheduled. | SAC [1] |
| 40 | Oral PK | PKPL1P | Listing of Derived CAB Plasma<br>Pharmacokinetic Parameters – Oral<br>Phase | | SAC [1] |
| 41 | Injection<br>(Week 41) PK | PKCL1P | Listing of CAB Plasma Pharmacokinetic Concentration-Time Data – Injection Phase (up to Week 41) | Please list all the concentration data including unscheduled. | W41 SAC [1],<br>SAC [1] |
| 42 | Injection<br>(Week 41) PK | PKPL1P | Listing of Derived CAB Plasma Pharmacokinetic Parameters – Injection Phase (up to Week 41) | | W41 SAC [1],<br>SAC [1] |
| 43 | Injection<br>(Week 89) PK | PKCL1P | Listing of CAB Plasma Pharmacokinetic Concentration-Time Data – Injection Phase (up to Week 89) | Please list all the concentration data including unscheduled. | SAC [1] |
| 44 | Injection<br>(Week 89) PK | PKPL1P | Listing of Derived CAB Plasma Pharmacokinetic Parameters – Injection Phase (up to Week 89) | | SAC [1] |

# 10.14.11. Non-ICH Listings

| Non-ICH: Listings | |
|---|---|
| NO PONIISTION I LITIO I LITIO I PROGRAMMING NOTOS | Deliverable<br>[Priority] |

## 10.15. Appendix 15: Example Mock Shells for Data Displays

Data Display Specification will be made available on Request

# 10.16. Appendix 16: Adverse Events of Special Interest Used for Data Summaries
| AESI Item | Product of Interest | PT Selection* |
|---|---|---|
| Hepatic Safety Profile: Assessment of risk of | CAB +RPV | Sub- SMQ** x2 |
| hepatoxicity | | |
| Hypersensitivity reactions (HSR) | САВ | SMQ (modified) plus selected |
| | | PTs from HLGT |
| Severe cutaneous adverse reactions (SCAR) | RPV | SMQ plus selected PTs from |
| | | HLTs |
| Prolongation of the corrected QT interval of the ECG | RPV | SMQ plus selected PT from HLT |
| in supratherapeutic doses | | |
| Neuropsychiatric Events | CAB +RPV | SMQ , Sub- SMQ or HLGT |
| <ul><li>Suicidal ideation/behaviour</li></ul> | | |
| •Depression | | |
| •Bipolar disorder | | |
| •Psychosis | | |
| •Mood disorders | | |
| •Anxiety | | |
| •Sleep disorders | | |
| Injection Site Reactions (ISR) | CAB +RPV | Use CRF terms for ISRs |
| Seizures and seizure-like events | CAB | SMQ plus selected PTs from |
| | | HLTs |
| Impact on Creatinine/Decline in Renal function | CAB+RPV | SMQ plus selected PTs from HLT |
| Safety in Pregnancy | CAB | Use AE terms co-reported in |
| | | pregnancy exposures to CAB |
| Protenuria | CAB+RPV | SMQ |
| Proximal Renal Tubule Dysfunctions | CAB+RPV | SMQ |

<sup>\*</sup> All PTs, SMQs, HLT, HLGTs from MedDRA V21

<sup>\*\*</sup> All SMQs use narrow terms unless otherwise specified

Hepatic failure, fibrosis and cirrhosis and other liver damage-

Notes: Medical concept of hepatic failure and hepatitis. Sub- SMQs (1) 'Hepatic failure, fibrosis and cirrhosis and other liver damage-related conditions' <u>and</u> (2) 'Hepatitis, non-infectious', both of parent SMQ 'Hepatic Disorders'; only narrow terms selected from sub-SMQs. Some preferred terms e.g PT 'hepatitis fulminant' are duplicated.

| related conditions (SMQ) | | 20000013 |
|--------------------------------------|----------|----------|
| PT | PT Code | |
| Acquired hepatocerebral degeneration | 10080860 | |
| Acute hepatic failure | 10000804 | |
| Acute on chronic liver failure | 10077305 | |
| Acute yellow liver atrophy | 10070815 | |
| Ascites | 10003445 | |
| Asterixis | 10003547 | |
| Bacterascites | 10068547 | |
| Biliary cirrhosis | 10004659 | |
| Biliary fibrosis | 10004664 | |
| Cholestatic liver injury | 10067969 | |
| Chronic hepatic failure | 10057573 | |
| Coma hepatic | 10010075 | |
| Cryptogenic cirrhosis | 10063075 | |
| Diabetic hepatopathy | 10071265 | |
| Drug-induced liver injury | 10072268 | |
| Duodenal varices | 10051010 | |
| Gallbladder varices | 10072319 | |
| Gastric variceal injection | 10076237 | |
| Gastric variceal ligation | 10076238 | |
| Gastric varices | 10051012 | |
| Gastric varices haemorrhage | 10057572 | |
| Hepatectomy | 10061997 | |
| Hepatic atrophy | 10019637 | |
| Hepatic calcification | 10065274 | |
| Hepatic cirrhosis | 10019641 | |
| Hepatic encephalopathy | 10019660 | |
| Hepatic encephalopathy prophylaxis | 10066599 | |
| Hepatic failure | 10019663 | |
| Hepatic fibrosis | 10019668 | |
| Hepatic hydrothorax | 10067365 | |
| Hepatic infiltration eosinophilic | 10064668 | |
| Hepatic lesion | 10061998 | |
| Hepatic necrosis | 10019692 | |
| Hepatic steato-fibrosis | 10077215 | |
| Hepatic steatosis | 10019708 | |
| Hepatitis fulminant | 10019772 | |
| Hepatobiliary disease | 10062000 | |
| Hepatocellular foamy cell syndrome | 10053244 | |
| Hepatocellular injury | 10019837 | |

| РТ | PT Code |
|---------------------------------------|----------|
| Hepatopulmonary syndrome | 10052274 |
| Hepatorenal failure | 10019845 |
| Hepatorenal syndrome | 10019846 |
| Hepatotoxicity | 10019851 |
| Intestinal varices | 10071502 |
| Intestinal varices haemorrhage | 10078058 |
| Liver and small intestine transplant | 10052280 |
| Liver dialysis | 10076640 |
| Liver disorder | 10024670 |
| Liver injury | 10067125 |
| Liver operation | 10062040 |
| Liver transplant | 10024714 |
| Lupoid hepatic cirrhosis | 10025129 |
| Minimal hepatic encephalopathy | 10076204 |
| Mixed liver injury | 10066758 |
| Nodular regenerative hyperplasia | 10051081 |
| Non-alcoholic fatty liver | 10029530 |
| Non-alcoholic steatohepatitis | 10053219 |
| Non-cirrhotic portal hypertension | 10077259 |
| Oedema due to hepatic disease | 10049631 |
| Oesophageal varices haemorrhage | 10030210 |
| Peripancreatic varices | 10073215 |
| Portal fibrosis | 10074726 |
| Portal hypertension | 10036200 |
| Portal hypertensive colopathy | 10079446 |
| Portal hypertensive enteropathy | 10068923 |
| Portal hypertensive gastropathy | 10050897 |
| Portal vein cavernous transformation | 10073979 |
| Portal vein dilatation | 10073209 |
| Portopulmonary hypertension | 10067281 |
| Primary biliary cholangitis | 10080429 |
| Regenerative siderotic hepatic nodule | 10080679 |
| Renal and liver transplant | 10052279 |
| Retrograde portal vein flow | 10067338 |
| Reye's syndrome | 10039012 |
| Reynold's syndrome | 10070953 |
| Splenic varices | 10067823 |
| Splenic varices haemorrhage | 10068662 |
| Steatohepatitis | 10076331 |
| Subacute hepatic failure | 10056956 |
| Varices oesophageal | 10056091 |
| Varicose veins of abdominal wall | 10072284 |
| White nipple sign | 10078438 |

| Hepatitis, non-infectious ( | 20000010 |
|--------------------------------------------|----------|
| PT | PT Code |
| Acute graft versus host disease in liver | 10066263 |
| Allergic hepatitis | 10071198 |
| Alloimmune hepatitis | 10080576 |
| Autoimmune hepatitis | 10003827 |
| Chronic graft versus host disease in liver | 10072160 |
| Chronic hepatitis | 10008909 |
| Graft versus host disease in liver | 10064676 |
| Hepatitis | 10019717 |
| Hepatitis acute | 10019727 |
| Hepatitis cholestatic | 10019754 |
| Hepatitis chronic active | 10019755 |
| Hepatitis chronic persistent | 10019759 |
| Hepatitis fulminant | 10019772 |
| Hepatitis toxic | 10019795 |
| Immune-mediated hepatitis | 10078962 |
| Ischaemic hepatitis | 10023025 |
| Lupus hepatitis | 10067737 |
| Non-alcoholic steatohepatitis | 10053219 |
| Radiation hepatitis | 10051015 |
| Steatohepatitis | 10076331 |

| Drug reaction with eosinophilia and systemic symptoms syndrome (SMQ) - | | 20000225 |
|---|---|---|
| PT | PT Code | |
| Drug reaction with eosinophilia and systemic symptoms | 10073508 | |
| Pseudolymphoma | 10037127 | |

| PTs (Selective) | |
|-----------------------------------|----------|
| Drug hypersensitivity | 10013700 |
| Hypersensitivity | 10020751 |
| Type IV Hypersensitivity reaction | 10053613 |
| Eosinophillia | 10014950 |
| Eye swelling | 10015967 |
| Eyelid oedema | 10015993 |
| Lip swelling | 10024570 |
| Angioedema | 10002424 |
| Circumoral oedema | 10052250 |
| Face oedema | 10016029 |
| Idiopathic angioedema | 10073257 |
| Lip oedema | 10024558 |
| Mouth swelling | 10075203 |
| Oedema mouth | 10030110 |
| Periorbital oedema | 10034545 |
| Swelling face | 10042682 |

Notes: Medical concept of hypersensitivity reactions/DRESS. Only narrow terms selected from Category A of SMQ 'Drug reaction with eosinophilia and systemic symptoms syndrome'. Algorithmic approach for this SMQ not used due to complexity in applying and poor specificity of remaining categories. Category A selected as PTs because more specific for concept (only narrow terms) and a pre-requisite for any combination in algorithmic search. Overlap of some preferred terms with SMQ 'Severe Cutaneous Adverse Reactions'. Plus additional preferred terms selected from HGLT 'Allergic conditions' under SOC 'Immune system disorders'

| Severe cutaneous adverse reactions ( | SMQ) | 20000020 |
|-------------------------------------------------------|----------|----------|
| PT | PT Code | |
| Acute generalised exanthematous pustulosis | 10048799 | |
| Cutaneous vasculitis | 10011686 | |
| Dermatitis bullous | 10012441 | |
| Dermatitis exfoliative | 10012455 | |
| Dermatitis exfoliative generalised | 10012456 | |
| Drug reaction with eosinophilia and systemic symptoms | 10073508 | |
| Epidermal necrosis | 10059284 | |
| Erythema multiforme | 10015218 | |
| Exfoliative rash | 10064579 | |
| Oculomucocutaneous syndrome | 10030081 | |
| Skin necrosis | 10040893 | |
| Stevens-Johnson syndrome | 10042033 | |
| Toxic epidermal necrolysis | 10044223 | |
| Toxic skin eruption | 10057970 | |

| PTs (Selective)G3 and higher | |
|------------------------------|----------|
| Eyelid rash | 10074620 |
| Genital rash | 10018175 |
| Mucocutaneous rash | 10056671 |
| Nodular rash | 10075807 |
| Perineal rash | 10075364 |
| Rash | 10037844 |
| Rash erythematous | 10037855 |
| Rash generalised | 10037858 |
| Rash macular | 10037867 |
| Rash maculo-papular | 10037868 |
| Rash maculovesicular | 10050004 |
| Rash morbilliform | 10037870 |
| Rash papular | 10037876 |
| Rash rubelliform | 10057984 |
| Rash scarlatiniform | 10037890 |
| Rash vesicular | 10037898 |
| Rash pruritic | 10037884 |
| Rash follicular | 10037857 |
| Rash pustular | 10037888 |
| Drug eruption | 10013687 |

Notes: Medical concept of severe cutaneous adverse reactions. Only narrow terms from SMQ 'Severe cutaneous adverse reactions' selected. <u>Plus</u> several additional preferred terms [only G3 and higher] selected from HLTs 'Rashes, eruptions and exanthems NEC', 'Pruritus NEC', 'Pustular conditions', 'Dermatitis ascribed to specific agent' all under SOC 'Skin and subcutaneous tissue disorders'

| Torsade de pointes/QT prolongation (SMQ) | 20000001 |
|------------------------------------------|----------|
| PT | PT Code |
| Electrocardiogram QT interval abnormal | 10063748 |
| Electrocardiogram QT prolonged | 10014387 |
| Long QT syndrome | 10024803 |
| Long QT syndrome congenital | 10057926 |
| Torsade de pointes | 10044066 |
| Ventricular tachycardia | 10047302 |

| 1 | de pointes/QT prolongation' selected <u>plus</u> one additional PT under HLT 'ECG investigations'. |
|---|---|
| | Notes: Medical concept of QT prolongation and complications. Only narrow terms from SMQ 'Torsade |

| PTs (Selective) | | rs (Selective) |
|---|---|---|
| | Electrocardiogram repolarisation abnormality | 10052464 |

| Suicide/self-injury (SMQ) | 20000037 |
|-------------------------------------------------|----------|
| PT | PT Code |
| Assisted suicide | 10079105 |
| Columbia suicide severity rating scale abnormal | 10075616 |
| Completed suicide | 10010144 |
| Depression suicidal | 10012397 |
| Intentional overdose | 10022523 |
| Intentional self-injury | 10022524 |
| Poisoning deliberate | 10036000 |
| Self-injurious ideation | 10051154 |
| Suicidal behaviour | 10065604 |
| Suicidal ideation | 10042458 |
| Suicide attempt | 10042464 |
| Suicide threat | 10077417 |

Notes: Medical concept of suicidal ideation and behaviour. Sub-SMQ 'Suicide/self-injury' (SMQ) from parent SMQ of 'Depression and Suicide/Self Injury'. Only narrow terms from the sub-SMQ selected.

| Depression (excl suicide and self injury) (SMQ) - | 20000167 |
|-----------------------------------------------------------|----------|
| PT | PT Code |
| Activation syndrome | 10066817 |
| Adjustment disorder with depressed mood | 10001297 |
| Adjustment disorder with mixed anxiety and depressed mood | 10001299 |
| Agitated depression | 10001496 |
| Anhedonia | 10002511 |
| Antidepressant therapy | 10054976 |
| Childhood depression | 10068631 |
| Decreased interest | 10011971 |
| Depressed mood | 10012374 |
| Depression | 10012378 |
| Depression postoperative | 10012390 |
| Depressive symptom | 10054089 |
| Dysphoria | 10013954 |
| Electroconvulsive therapy | 10014404 |
| Feeling guilty | 10049708 |
| Feeling of despair | 10016344 |
| Feelings of worthlessness | 10016374 |
| Helplessness | 10077169 |
| Major depression | 10057840 |
| Menopausal depression | 10067371 |
| Mixed anxiety and depressive disorder | 10080836 |
| Perinatal depression | 10078366 |
| Persistent depressive disorder | 10077804 |
| Post stroke depression | 10070606 |
| Postictal depression | 10071324 |

| HLGT Manic and Bipolar mood disorders and disturbances | |
|--------------------------------------------------------|----------|
| PT | PT Code |
| Bipolar I disorder | 10004939 |
| Bipolar II disorder | 10004940 |
| Bipolar disorder | 10057667 |
| Cyclothymic disorder | 10011724 |
| Hypomania | 10021030 |
| Mania | 10026749 |

Notes: Medical concept of bipolar disorder. All preferred terms from HLGT 'Manic and Bipolar mood disorders and disturbances' under SOC 'Psychiatric disorders'.

20000117 selected. Psychosis and psychotic disorders (SMQ) 20000117 PT PT Code Acute psychosis 10001022 Alcoholic psychosis 10001632 Alice in wonderland syndrome 10001666 Brief psychotic disorder with marked stressors 10048549 10056395 Brief psychotic disorder without marked stressors Brief psychotic disorder, with postpartum onset 10006362 Charles Bonnet syndrome 10063354 Childhood psychosis 10061040 10009232 Clang associations Cotard's syndrome 10059591 Delusion 10012239 Delusion of grandeur 10012241 10012244 Delusion of reference Delusion of replacement 10012245 Delusional disorder, erotomanic type 10012249 Delusional disorder, grandiose type 10012250 Delusional disorder, jealous type 10012251 Delusional disorder, mixed type 10012252 Delusional disorder, persecutory type 10053195 Delusional disorder, somatic type 10012254 10012255 Delusional disorder, unspecified type **Delusional perception** 10012258 Dementia of the Alzheimer's type, with delusions 10012295 Depressive delusion 10063033 Derailment 10012411 Epileptic psychosis 10059232 10015134 Erotomanic delusion 10016777 Flight of ideas Hallucination 10019063 Hallucination, auditory 10019070 Hallucination, gustatory 10019071 Hallucination, olfactory 10019072 10062824 Hallucination, synaesthetic 10019074 Hallucination, tactile Hallucination, visual 10019075 10019079 Hallucinations, mixed

Hypnagogic hallucination

Hysterical psychosis

Hypnopompic hallucination

Notes: Medical concept of psychosis. Only narrow terms from SMQ 'Psychosis and psychotic disorders'

10020927

| PT | PT Code |
|-------------------------------------------------------|----------|
| Ideas of reference | 10021212 |
| Illusion | 10021403 |
| Jealous delusion | 10023164 |
| Loose associations | 10024825 |
| Mixed delusion | 10076429 |
| Neologism | 10028916 |
| Neuroleptic-induced deficit syndrome | 10075295 |
| Paranoia | 10033864 |
| Paranoid personality disorder | 10033869 |
| Parkinson's disease psychosis | 10074835 |
| Paroxysmal perceptual alteration | 10063117 |
| Persecutory delusion | 10034702 |
| Postictal psychosis | 10070669 |
| Post-injection delirium sedation syndrome | 10072851 |
| Posturing | 10036437 |
| Psychosis postoperative | 10065617 |
| Psychotic behaviour | 10037249 |
| Psychotic disorder | 10061920 |
| Psychotic disorder due to a general medical condition | 10061921 |
| Reactive psychosis | 10053632 |
| Rebound psychosis | 10074833 |
| Schizoaffective disorder | 10039621 |
| Schizoaffective disorder bipolar type | 10068889 |
| Schizoaffective disorder depressive type | 10068890 |
| Schizophrenia | 10039626 |
| Schizophreniform disorder | 10039647 |
| Schizotypal personality disorder | 10039651 |
| Senile psychosis | 10039987 |
| Shared psychotic disorder | 10040535 |
| Somatic delusion | 10041317 |
| Somatic hallucination | 10062684 |
| Substance-induced psychotic disorder | 10072388 |
| Tangentiality | 10043114 |
| Thought blocking | 10043495 |
| Thought broadcasting | 10052214 |
| Thought insertion | 10043496 |
| Thought withdrawal | 10043497 |
| Transient psychosis | 10056326 |
| Waxy flexibility | 10047853 |

| HLGT Mood disorders and disturbances NEC, Psychiatric disorders SOC | |
|---|---|
| PT | PT Code |
| Crying | 10011469 |
| Mood swings | 10027951 |
| Boredom | 10048909 |
| Mood altered | 10027940 |
| Apathy | 10002942 |
| Affective ambivalence | 10077173 |
| Emotional poverty | 10014557 |
| Euphoric mood | 10015535 |
| Premenstrual dysphoric disorder | 10051537 |
| Alexithymia | 10077719 |
| Laziness | 10051602 |
| Blunted affect | 10005885 |
| Constricted affect | 10010778 |
| Affect lability | 10054196 |
| Anger | 10002368 |
| Affective disorder | 10001443 |
| Lethargy | 10024264 |
| Listless | 10024642 |
| Inappropriate affect | 10021588 |
| Dysphoria | 10013954 |
| Mood disorder due to a general medical con | 10027944 |
| Morose | 10027977 |
| Screaming | 10039740 |
| Steroid withdrawal syndrome | 10042028 |
| Emotional disorder | 10014551 |
| Irritability | 10022998 |
| Moaning | 10027783 |
| Premenstrual syndrome | 10036618 |
| Neuroleptic-induced deficit syndrome | 10075295 |
| Substance-induced mood disorder | 10072387 |
| Flat affect | 10016759 |
| Diencephalic syndrome of infancy | 10012774 |
| Emotional distress | 10049119 |
| Frustration tolerance decreased | 10077753 |
| Seasonal affective disorder | 10039775 |

| HLGT Anxiety disorders and symper | PT Code |
|-----------------------------------------------------|----------|
| Acrophobia Acrophobia | 10000605 |
| Activation syndrome | 10066817 |
| Acute stress disorder | 10000017 |
| Aerophobia | 10080300 |
| Agitation | 10001497 |
| Agitation neonatal | 10001500 |
| Agitation postoperative | 10049989 |
| Agoraphobia | 10001502 |
| Akathisia | 10001540 |
| Algophobia | 10078056 |
| Animal phobia | 10002518 |
| Anniversary reaction | 10074066 |
| Anticipatory anxiety | 10002758 |
| Anxiety | 10002855 |
| Anxiety disorder | 10057666 |
| Anxiety disorder due to a general medical condition | 10002859 |
| Arachnophobia | 10051408 |
| Astraphobia | 10078372 |
| Autophobia | 10071070 |
| Body dysmorphic disorder | 10052793 |
| Burnout syndrome | 10065369 |
| Claustrophobia | 10009244 |
| Compulsions | 10010219 |
| Compulsive cheek biting | 10076510 |
| Compulsive handwashing | 10071263 |
| Compulsive hoarding | 10068007 |
| Compulsive lip biting | 10066241 |
| Compulsive shopping | 10067948 |
| Dermatillomania | 10065701 |
| Dysmorphophobia | 10049096 |
| Emetophobia | 10070637 |
| Fear | 10016275 |
| Fear of animals | 10016276 |
| Fear of closed spaces | 10016277 |
| Fear of crowded places | 10050365 |
| Fear of death | 10066392 |
| Fear of disease | 10016278 |
| Fear of eating | 10050366 |

Notes: Medical concept of anxiety disorders. All preferred terms from HLGT 'Anxiety disorders and symptoms', under SOC 'Psychiatric disorders'.

| PT | PT Code |
|--------------------------------------------------------|----------|
| Fear of falling | 10048744 |
| Fear of injection | 10073753 |
| Fear of open spaces | 10016279 |
| Fear of pregnancy | 10067035 |
| Fear of weight gain | 10016280 |
| Fear-related avoidance of activities | 10080136 |
| Generalised anxiety disorder | 10018075 |
| Glossophobia | 10080077 |
| Haemophobia | 10073458 |
| Haphephobia | 10067580 |
| Hydrophobia | 10053317 |
| Hyperarousal | 10080831 |
| Immunisation anxiety related reaction | 10075205 |
| Kinesiophobia | 10078430 |
| Limited symptom panic attack | 10024511 |
| Mysophobia | 10078769 |
| Nail picking | 10066779 |
| Nervousness | 10029216 |
| Neurosis | 10029333 |
| Noctiphobia | 10057946 |
| Nocturnal fear | 10057948 |
| Nosophobia | 10063546 |
| Obsessive need for symmetry | 10077179 |
| Obsessive rumination | 10056264 |
| Obsessive thoughts | 10029897 |
| Obsessive-compulsive disorder | 10029898 |
| Obsessive-compulsive symptom | 10077894 |
| Ochlophobia | 10050095 |
| Osmophobia | 10060765 |
| Paediatric autoimmune neuropsychiatric disorders assoc | 10072147 |
| Panic attack | 10033664 |
| Panic disorder | 10033666 |
| Panic reaction | 10033670 |
| Paruresis | 10069024 |
| Performance fear | 10034432 |
| Phagophobia | 10050096 |
| Pharmacophobia | 10069423 |
| Phobia | 10034912 |
| Phobia of driving | 10056676 |
| Phobia of exams | 10034913 |
| Phobic avoidance | 10034918 |

| PT | PT Code |
|--------------------------------|----------|
| Phonophobia | 10054956 |
| Photaugiaphobia | 10064420 |
| Post-traumatic stress disorder | 10036316 |
| Postpartum neurosis | 10036419 |
| Postpartum stress disorder | 10056394 |
| Procedural anxiety | 10075204 |
| Pseudoangina | 10056610 |
| Selective mutism | 10039917 |
| Separation anxiety disorder | 10040045 |
| Sitophobia | 10080170 |
| Social anxiety disorder | 10041242 |
| Social fear | 10041247 |
| Stress | 10042209 |
| Tension | 10043268 |
| Terminal agitation | 10077416 |
| Thanatophobia | 10064723 |
| Thermophobia | 10075147 |
| Trichotemnomania | 10072752 |
| Trichotillomania | 10044629 |

Notes: Medical concept of sleep disorders. All preferred terms from (1) HLGT 'Sleep Disorders and Disturbances', 'Psychiatric disorders' SOC <u>plus</u> (2)HLGT 'Sleep disturbances (incl subtypes)', 'Nervous system' SOC. Numerous duplicated preferred terms e.g. middle insomnia

### **HLGT Sleep Disorders and Disturbances**

| PT | PT Code |
|-------------------------------------------------------------------|----------|
| Behavioural insomnia of childhood | 10072072 |
| Hyposomnia | 10067530 |
| Initial insomnia | 10022035 |
| Insomnia | 10022437 |
| Middle insomnia | 10027590 |
| Terminal insomnia | 10068932 |
| Breathing-related sleep disorder | 10006344 |
| Dyssomnia | 10061827 |
| Hypersomnia | 10020765 |
| Periodic limb movement disorder | 10064600 |
| Pickwickian syndrome | 10035004 |
| Poor quality sleep | 10062519 |
| Sleep apnoea syndrome | 10040979 |
| Somnolence | 10041349 |
| Somnolence neonatal | 10041350 |
| Stupor | 10042264 |
| Upper airway resistance syndrome | 10063968 |
| Cataplexy | 10007737 |
| Hypnagogic hallucination | 10020927 |
| Hypnopompic hallucination | 10020928 |
| Narcolepsy | 10028713 |
| Sleep attacks | 10040981 |
| Sleep paralysis | 10041002 |
| Abnormal dreams | 10000125 |
| Abnormal sleep-related event | 10061613 |
| Confusional arousal | 10067494 |
| Exploding head syndrome | 10080684 |
| Loss of dreaming | 10065085 |
| Nightmare | 10029412 |
| Parasomnia | 10061910 |
| Rapid eye movement sleep behaviour disorder | 10077299 |
| Rapid eye movements sleep abnormal | 10037841 |
| Sleep inertia | 10067493 |
| Sleep sex | 10067492 |
| Sleep talking | 10041009 |
| Sleep terror | 10041010 |
| Sleep-related eating disorder | 10067315 |
| Somnambulism | 10041347 |
| Hypersomnia related to another mental condition | 10020767 |
| Hypersomnia-bulimia syndrome | 10053712 |
| Insomnia related to another mental condition | 10022443 |
| Sleep disorder | 10040984 |
| Sleep disorder due to a general medical condition | 10063910 |
| Sleep disorder due to general medical condition, hypersomnia type | 10040985 |
| Sleep disorder due to general medical condition, insomnia type | 10040986 |
| Sleep disorder due to general medical condition, mixed type | 10040987 |
| Sleep disorder due to general medical condition, parasomnia type | 10040988 |

| PT | PT Code |
|--------------------------------------|----------|
| Sopor | 10058709 |
| Advanced sleep phase | 10001423 |
| Circadian rhythm sleep disorder | 10009191 |
| Delayed sleep phase | 10012209 |
| Irregular sleep phase | 10022995 |
| Irregular sleep wake rhythm disorder | 10080301 |
| Non-24-hour sleep-wake disorder | 10078086 |
| Shift work disorder | 10078088 |

| HLGT Sleep disturbances (incl subtypes) | |
|---------------------------------------------|----------|
| PT | PT Code |
| Abnormal dreams | 10000125 |
| Abnormal sleep-related event | 10061613 |
| Confusional arousal | 10067494 |
| Loss of dreaming | 10065085 |
| Sleep inertia | 10067493 |
| Sleep paralysis | 10041002 |
| Sleep sex | 10067492 |
| Sleep talking | 10041009 |
| Sleep terror | 10041010 |
| Sleep-related eating disorder | 10067315 |
| Somnambulism | 10041347 |
| Behavioural insomnia of childhood | 10072072 |
| Hyposomnia | 10067530 |
| Initial insomnia | 10022035 |
| Insomnia | 10022437 |
| Middle insomnia | 10027590 |
| Terminal insomnia | 10068932 |
| Advanced sleep phase | 10001423 |
| Circadian rhythm sleep disorder | 10009191 |
| Delayed sleep phase | 10012209 |
| Irregular sleep phase | 10022995 |
| Irregular sleep wake rhythm disorder | 10080301 |
| Non-24-hour sleep-wake disorder | 10078086 |
| Shift work disorder | 10078088 |
| Cataplexy | 10007737 |
| Hypersomnia | 10020765 |
| Narcolepsy | 10028713 |
| Central-alveolar hypoventilation | 10007982 |
| Sleep apnoea syndrome | 10040979 |
| Breathing-related sleep disorder | 10006344 |
| Dyssomnia | 10061827 |
| Fatal familial insomnia | 10072077 |
| Microsleep | 10076954 |
| Periodic limb movement disorder | 10064600 |
| Pickwickian syndrome | 10035004 |
| Poor quality sleep | 10062519 |
| Rapid eye movement sleep behaviour disorder | 10077299 |
| Rapid eye movements sleep abnormal | 10037841 |
| Sleep deficit | 10080881 |
| Sudden onset of sleep | 10050014 |

CONFIDENTIAL 2020N435253\_00 206898

| PT | PT Code |
|----------------------------------|----------|
| Upper airway resistance syndrome | 10063968 |

| Convulsions (SMQ) | 20000079 |
|-----------------------------------------------------------------|----------|
| PT | PT Code |
| 2-Hydroxyglutaric aciduria | 10078971 |
| Acquired epileptic aphasia | 10052075 |
| Acute encephalitis with refractory, repetitive partial seizures | 10076948 |
| Alcoholic seizure | 10056347 |
| Aspartate-glutamate-transporter deficiency | 10079140 |
| Atonic seizures | 10003628 |
| Atypical benign partial epilepsy | 10056699 |
| Automatism epileptic | 10003831 |
| Autonomic seizure | 10049612 |
| Baltic myoclonic epilepsy | 10054895 |
| Benign familial neonatal convulsions | 10067866 |
| Benign rolandic epilepsy | 10070530 |
| Biotinidase deficiency | 10071434 |
| Change in seizure presentation | 10075606 |
| Clonic convulsion | 10053398 |
| Convulsion in childhood | 10052391 |
| Convulsion neonatal | 10010911 |
| Convulsions local | 10010920 |
| Convulsive threshold lowered | 10010927 |
| CSWS syndrome | 10078827 |
| Deja vu | 10012177 |
| Double cortex syndrome | 10073490 |
| Dreamy state | 10013634 |
| Drug withdrawal convulsions | 10013752 |
| Early infantile epileptic encephalopathy with burst-suppression | 10071545 |
| Eclampsia | 10014129 |
| Epilepsy | 10015037 |
| Epilepsy surgery | 10079824 |
| Epileptic aura | 10015049 |
| Epileptic psychosis | 10059232 |
| Febrile convulsion | 10016284 |
| Febrile infection-related epilepsy syndrome | 10079438 |
| Focal dyscognitive seizures | 10079424 |
| Frontal lobe epilepsy | 10049424 |
| Generalised non-convulsive epilepsy | 10018090 |
| Generalised tonic-clonic seizure | 10018100 |
| Glucose transporter type 1 deficiency syndrome | 10078727 |
| Gray matter heterotopia | 10080533 |
| Hemimegalencephaly | 10078100 |
| Hyperglycaemic seizure | 10071394 |

Notes: Medical concept of seizures. Only narrow terms from SMQ 'Convulsions' selected <u>plus</u> selected PTs of possible seizure events from HLT 'Disturbances in consciousness NEC' under SOC 'Nervous systems disorders' and HLT 'Confusion and disorientation' under SOC 'Psychiatric disorders'.

| PT | PT Code |
|------------------------------------------------|----------|
| Hypocalcaemic seizure | 10072456 |
| Hypoglycaemic seizure | 10048803 |
| Hyponatraemic seizure | 10073183 |
| Idiopathic generalised epilepsy | 10071081 |
| Infantile spasms | 10021750 |
| Juvenile myoclonic epilepsy | 10071082 |
| Lafora's myoclonic epilepsy | 10054030 |
| Lennox-Gastaut syndrome | 10048816 |
| Migraine-triggered seizure | 10076676 |
| Molybdenum cofactor deficiency | 10069687 |
| Multiple subpial transection | 10079825 |
| Myoclonic epilepsy | 10054859 |
| Myoclonic epilepsy and ragged-red fibres | 10069825 |
| Partial seizures | 10061334 |
| Partial seizures with secondary generalisation | 10056209 |
| Petit mal epilepsy | 10034759 |
| Polymicrogyria | 10073489 |
| Post stroke epilepsy | 10076982 |
| Post stroke seizure | 10076981 |
| Postictal headache | 10052470 |
| Postictal paralysis | 10052469 |
| Postictal psychosis | 10070669 |
| Postictal state | 10048727 |
| Post-traumatic epilepsy | 10036312 |
| Schizencephaly | 10073487 |
| Seizure | 10039906 |
| Seizure anoxic | 10039907 |
| Seizure cluster | 10071350 |
| Seizure like phenomena | 10071048 |
| Severe myoclonic epilepsy of infancy | 10073677 |
| Simple partial seizures | 10040703 |
| Status epilepticus | 10041962 |
| Sudden unexplained death in epilepsy | 10063894 |
| Temporal lobe epilepsy | 10043209 |
| Tonic clonic movements | 10051171 |
| Tonic convulsion | 10043994 |
| Tonic posturing | 10075125 |
| Topectomy | 10073488 |
| Tuberous sclerosis complex | 10080584 |
| Uncinate fits | 10045476 |

| PTs (Select | ive) |
|-------------------|----------|
| Confusional state | 10010305 |

| PT | PT Code |
|----------------------------------|----------|
| Loss of consciousness | 10024855 |
| Syncope | 10042772 |
| Sopor | 10058709 |
| Stupor | 10042264 |
| Altered state of consciousness | 10050093 |
| Depressed level of consciousness | 10012373 |
| Consciousness fluctuating | 10050093 |

| Acute renal failure (SMQ) | 20000 | Notes: Medical concept of worsening renal function/renal failure in the context of impact of creatinine. Only narrow terms from SMQ 'Acute renal failure' plus all PTs from HLT 'Renal failure impairment', under SOC 'Renal and urinary disorders'. Numerous duplicated preferred terms renal failure |
|---|---|---|
| PT | PT Code | |
| Acute kidney injury | 10069339 | |
| Acute phosphate nephropathy | 10069688 | |
| Anuria | 10002847 | |
| Azotaemia | 10003885 | |
| Continuous haemodiafiltration | 10066338 | |
| Dialysis | 10061105 | |
| Foetal renal impairment | 10078987 | |
| Haemodialysis | 10018875 | |
| Haemofiltration | 10053090 | |
| Hyponatriuria | 10077515 | |
| Neonatal anuria | 10049778 | |
| Nephropathy toxic | 10029155 | |
| Oliguria | 10030302 | |
| Peritoneal dialysis | 10034660 | |
| Prerenal failure | 10072370 | |
| Renal failure | 10038435 | |
| Renal failure neonatal | 10038447 | |
| Renal impairment | 10062237 | |
| Renal impairment neonatal | 10049776 | |

| Renal Failure and Impairment HLT | |
|--------------------------------------|----------|
| PT | PT Code |
| Acute Kidney injury | 10069339 |
| Anuria | 10002847 |
| Atypical haemolytic uraemic syndrome | 10079840 |
| Cardiorenal syndrome | 10068230 |
| Chronic kidney disease | 10064848 |
| Crush syndrome | 10050702 |
| Diabetic end stage renal disease | 10012660 |
| End stage renal disease | 10077512 |
| Foetal renal impairment | 10078987 |
| Haemolytic uraemic syndrome | 10018932 |
| Hepatorenal failure | 10019845 |
| Hepatorenal syndrome | 10019846 |

| | 10038447 |
|----------------|--------------|
| | 10062237 |
| al | 10049776 |
| Failure and Im | pairment HLT |
| | PT Code |
| | 10069339 |
| | 10002847 |
| nic syndrome | 10079840 |
| | 10068230 |
| | 10064848 |
| | 10050702 |
| disease | 10012660 |
| | 10077512 |
| | 10078987 |
| rome | 10018932 |
| | 10019845 |
| | 10019846 |

| PT | PT Code |
|-----------------------------|----------|
| Nail-patella syndrome | 10063431 |
| Neonatal anuria | 10049778 |
| Oliguria | 10030302 |
| Pancreatorenal syndrome | 10056277 |
| Postoperative renal failure | 10056675 |
| Postrenal failure | 10059345 |
| Prerenal failure | 10072370 |
| Propofol infusion syndrome | 10063181 |
| Renal failure | 10038435 |
| Renal failure neonatal | 10038447 |
| Renal impairment | 10062237 |
| Renal impairment neonatal | 10049776 |
| Renal injury | 10061481 |
| Scleroderma renal crisis | 10062553 |
| Traumatic anuria | 10044501 |

| Tubulointerstitial diseases (SMQ) | 20000221 | Notes: Mea | lical concept of Proximal R |
|---|---|---|---|
| | | 'Tubuloir | nterstitial diseases'. |
| | PT Code | | |
| Acidosis hyperchloraemic | 10000489 | | |
| Acquired aminoaciduria | 10073515 | | |
| Acute phosphate nephropathy | 10069688 | | |
| Aminoaciduria | 10001939 | | |
| Beta-N-acetyl-D-glucosaminidase increased | | | |
| Crystal nephropathy | 10071503 | | |
| Eosinophils urine present | 10058363 | | |
| Fanconi syndrome acquired | 10052607 | | |
| Hyperphosphaturia | 10051232 | | |
| Isosthenuria | 10023077 | | |
| Nephritis allergic | 10029120 | | |
| Nephrogenic diabetes insipidus | 10029147 | | |
| Nephropathy toxic | 10029155 | | |
| Renal glycosuria | 10038457 | | |
| Renal papillary necrosis | 10038491 | | |
| Renal tubular acidosis | 10038535 | | |
| Renal tubular atrophy | 10038536 | | |
| Renal tubular disorder | 10038537 | | |
| Renal tubular dysfunction | 10050335 | | |
| Tubulointerstitial nephritis | 10048302 | | |
| Tubulointerstitial nephritis and uveitis syndro | 10069034 | | |
| Urine phosphorus increased | 10055030 | | |
| Urine retinol binding protein increased | 10061432 | | |

| Proteinuria (SMQ) | 20000220 | Notes: Medical concept of Proteinuria. Only narrow terms from narrow SMQ 'Proteinuria' included. |
|---|---|---|
| PT | PT Code | |
| Albumin globulin ratio increased | 10001567 | |
| Albumin urine present | 10001582 | |
| Albuminuria | 10001580 | |
| Bence Jones protein urine present | 10053112 | |
| Bence Jones proteinuria | 10004231 | |
| Beta 2 microglobulin urine increased | 10004501 | |
| Globulinuria | 10018352 | |
| Microalbuminuria | 10027525 | |
| Myoglobinuria | 10028629 | |
| Orthostatic proteinuria | 10031129 | |
| Protein urine | 10037018 | |
| Protein urine present | 10053123 | |
| Proteinuria | 10037032 | |
| Urine albumin/creatinine ratio increased | 10053541 | |
| Urine protein/creatinine ratio abnormal | 10053539 | |
| Urine protein/creatinine ratio increased | 10053538 | |

#### The GlaxoSmithKline group of companies

206898

| Division | : Worldwide Development |
|------------------|-------------------------------------|
| Information Type | : Reporting and Analysis Plan (RAP) |

Title : Reporting and Analysis Plan for 206898: An Open Label, Phase 1 Study to Evaluate the PK, Safety, Tolerability and Acceptability of Long Acting Injections of the HIV Integrase Inhibitor, Cabotegravir (CAB; GSK1265744) in HIV Uninfected Chinese Men

Compound Number : GSK1265744

Effective Date : 28-SEP-2018

### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 206898.
- This RAP is intended to describe the safety, tolerability, and pharmacokinetic (PK) analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

#### **Author's Name and Functional Area:**

| PPD | 11-SEP-2018 |
|-------------------------|-------------|
| Biostatistician II, PPD | 11-SEF-2016 |

| PPD | | 11-SEP-2018 |
|-----------------|---------------------------|-------------|
| Pharmacokinetic | cist (Biostatistics, PPD) | 11-SEF-2016 |

### Approved by:

| PPD | 20 CED 2010 |
|--------------------------------|-------------|
| Statistician, GSK 28-SEP-2018 | |
| PPD | 20 CED 2010 |
| Manager Statistics 28-SEP-2018 | |

Copyright 2018 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

206898

### **TABLE OF CONTENTS**

| | | | | | PAGE |
|---|---|---|---|---|---|
| 1. | REPOR | TING & | ANALYSIS | PLAN SYNOPSIS | 5 |
| 2. | SUMMA | ARY OF I | KEY PROT | OCOL INFORMATION | 9 |
| | | | | tocol Defined Statistical Analysis Plan | |
| | | | | and Endpoint(s) | |
| | | | | es | |
| 3. | PLANN | ED ANAI | YSES | | 12 |
| | 3.1. I | nterim A | nalyses | | 12 |
| | 3.2. F | Final Ana | alyses | | 12 |
| 4. | ANALYS | SIS POP | ULATIONS | S | 13 |
| | 4.1. F | Protocol | Deviations | | 14 |
| 5. | CONSIE | DERATIO | ONS FOR I | DATA ANALYSES AND DATA HANDLING | |
| | | | | | 15 |
| 6. | STUDY | POPUL | ATION AN | ALYSES | 16 |
| | 6.1. | Overview | of Planne | d Analyses | 16 |
| | 6 | 3.1.1. | | n | |
| | | 3.1.2. | | phics | |
| | | 3.1.3. | Medical H | istory | 17 |
| | - | 5.1.4. | | Concomitant Medications | |
| | 6 | 6.1.5. | Protocol L | Deviation | 17 |
| 7. | | | | NALYSES | |
| | | | nalyses of | CAB LA | 18 |
| | | 7.1.1. | | Site Reaction | |
| | | 7.1.2. | | vents | |
| | | 7.1.3. | | aboratory Tests | |
| | - | 7.1.4. | | Assessments | |
| | | 7.1.5. | | f OAD I A | |
| | | | | s of CAB LA | |
| | | | | inetic Analyses | |
| | | 7.3.1.<br>7.3.2. | | of Planned Primary Pharmacokinetic Analyses rug Concentration Measures | |
| | | 7.3.2.<br>7.3.3. | | harmacokinetic Parameters | |
| | , | 1.3.3. | 7.3.3.1. | Deriving Primary Pharmacokinetic Parameters | |
| | | | 7.3.3.1. | Statistical Analysis of Primary Pharmacokinetic | |
| | | | | Parameters | 25 |
| 8. | | | | AL ANALYSES | |
| | 8.1. | Seconda | ry Pharma | cokinetic Analyses | 27 |

| | | | | 206898 |
|---|---|---|---|---|
| | | 8.1.1. | Overview of Planned Secondary Pharmacokinetic | |
| | | | Analyses | 27 |
| | | 8.1.2. | Secondary Drug Concentration Measures | |
| | | 8.1.3. | Secondary Pharmacokinetic Parameters | 27 |
| | | | 8.1.3.1. Deriving Secondary Pharmacokinetic | |
| | | | Parameters | 27 |
| | 8.2. | Safety a | nd Tolerability Analyses of Oral CAB | 28 |
| | 8.3. | | bility of CAB LA | |
| | 8.4. | | ration-effect Relationships for Safety and Tolerability | |
| | | | ters | 30 |
| | 8.5. | | Safety Analyses | |
| | | 8.5.1. | Extent of Exposure to CAB | |
| | | 8.5.2. | Possible suicidality-related Adverse Events | |
| | | 8.5.3. | Social Harms | |
| | | 8.5.4. | ECG | |
| | | 8.5.5. | Cardiovascular Events | |
| | | 8.5.6. | Liver Events | |
| | | 0.0.0. | | |
| 9. | REFE | RENCES | | 35 |
| 10 | 4 DDE | NDICEC | | 20 |
| 10. | | | . 4. Destroy Deviation Management and Definitions for Dev | 36 |
| | 10.1. | | x 1: Protocol Deviation Management and Definitions for Per | 07 |
| | | Protocol | Population | 37 |
| | 40.0 | | Exclusions from Per Protocol Population | |
| | 10.2. | | x 2: Time & Events | |
| | | | Protocol Defined Time & Events | |
| | 10.3. | | x 3: Assessment Windows | |
| | | 10.3.1. | | |
| | 10.4. | | x 4: Study Phase and State | |
| | | 10.4.1. | | |
| | | 10.4.2. | Treatment States | |
| | | | 10.4.2.1. Treatment States for AE Data | |
| | 10.5. | Appendi | x 5: Data Display Standards & Handling Conventions | 44 |
| | | 10.5.1. | | 44 |
| | | 10.5.2. | Baseline Definition & Derivations | 44 |
| | | | 10.5.2.1. Baseline Definitions | 44 |
| | | | 10.5.2.2. Derivations and Handling of Missing Baseline | |
| | | | Data | |
| | | | Reporting Process & Standards | |
| | 10.6. | Appendi | x 6: Derived and Transformed Data | 47 |
| | | 10.6.1. | General | |
| | | 10.6.2. | Study Population | 47 |
| | | 10.6.3. | Safety | 48 |
| | 10.7. | Appendi | x 7: Premature Withdrawals & Handling of Missing Data | |
| | | 10.7.1. | Premature Withdrawals | |
| | | 10.7.2. | Handling of Missing Data | |
| | | | 10.7.2.1. Handling of Missing Dates | |
| | | | 10.7.2.2. Handling of Partial Dates | |

| | | 206898 |
|---|---|---|
| | 10.7.2.3. Handling of Missing Data for Statistical | |
| | Analysis | 50 |
| 10.8. | Appendix 8: Values of Potential Clinical Importance | |
| | 10.8.1. Laboratory Values | |
| | 10.8.2. ECG | |
| | 10.8.3. Vital Signs | |
| 10.9. | Appendix 9: Multicenter Studies | |
| | 10.9.1. Methods for Handling Centres | |
| 10.10. | Appendix 10: Examination of Covariates, Subgroups & Other Strata | 54 |
| | 10.10.1. Handling of Covariates, Subgroups & Other Strata | 54 |
| 10.11. | Appendix 11: Multiple Comparisons & Multiplicity | 55 |
| | 10.11.1. Handling of Multiple Comparisons & Multiplicity | 55 |
| 10.12. | Appendix 12: Model Checking and Diagnostics for Statistical | |
| | Analyses | 56 |
| | 10.12.1. Statistical Analysis Assumptions | |
| 10.13. | Appendix 13 – Abbreviations & Trade Marks | 57 |
| | 10.13.1. Abbreviations | |
| | 10.13.2. Trademarks | |
| 10.14. | Appendix 14: List of Data Displays | |
| | 10.14.1. Data Display Numbering | |
| | 10.14.2. Mock Example Shell Referencing | |
| | 10.14.3. Deliverable [Priority] | |
| | 10.14.4. Study Population Tables | |
| | 10.14.5. Safety Tables | |
| | 10.14.6. Tolerability Tables | |
| | 10.14.7. Acceptability Tables | |
| | 10.14.8. Pharmacokinetic Tables | |
| | 10.14.9. Pharmacokinetic Figures | |
| | 10.14.10.ICH Listings | |
| 40.45 | 10.14.11.Non-ICH Listings | |
| 10.15. | Appendix 15: Example Mock Shells for Data Displays | /5 |

206898

# 1. REPORTING & ANALYSIS PLAN SYNOPSIS

| Overview | Key Elements of the RAP |
|---|---|
| Purpose | <ul> <li>The purpose of this reporting and analysis plan (RAP) is to describe any<br/>planned analyses and output to be included in the clinical study report for<br/>Protocol 206898.</li> </ul> |
| Protocol | This RAP is based on the Protocol Amendment 1 (Dated: 06JUN2018) of study Protocol 206898 (GSK Document No.: 2016N293702_00] and eCRF Version (1.00, Dated: 09MAR2018). |
| Primary<br>Objective | Evaluate the safety and tolerability of the injectable agent, cabotegravir (GSK1265744) long acting (CAB LA) injectable (600 mg dose administered every 4 weeks for 2 doses followed by every 8 weeks for 3 doses) through Week 5-41 in HIV-1 uninfected Chinese men. |
| | <ul> <li>Evaluate the plasma pharmacokinetics of CAB following repeat oral<br/>administration (Day 1 to Week 4) and CAB LA IM injections throughout the<br/>Injection Phase (Weeks 5-41).</li> </ul> |
| Primary<br>Endpoint | <ul> <li>Safety and tolerability parameters, including adverse events, clinical laboratory<br/>tests, study withdrawals due to AEs, vital signs assessments, and evaluation of<br/>injection site reactions (ISRs), for injection phase (Week 5-41).</li> </ul> |
| | <ul> <li>Plasma CAB AUC(0-τ), Cmax, Cτ, tmax, λz, t½, CL/F, and Vz/F following daily oral administration of CAB through Day 1 to Week 4.</li> </ul> |
| | <ul> <li>Plasma CAB AUC(0-τ), Cmax, Cτ, and tmax following IM injections of CAB LA<br/>once every 8 weeks through Weeks 5-41.</li> </ul> |
| Secondary<br>Objective | <ul> <li>Evaluate the plasma pharmacokinetics of CAB LA throughout the Injection and<br/>Long-term Follow-up Phases (Week 5 to Week 89).</li> </ul> |
| | <ul> <li>Evaluate the safety and tolerability of oral CAB in HIV uninfected Chinese men<br/>during the oral lead-in Phase (Day 1 to Week 4)</li> </ul> |
| | Evaluate the acceptability of CAB LA injections through 41 weeks. |
| | Explore concentration-effect relationships for various safety and tolerability parameters if relevant. |
| Secondary<br>Endpoint | <ul> <li>Plasma CAB AUC(0-τ), Cmax, Cτ, tmax, λz, t½, CL/F, and Vz/F through Weeks<br/>5-89.</li> </ul> |
| | <ul> <li>Safety and tolerability parameters, including adverse events, study withdrawals due to AEs, vital signs assessments, and clinical laboratory assessments, for oral lead-in phase (Day 1 to Week 4).</li> </ul> |
| | <ul> <li>Injection discontinuation rate, the number and severity of ISRs and additional<br/>acceptability measures.</li> </ul> |

| Overview | Key | Elements of the RAP |
|---|---|---|
| | • | Evaluation of relationships between significant safety and tolerability parameters and CAB PK may be explored. |
| Study<br>Design | • | This will be an open label, non-randomized, single arm study. Participants will receive daily oral CAB (30mg tablets) for 4 weeks during the Oral Phase of the study and intramuscular (IM) injections of 600 mg of CAB LA at Week 5, Week 9, Week 17, Week 25 and Week 33. |
| | • | Starting at 8 weeks post last injection, participants will be seen once every 12 weeks for 48 weeks during the follow-up phase. |
| | • | Subjects who volunteer to participate in the intensive PK assessment will have serial blood sampling for measurement of plasma CAB concentrations following oral administration over a 24 h window starting on Day 27 and ending on Day 28 |
| | • | PK samples at trough for Oral Phase will be collected for all subjects prior to dose within 20 to 28 hours following oral administration the day prior; Intensive oral PK samples will be collected from approximately 16 participants. |
| | • | PK Samples for Injection Phase will be collected prior to CAB LA injections at Week 5, 9, 17, 25, and 33 with the exception of 1-week post injection samples at Weeks 6, 10, 18, 26, 34, 37 (4-week post injection sample) and Week 41 |
| | • | Long-term follow up PK samples will be collected at Week 53, 65, 77, and 89. |
| Planned<br>Analyses | • | The primary safety analysis and PK analyses including both oral phase and injection phase through Weeks 5 to 41 will be performed after all ongoing participants complete the Week 41 visit or withdraw from the study treatment, whichever comes first. |
| | • | The end of study analysis will be performed after all ongoing participants complete the Week 89 visit or withdraw from the study treatment, whichever comes first. |
| Analysis<br>Populations | • | The All Subjects Screened Population will include all subjects who consent to participate in the clinical study. Subjects in this population will be used for disposition summary |
| | • | The Safety Population will include all subjects who receive at least one dose of the study treatment. Subjects in this population will be used for all demographic and safety summaries or listings, as well as for the analysis of acceptability of CAB LA. |
| | • | Safety Injection Population will include all subjects received at least one CAB LA injection. Subjects in this population will be used to evaluate the safety and tolerability of CAB LA injection in primary analysis. |
| | • | Oral PK Population: subjects in the 'Safety population' for whom an intensive oral pharmacokinetic sample was obtained and analysed. PK samples that may |

| Overview | Key Elements of the RAP |
|---|---|
| | be affected by protocol deviations will be reviewed by the study team to determine whether or not the sample will be excluded. This population will be used for reporting of Oral PK data. |
| | <ul> <li>Injection (Week 41) PK Population: subjects in the 'Safety population' for whom<br/>an injection pharmacokinetic sample was obtained and analysed during Weeks<br/>5 to 41. PK samples that may be affected by protocol deviations will be<br/>reviewed by the study team to determine whether or not the sample will be<br/>excluded. This population will be used for reporting of Injection PK data from<br/>Weeks 5 to 41.</li> </ul> |
| | <ul> <li>Injection (Week 89) PK Population: subjects in the 'Safety population' for whom<br/>an injection pharmacokinetic sample was obtained and analysed during Weeks<br/>5 to 89. PK samples that may be affected by protocol deviations will be<br/>reviewed by the study team to determine whether or not the sample will be<br/>excluded. This population will be used for reporting of Injection PK data from<br/>Weeks 5 to 89.</li> </ul> |
| Hypothesis | No formal statistical hypotheses will be evaluated. |
| Primary<br>Analyses | To assess safety of CAB LA, the number and the percent of participants experiencing each safety endpoint will be tabulated including adverse events, clinical laboratory tests, study withdrawals due to AEs, and vital signs assessments. |
| | To assess tolerability of CAB LA, the proportion of participants who terminate from receiving injections prior to the full course due to AE, intolerability of injection, frequency of injections, or burden of procedures related to injections out of those participants that received at least one injection. |
| | To assess the plasma pharmacokinetics of CAB following repeat oral administration (Day 1 to Week 4) and CAB LA IM injections throughout the Injection Phase (Week 5 to Week 41). |
| Secondary<br>Analyses | To assess the plasma pharmacokinetics of CAB LA throughout the Injection and Long-term Follow-up Phases (Week 5 to Week 89). |
| | To assess the safety and tolerability of oral CAB, each safety and tolerability endpoint will be tabulated including adverse events, study withdrawals due to AEs, vital signs assessments and clinical laboratory assessments. |
| | To assess the acceptability of the CAB LA, injection discontinuation rate, the number and severity of ISRs, and the proportion (with 95% CI for the CAB LA arm) of participants who would consider using CAB LA for HIV prevention in the future will be tabulated among all enrolled participants (including those who terminated product use during the trial. |
| | Overall treatment satisfaction score and answers to each individual question on |

| Overview | Key Elements of the RAP |
|----------|----------------------------------------------------------|
| | HIV-PrevTSQc will be summarized to evaluate tolerability |

206898

## 2. SUMMARY OF KEY PROTOCOL INFORMATION

# 2.1. Changes to the Protocol Defined Statistical Analysis Plan

There were no changes or deviations to the originally planned statistical analysis specified in the protocol (Dated: 06/JUN/2018).

## 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| Evaluate the safety and tolerability of the injectable agent, cabotegravir (GSK1265744) long acting (CAB LA) injectable (600 mg dose administered every 4 weeks for 2 doses followed by every 8 weeks for 3 doses) through Week 5-41 in HIV-1 uninfected Chinese men. | Safety and tolerability parameters, including adverse events, clinical laboratory tests, study withdrawals due to AEs, vital signs assessments, and evaluation of injection site reactions (ISRs). |
| Evaluate the plasma pharmacokinetics of CAB following repeat oral administration (Day 1 to Week 4) and CAB LA IM injections throughout the Injection Phase (Week 5 to Week 41). | Plasma CAB AUC(0-τ), Cmax, Cτ, tmax, λz, t½, CL/F, and Vz/F at Week 4 following daily oral administration of CAB. Plasma CAB AUC(0-τ), Cmax, Cτ, and tmax at Week 41 following IM injections of CAB LA. |
| Secondary Objectives | Secondary Endpoints |
| Evaluate the plasma pharmacokinetics of CAB LA throughout the Injection and Longterm Follow-up Phases (Week 5 to Week 89) | Plasma CAB AUC(0- $\tau$ ), Cmax, C $\tau$ , tmax, $\lambda z$ , t½, CL/F, and Vz/F |
| Evaluate the safety and tolerability of oral CAB in HIV uninfected Chinese men during the oral lead-in Phase (Day 1 to Week 4) | Safety and tolerability parameters, including adverse events, study withdrawals due to AEs, vital signs assessments and clinical laboratory assessments. |
| Evaluate the acceptability of CAB LA injections through 41 weeks. | Injection discontinuation rate, the number and severity of ISRs and additional acceptability measures. |
| Explore concentration-effect relationships for various safety and tolerability parameters if relevant. | Evaluation of relationships between significant safety and tolerability parameters and CAB PK may be explored. |

206898

### 2.3. Study Design



### 2.4. Statistical Hypotheses

No formal statistical hypotheses will be evaluated. The study is designed to evaluate the PK, safety, tolerability, and acceptability of the injectable agent, CAB LA (600 mg dose administered at 8-week intervals after 2 initial doses 4 weeks apart) in HIV-uninfected men in China where at least 60% of the men are of a population who have sex with men.
206898

Where appropriate, an estimation approach will be taken, and point estimates and confidence intervals will be constructed.

206898

# 3. PLANNED ANALYSES

# 3.1. Interim Analyses

No formal interim analysis is planned in the study.

However, two preliminary PK analyses during the study will be performed in an informal manner. One will be after all planned participants complete the oral phase, and the other one will be after 50% of planned participants complete Week 17 visit. Study team will review preliminary safety and PK data.

# 3.2. Final Analyses

The primary safety analysis and PK analyses including both oral phase and injection phase through Weeks 5 to 41 will be performed after all ongoing participants complete the Week 41 visit and datasets have been authorized. Other secondary analyses as mentioned, where appropriate, will also be performed. The end of study analysis will be performed after all ongoing participants complete the Week 89 visit. All planned primary and secondary analyses will be included in the second formal analyses.

The planned analyses will be performed after the completion of the following sequential steps:

- a. All subjects have completed the specific study visit (i.e. week 41 or week 89) as defined in the protocol.
- b. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.

206898

# 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All Subjects<br>Screened | Comprise of all subjects who consent to participate in the clinical study. | Disposition summary |
| Safety | Comprise of all subjects who receive at least one dose of the study treatment. | <ul> <li>All demographic</li> <li>General safety analyses</li> <li>Safety analysis for the oral phase</li> <li>Analysis of acceptability of CAB LA</li> </ul> |
| Safety Injection | Comprise of all subjects received at<br>least one CAB LA injection | <ul> <li>Safety and tolerability<br/>analyses of CAB LA in<br/>primary and extended<br/>analyses</li> </ul> |
| Oral<br>Pharmacokinetic<br>(PK) | Will consist of all subjects in the 'Safety population' for whom an intensive oral pharmacokinetic sample was obtained and analysed. PK samples that may be affected by protocol deviations will be reviewed by the study team to determine whether or not the sample will be excluded. | <ul> <li>Oral PK Concentration</li> <li>Oral PK Parameters</li> </ul> |
| Injection (Week 41) Pharmacokinetic (PK) | Will consist of all subjects in the 'Safety population' for whom an injection pharmacokinetic sample was obtained and analysed during Weeks 5 to 41. PK samples that may be affected by protocol deviations will be reviewed by the study team to determine whether or not the sample will be excluded. | <ul> <li>Injection PK Concentration</li> <li>Injection PK Parameters</li> </ul> |
| Injection (Week 89) Pharmacokinetic (PK) | Will consist of all subjects in the 'Safety population' for whom an injection pharmacokinetic sample was obtained and analysed during Weeks 5 to 89. PK samples that may be affected by protocol deviations will be reviewed by the study team to determine whether or not the sample will be excluded. | <ul> <li>Injection PK Concentration</li> <li>Injection PK Parameters</li> </ul> |

# NOTES:

Please refer to Appendix 14: List of Data Displays which details the population to be used for each display being generated.

206898

# 4.1. Protocol Deviations

- Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.
- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.
  - o Data will be reviewed prior to freezing the database to ensure all important deviations are captured and categorised on the protocol deviations dataset.
  - This dataset will be the basis for the summaries and listings of protocol deviations.
- A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the eCRF.

206898

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Table 1 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 1 Overview of Appendices

| Section | Component |
|---|---|
| 10.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population |
| 10.2 | Appendix 2: Time & Events |
| 10.3 | Appendix 3: Assessment Windows |
| 10.4 | Appendix 4: Treatment States and Phases |
| 10.5 | Appendix 5: Data Display Standards & Handling Conventions |
| 10.6 | Appendix 6: Derived and Transformed Data |
| 10.7 | Appendix 7: Premature Withdrawals & Handling of Missing Data |
| 10.8 | Appendix 8: Values of Potential Clinical Importance |
| 10.9 | Appendix 9: Multicenter Studies |
| 10.10 | Appendix 10: Examination of Covariates, Subgroups & Other Strata |
| 10.11 | Appendix 11: Multiple Comparisons & Multiplicity |
| 10.12 | Appendix 12: Model Checking and Diagnostics for Statistical Analyses. |
| 10.13 | Appendix 13: Abbreviations & Trade Marks |
| 10.14 | Appendix 14: List of Data Displays |

206898

#### 6. STUDY POPULATION ANALYSES

# 6.1. Overview of Planned Analyses

The study population analyses will be based on the safety population, unless otherwise specified. All summary data and statistics are calculated from available data, unless otherwise specified.

Table 2 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 14: List of Data Displays.

Table 2 Overview of Planned Study Population Analyses

| Display Type | Data | Displays Gene | rated |
|---|---|---|---|
| | Table | Figure | Listing |
| Disposition | | | |
| Retention Rate and Reasons for Withdrawals | Υ | | Υ |
| Demography and Baseline Characteristics | | | |
| General Demographics Characteristics | Υ | | Υ |
| Medical History and Concomitant Medications | | | |
| Medical History | Υ | | Υ |
| Prior Medications | Υ | | Υ |
| Concomitant Medications | Υ | | Υ |
| Protocol Deviations | | | |
| Deviation of Inclusion/Exclusion Criteria | Y | | Υ |
| Important Protocol Deviations | Y | | Y |

#### NOTES:

• Y = Yes display generated.

# 6.1.1. Disposition

The reasons of screening failure will be summarized based on the screened population. The number and percentage of each reason will be tabulated.

A summary of subject disposition by phase will be provided, including the number and percentage of subjects entering oral/injection phase, the number and percentage of subjects completing oral/injection phase and the number and percentage of subjects withdrawing from oral/injection phase.

Subject disposition data will be presented in a listing.

# 6.1.2. Demographics

General demographics including age, self-identified gender when entering the study, and ethnicity will be summarized.

206898

A subject's age is calculated using the year part of informed consent form (ICF) – year of birth collected in CRF.

## 6.1.3. Medical History

Summaries of medical history will be presented by GSK pre-specified body system categories as collected in the eCRF. Number and percentage of subjects in each category will be tabulated.

#### 6.1.4. Prior and Concomitant Medications

Medications will be coded to therapeutic drug classes and generic drug names using the GSKDRUG 1.4 or later. Medications initiated prior to the Day 1 of the study will be counted as prior medications. Concomitant medications are defined as medications that are taken on or after the Day 1. Medications initiated prior to the Day 1 and continued after the Day 1 will be counted as both prior and concomitant medications.

Summaries showing the number and percentage of subjects who take prior or concomitant medications will be presented by therapeutic drug class and generic drug name.

#### 6.1.5. Protocol Deviation

Important protocol deviations (PD) will be summarized PD category and subcategory, and will also be presented in a listing. A separate summary table and a listing will be provided for subjects with deviation of the inclusion/exclusion criteria in the safety population

206898

# 7. PRIMARY STATISTICAL ANALYSES

# 7.1. Safety Analyses of CAB LA

Four study phases are defined for this study: screening phase, oral phase, injection phase and follow-up phase (see Appendix 4 for the definition of each phase).

The primary safety analysis will be conducted after all ongoing participants complete the Week 41 visit and datasets have been authorized. All data from injected participants collected from Week 5 to Week 41 (i.e., in the injection phase) will be analysed. Analysis endpoints will include Grade 2 or higher clinical and laboratory events that occur from the initial injection to 8 weeks after the last injection among participants who receive at least one injection.

The extended safety analysis will be conducted after all ongoing participants complete the Week 89 visit and datasets have been authorized. All data from injected participants collected from Week 5 to Week 89 (i.e., in the injection phase and the follow-up phase) will be analysed. Analysis endpoints are the same as in the primary safety analysis.

To assess safety, the number and the percent of participants experiencing each safety endpoint will be tabulated. Each participant will contribute once in each category (i.e., only for the highest severity AE) for the evaluation of safety.

# 7.1.1. Injection Site Reaction

The number and percentage of participants experiencing each type of injection site reaction sign or symptom will be tabulated by severity from the safety injection population. For a given sign or symptom, each participant's ISR will be counted once under the maximum severity for all injection visits. Overall summary of ISR and summary of ISR by needle length will both be provided. ISR related details, such as cardiovascular activity, strength training exercise, will be listed only.

Table 3 provides an overview of the planned ISR analyses, with full details of data displays being presented in Appendix 14: List of Data Displays.

206898

Table 3 Overview of Planned ISR Analyses

| Display Type | | Data Displays Generated | | | | | |
|---|---|---|---|---|---|---|---|
| | S | tats Analysis | 3 | Sum | mary | Individual | |
| | Т | F | L | T | F | F | L |
| ISR Analyses | | | | | | | |
| All ISR Symptoms | | | | Υ | | | Υ |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

#### 7.1.2. Adverse Events

Adverse events will be tabulated using MedDRA (v20.0 or above) system organ class (SOC) and preferred terms (PT), or preferred terms alone, by study phase. The number and percentage of participants experiencing each specific AEs (Grade 2 or higher, All AEs, SAEs, AEs leading to permanent treatment discontinuation or study withdrawal) will be tabulated. Number of subjects in the safety population who entered the study phase will be used as denominator in the calculation of percentages.

Drug-related AEs, SAEs, and Grade 2-4 AEs will also be tabulated. Any AE is assumed to be study treatment-related if relationship is marked 'YES' on CRF or value is missing. In addition, a summary table will be created for AEs by maximum severity by study phase. Common AEs are defined as AEs occurring in >=5% subjects during the study (based on preferred term). Common AEs, common non-serious AEs, common Grade 2-4 AEs, and common drug-related Grade 2-4 AEs will be tabulated.

All AE tables will be presented in a decreasing frequency order of SOC or PT unless otherwise specified.

Table 4 provides an overview of the planned AE analyses, with full details of data displays being presented in Appendix 14: List of Data Displays.

Table 4 Overview of Planned AE Analyses

| | Data Displays Generated | | | | | | |
|---|---|---|---|---|---|---|---|
| Display Type | S | tats Analysis | S | Sum | mary | Individual | |
| | T | F | L | T | F | F | L |
| AE Analyses | | | | | | | |
| All AEs | | | | Υ | | | Υ |
| Grade 2 or higher AEs | | | | Υ | | | Υ |
| SAEs | | | | Υ | | | Υ |
| AE leading to | | | | Υ | | | Υ |
| treatment | | | | | | | |

206898

| | Data Displays Generated | | | | | | |
|---|---|---|---|---|---|---|---|
| Display Type | S | tats Analysis | 3 | Sum | mary | Individual | |
| | T | F | Ш | Τ | F | F | L |
| discontinuation or | | | | | | | |
| study withdrawal | | | | | | | |
| Drug-related AEs | | | | Υ | | | |
| Drug-related SAEs | | | | Υ | | | |
| Drug-related Grade 2 | | | | Υ | | | |
| or higher AEs | | | | | | | |
| Common AEs | | | | Υ | | | |
| Common non-serious | | | | Υ | | | |
| AEs | | | | | | | |
| Common Grade 2-4 | | | | Υ | | | |
| AEs | | | | | | | |
| Common drug-related | | | | Υ | | | |
| Grade 2-4 AEs | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

# 7.1.3. Clinical Laboratory Tests

All clinical laboratory tests will be graded according to the Appendix 7 from the study protocol. Grade 2 or higher laboratory events will be tabulated by number and percentage of subjects with the event by study phase.

Change from baseline in hematology, fasting chemistry, fasting lipid profile, and coagulation profile will be summarized by visit. For the definition of baseline, refer to Section 10.5.2. Urinalysis and urine chemistry results will be summarized by visit as either categorical values or as continuous values, depending on the type of the parameter.

For each lab test, shift from baseline table will be provided based on toxicity grade, both by visit and for the shift to maximum toxicity grade in each study phase. Data collected at unscheduled visits will not be included in the by-visit summary, but will be used in the calculation of maximum grade in each study phase. Subjects having both high and low values will be counted in both High and Low categories for the summary by study phase.

All lab data, as well as lab data for subjects with Grade 2 or higher abnormalities, will be listed. Abnormal data will be listed with an indicator, which is low/high relative to normal range. All laboratory results from local labs, if any, will be listed only

Table 4 provides an overview of the planned lab test analyses, with full details of data displays being presented in Appendix 14: List of Data Displays.

206898

Table 5 Overview of Planned Lab Test Analyses

| | | Abs | olute | | С | hange fro | m Baselin | е |
|---|---|---|---|---|---|---|---|---|
| Display Type | Summary | | Indiv | idual | Sumi | mary | Individual | |
| | T | F | F | L | Т | F | F | L |
| Laboratory Test Analyses | | | | | | | | |
| Grade 2 or high | Υ | | | | | | | |
| laboratory events | | | | | | | | |
| Clinical Chemistry | | | | Υ | Υ | | | |
| Hematology | | | | Υ | Υ | | | |
| Fasting Lipid Profile | | | | Υ | Υ | | | |
| Coagulation Profile | | | | Υ | Υ | | | |
| Urinalysis and Urine | Υ | | | Υ | Υ | | | |
| Chemistry | | | | | | | | |
| Other lab data | | | | Υ | | | | |
| including local lab | | | | | | | | |

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

### 7.1.4. Vital Sign Assessments

Change from baseline in vital signs, including temperature, systolic and diastolic blood pressure, and pulse rate and respiratory rate will be summarized by study visit. For the definition of baseline, refer to Section 10.5.2. Shift from baseline table (with respect to clinical concern range) will also be provided.

All vital signs, as well as vital signs for subjects with abnormalities of potential clinical importance, will be listed with an indicator, which is low/high relative to clinical concern range.

Table 6 provides an overview of the planned vital sign analyses, with full details of data displays being presented in Appendix 14: List of Data Displays.

Table 6 Overview of Planned Vital Sign Analyses

| Display Type | | Abso | olute | | Change from Baseline | | | |
|---|---|---|---|---|---|---|---|---|
| | Summary | | Indiv | idual | Sumi | mary | Individual | |
| | T | F | F | L | Т | F | F | L |
| Vital Signs | Vital Signs | | | | | | | |
| Vital signs | | | | Υ | Υ | | | |

#### NOTES

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

206898

#### 7.1.5. Death

Both primary and secondary causes, if any, will be listed for each deceased participant.

Table 7 provides an overview of the planned death analyses, with full details of data displays being presented in Appendix 14: List of Data Displays.

Table 7 Overview of Planned Death Analyses

| | Data Displays Generated | | | | | | |
|---|---|---|---|---|---|---|---|
| Display Type | S | tats Analysis | 3 | Sum | mary | Individual | |
| | T | F L | | T F | | F | L |
| Death Analysis | Death Analysis | | | | | | |
| Death | | | | | | | Υ |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

# 7.2. Tolerability Analyses of CAB LA

The tolerability analyses will be based on the safety injection population, unless otherwise specified. All summary data and statistics are calculated from available data, unless otherwise specified.

To assess tolerability of CAB LA, the proportion (with 95% confidence interval) of participants who terminate from receiving injections prior to the full course due to AE, intolerability of injection, frequency of injections, or burden of procedures related to injections will be calculated out of those participants that received at least one injection.

A questionnaire will also be used to assess participant tolerability and satisfaction to the treatment. For each question, the responses will be summarized by the proportion of participants reporting the response out of all those that answered the question. An overall treatment satisfaction score will be calculated for each participant.

Total score is defined as the sum of the scores for individual questions. If less than or equal to 50% of the questions for an individual participant are missing, the missing total scores will be estimated using the average of the existing questions multiplied by twelve; if more than 50% of the questions for an individual participant are missing, the total score will not be estimated and will be considered as missing. When calculating total scores,

question will be used and question ccl will be used and question ccl will be excluded.

206898

Table 8 provides an overview of the planned tolerability analyses, with further details of data displays being presented in Appendix 14: List of Data Displays.

Table 8 Overview of Planned Tolerability Analyses

| | Data Displays Generated | | | | | | |
|---|---|---|---|---|---|---|---|
| Display Type | S | tats Analysis | 3 | Sum | mary | Individual | |
| | Т | F | L | T | F | F | L |
| <b>CAB LA Discontinuat</b> | CAB LA Discontinuation | | | | | | |
| Injection | | | | Y | | | Υ |
| Discontinuation Rate | | | | | | | |
| Treatment Satisfaction | n Questio | nnaire | | | | | |
| Each question in the | | | | Υ | | | Υ |
| questionnaire | | | | | | | |
| Treatment total | | | | Υ | | | Y |
| satisfaction score | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data

# 7.3. Primary Pharmacokinetic Analyses

# 7.3.1. Overview of Planned Primary Pharmacokinetic Analyses

The primary pharmacokinetic (PK) analyses will be based on the Oral PK and Injection (Week 41) PK populations, unless otherwise specified.

Table 9 provides an overview of the planned efficacy analyses, with full details of data displays being presented in Appendix 14: List of Data Displays.

Table 9 Overview of Planned Primary Pharmacokinetic Analyses

| Display Type | | Untransformed | | | | | | | Log-Transformed | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stats Analysis | | Summary Individual | | Stats Analysis | | Summary | | Individual | | | | | |
| | Τ | F | L | Т | F | F | L | Т | F | L | Т | F | F | L |
| Oral/Injection | | | | | | | | | | | | | | |
| PK Concentrations | | | | Υ | <b>Y</b> [1] | <b>Y</b> [1] | Υ | | | | | | | |
| Plasma PK Parameters | Υ | | | Υ | | | Υ | _ | | Υ | Υ | | | |

#### NOTES

- T = Table, F = Figure, L = Listings, Y = Display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

<sup>[1]</sup> Linear and Semi-Logarithmic plots will be created on the same display.

206898

# 7.3.2. Primary Drug Concentration Measures

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 10.5.3 Reporting Process & Standards).

# 7.3.3. Primary Pharmacokinetic Parameters

#### 7.3.3.1. Deriving Primary Pharmacokinetic Parameters

- Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 10.5.3 Reporting Process & Standards).
- The pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using Phoenix WinNonlin Version 6.4 or higher.
- All calculations of non-compartmental parameters will be based on actual sampling times, and all concentrations will be included in the estimation of PK parameters regardless of whether samples are collected within the specified time window or not.
- Pharmacokinetic parameters described in Table 10 will be determined from the plasma concentration-time data, as data permits.

206898

Table 10 Derived Primary Pharmacokinetic Parameters

| Parameter | Parameter Description |
|---|---|
| AUC(0-τ) | Area under the concentration-time curve over the dosing interval will be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. |
| Cmax | Maximum observed concentration, determined directly from the concentration-time data. |
| tmax | Time to reach Cmax, determined directly from the concentration-time data. |
| Сτ | Observed concentration at the end of the dosing interval, determined directly from the concentration-time data. |
| t½ | Terminal absorption elimination half-life will be calculated as: $t\frac{1}{2} = \ln 2 / \lambda z$ |
| λz | Terminal absorption elimination rate constant |
| CL/F | Clearance (adjusted for bioavailability, F) will be calculated as: $CL/F = Dose \ / \ AUC(0-\tau)$ |
| Vz/F | Volume of distribution (adjusted for bioavailability, F) will be calculated as: $Vz/F = CL \ / \ \lambda z$ |

#### NOTES:

- · Additional parameters may be included as required.
- λz, CL/F, Vss and t½ will be determined for the Oral PK population only in the primary analysis; these
  parameters will be further explored for the Injection (Week 89) PK population (Section 8.1.3.1).

#### 7.3.3.2. Statistical Analysis of Primary Pharmacokinetic Parameters

The following pharmacokinetic statistical analyses will only be performed, if sufficient data is available (i.e. if subjects have well defined plasma profiles).

# Pharmacokinetic Statistical Analyses

#### Endpoint(s)

• Plasma primary PK endpoints include  $C\tau$ , as data permit

# **Model Specification**

Assessment of Accumulation (Injection Phase only):

To determine accumulation of plasma CAB following treatment with CAB LA, the log-transformed Cτ values for CAB will be analyzed using a mixed effects model (ANOVA) as appropriate to the study design, fitting fixed effect terms for visit and treating subject as a random effect. Point estimates and 90% confidence intervals (CIs) for the differences of interest (i.e. accumulation of CAB based on AUC(0-τ): Week 34 / Week 6) will be constructed using the residual variance.

Attainment of Steady state (Injection Phase only):

If data permit, a statistical analysis of steady-state trough concentrations (Cτ) will be performed

206898

# **Pharmacokinetic Statistical Analyses**

after log-transformation of  $C_{\tau}$  on Weeks 17, 25, 33, and 41 to evaluate whether steady state was achieved using the Helmert transformation approach. A mixed effect model (ANOVA) will be fitted by visit (as a categorical covariate) as a fixed effect term and subject as a random effect term. The comparison will begin with Week 17 vs. the average of Weeks 25 through Week 41. If the p-value for Week 17 vs. the average of Week 25 through Week 41 comparison is  $\leq$ 0.05 (i.e. steady state not achieved at Week 17), then the comparison will continue with Week 25 vs. Week 33 through Week 41.

# **Model Checking & Diagnostics**

Refer to Appendix 12: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

- Statistical analysis of accumulation of plasma CAB following treatment with CAB LA will be presented in tabular format with geometric mean ratios between Week 34 and Week 6, and 90% CIs for the ratios of  $C\tau$  for CAB.
- In steady-state analysis, the ratio of Geometric LS means and its 95% CI will be presented for the comparison(s).

206898

#### 8. SECONDARY STATISTICAL ANALYSES

# 8.1. Secondary Pharmacokinetic Analyses

# 8.1.1. Overview of Planned Secondary Pharmacokinetic Analyses

The secondary pharmacokinetic (PK) analyses will be based on the Injection (Week 89) PK population, unless otherwise specified.

Table 11 provides an overview of the planned analyses, with full details being presented in Appendix 14: List of Data Displays.

Table 11 Overview of Planned Secondary Pharmacokinetic Analyses

| Display Type | | Untransformed | | | | Log-Transformed | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stat | Stats Analysis | | Summary Individual | | idual | Stats Analysis | | Summary | | Individual | | | |
| | T | F | L | Т | F | F | L | Т | F | L | Т | F | F | L |
| Oral/Injection | Oral/Injection | | | | | | | | | | | | | |
| PK Concentrations | | | | Υ | <b>Y</b> [1] | <b>Y</b> [1] | Υ | | | | | | | |
| Plasma PK Parameters | Υ | | | Υ | | | Υ | | | Υ | Υ | | | |

#### NOTES:

- T = Table, F = Figure, L = Listings, Y = Display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

#### 8.1.2. Secondary Drug Concentration Measures

Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 10.5.3 Reporting Process & Standards).

# 8.1.3. Secondary Pharmacokinetic Parameters

# 8.1.3.1. Deriving Secondary Pharmacokinetic Parameters

- Refer to Appendix 5: Data Display Standards & Handling Conventions (Section 10.5.3 Reporting Process & Standards).
- The pharmacokinetic parameters will be calculated by standard non-compartmental analysis according to current working practices and using Phoenix WinNonlin Version 6.4 or higher.
- All calculations of non-compartmental parameters will be based on actual sampling times, and all concentrations will be included in the estimation of PK parameters regardless of whether samples are collected within the specified time window or not.

<sup>[1]</sup> Linear and Semi-Logarithmic plots will be created on the same display.

206898

• Pharmacokinetic parameters described in Table 12 will be determined from the plasma concentration-time data, as data permits.

Table 12 Derived Secondary Pharmacokinetic Parameters

| Parameter | Parameter Description |
|---|---|
| AUC(0-τ) | Area under the concentration-time curve over the dosing interval will be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. |
| Cmax | Maximum observed concentration, determined directly from the concentration-time data. |
| tmax | Time to reach Cmax, determined directly from the concentration-time data. |
| Сτ | Observed concentration at the end of the dosing interval, determined directly from the concentration-time data. |
| t½ | Terminal absorption elimination half-life will be calculated as: $t\frac{1}{2} = \ln 2 / \lambda z$ |
| λz | Terminal absorption elimination rate constant |
| CL/F | Clearance (adjusted for bioavailability, F) will be calculated as: $ CL/F = Dose \ / \ AUC(0-\tau) $ |
| Vz/F | Volume of distribution (adjusted for bioavailability, F) will be calculated as: $Vz/F = CL \ / \ \lambda z$ |

#### NOTES:

Additional parameters may be included as required.

# 8.2. Safety and Tolerability Analyses of Oral CAB

The safety and tolerability analyses of oral CAB will include Grade 2 or higher clinical and laboratory events occurred during the oral phase. Analysis time frame is from the first date of taking oral CAB tablet to the date right before the first CAB LA injection. For subjects who withdraw treatment from the oral phase, the analysis will include all safety and tolerability assessments from the first date of taking oral CAB tablet up to the date of last study visit.

Safety endpoints including adverse events, laboratory test, vital signs, and death will be analysed. The same analysis approaches will be conducted as in the primary analysis, but with different time frame.

Table 13 provides an overview of the planned analyses, with full details of data displays being presented in Appendix 14: List of Data Displays.

206898

Table 13 Overview of Planned AE, LB, VS, and Death Analyses

| | Data Displays Generated | | | | | | |
|---|---|---|---|---|---|---|---|
| Display Type | S | tats Analysis | S | Sum | mary | Indiv | ridual |
| | Т | F | L | T | F | F | L |
| AE Analyses | | | | | | | |
| All AEs | | | | Υ | | | Υ |
| Grade 2 or higher AEs | | | | Υ | | | Υ |
| SAEs | | | | Υ | | | Υ |
| AE leading to | | | | Υ | | | Υ |
| treatment | | | | | | | |
| discontinuation or | | | | | | | |
| study withdrawal | | | | | | | |
| Drug-related AEs | | | | Υ | | | |
| Drug-related SAEs | | | | Υ | | | |
| Drug-related Grade 2 | | | | Y | | | |
| or higher AEs | | | | | | | |
| Common AEs | | | | Υ | | | |
| Common non-serious<br>AEs | | | | Y | | | |
| Common Grade 2-4 | | | | Υ | | | |
| AEs | | | | | | | |
| Common drug-related | | | | Υ | | | |
| Grade 2-4 AEs | | | | | | | |
| Laboratory Tests | | | | | | | |
| Grade 2 or higher | | | | Υ | | | |
| laboratory events | | | | | | | |
| Clinical Chemistry | | | | Υ | | | Υ |
| Hematology | | | | Υ | | | Υ |
| Fasting Lipid Profile | | | | Υ | | | Υ |
| Urinalysis | | | | Y | | | Υ |
| Coagulation Profile | | | | Υ | | | Υ |
| Other lab data | | | | | | | Υ |
| including local lab | | | | | | | |
| Vital Sign Analysis | | | | | | | |
| Vital Signs | | | | Υ | | | Υ |
| Death Analysis | 1 | 1 | | 1 | , | , | , |
| Death | | | | | | | Υ |

# NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

206898

# 8.3. Acceptability of CAB LA

The secondary acceptability analyses will be based on safety population, unless otherwise specified. All summary data and statistics are calculated from available data, unless otherwise specified.

To assess acceptability of the CAB LA, the proportion (with 95% confidence interval) of participants who would consider using CAB LA for HIV prevention in the future will be calculated among all subjects in the safety population (including those who terminated product use during the trial). Participants will be asked if they would consider using CAB LA for HIV prevention in the future at their Week 41 visit or at their withdrawal visit, whichever occurs first. Patients who are lost to follow up or with missing responses will be presented as such in a separate category.

Table 14 provides an overview of the planned acceptability analyses, with further details of data displays being presented in Appendix 14: List of Data Displays.

Table 14 Overview of Planned Acceptability Analyses

| | Data Displays Generated | | | | | | |
|---|---|---|---|---|---|---|---|
| Display Type | S | tats Analysis | 3 | Summary | | Individual | |
| | T | F | L | T | F | F | L |
| Acceptability of the CAB LA | | | | | | | |
| participants who | | | | Υ | | | Υ |
| would consider using | | | | | | | |
| CAB LA | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

# 8.4. Concentration-effect Relationships for Safety and Tolerability Parameters

Evaluation of relationships between significant safety and tolerability parameters and CAB PK may be explored.

# 8.5. General Safety Analyses

This section will describe safety analyses that are not mentioned in Section 7.1 or Section 8.2, but usually are performed as safety assessment.

206898

# 8.5.1. Extent of Exposure to CAB

Duration of exposure to CAB and cumulative dose (see Section 10.6.2 for the definition) will be summarized for the oral phase and the injection phase separately. Overall exposure to the study drug and to the study (for safety evaluation) will also be calculated and summarized. Exposure data will also be listed.

Table 15 provides an overview of the planned analyses, with full details of data displays being presented in Appendix 14: List of Data Displays.

206898

Table 15 Overview of Planned Analyses for Extent of Exposure

| | Data Displays Generated | | | | | | |
|---|---|---|---|---|---|---|---|
| Display Type | S | tats Analysis | S | Sum | mary | Individual | |
| | Т | F | L | T F | | F | L |
| Extent of Exposure | | | | | | | |
| Extent of exposure | | | | Υ | | | Υ |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

# 8.5.2. Possible suicidality-related Adverse Events

Possible suicidality-related will be listed.

Table 16 provides an overview of the planned analyses, with full details of data displays being presented in Appendix 14: List of Data Displays.

Table 16 Overview of Analyses for possible suicidality-related AEs

| | Data Displays Generated | | | | | | |
|---|---|---|---|---|---|---|---|
| Display Type | S | tats Analysis | S | Summary | | Individual | |
| | T | F | L | T | F | F | L |
| AE Analyses | AE Analyses | | | | | | |
| Possible Suicidality- | | | | | | | Υ |
| Related Adverse Event | | | | | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

#### 8.5.3. Social Harms

Details of social harms collected on the eCRF will be listed for each participant.

Table 17 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 14: List of Data Displays.

206898

Table 17 Overview of Planned Study Population Analyses

| Display Type | Data | Data Displays Generated | |
|------------------|-------|-------------------------|---------|
| | Table | Figure | Listing |
| Social Harms | | | |
| All Social Harms | | | Υ |

#### NOTES:

• Y = Yes display generated.

#### 8.5.4. ECG

ECG test will be performed at Screening only. Details collected on the eCRF will be listed for each subject. Baseline ECG findings (normal, abnormal – not clinically significant, or abnormal - clinically significant) will be summarized by number and percentage of subjects and presented as part of the 'Demographic Characteristics' table.

Table 18 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 14: List of Data Displays.

Table 18 Overview of Planned Study Population Analyses

| Display Type | Data Displays Generated | | |
|---|---|---|---|
| | Table | Figure | Listing |
| ECG | | | |
| ECG Parameters and Results | Y | | Υ |

#### NOTES:

• Y = Yes display generated.

# 8.5.5. Cardiovascular Events

Any cardiovascular events will be listed only.

Table 19 provides an overview of the planned cardiovascular event analyses, with full details of data displays being presented in Appendix 14: List of Data Displays.

Table 19 Overview of Planned Cardiovascular Event Analyses

| | Data Displays Generated | | | | | | |
|---|---|---|---|---|---|---|---|
| Display Type | S | tats Analysis | 3 | Sum | mary | Individual | |
| | T | F | L | T F | | F | L |
| CV Event Analyses | | | | | | | |
| All CV events | | | | | | | Υ |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.

206898

| | Data Displays Generated | | | | |
|---|---|---|---|---|---|
| Display Type | Stats Analysis | Sum | mary | Individual | |
| | T F L | T | F | F | L |

• Individual = Represents FL related to any displays of individual subject observed raw data.

#### 8.5.6. Liver Events

Number and percentage of subjects with liver events will be tabulated by study phase. Number and percentage of subjects with clinical significant hepatobiliary laboratory abnormalities during the study will also be tabulated. Full information of liver events will be listed.

Table 20 provides an overview of the planned liver event analyses, with full details of data displays being presented in Appendix 14: List of Data Displays.

Table 20 Overview of Planned Liver Event Analyses

| | Data Displays Generated | | | | | | |
|---|---|---|---|---|---|---|---|
| Display Type | S | Stats Analysis | S | Sum | mary | Individual | |
| | T | F | L | T | F | F | L |
| Liver Event Analyses | | | | | | | |
| All liver events | | | | Υ | | | Υ |
| Hepatobiliary | | | | Υ | | | |
| laboratory | | | | | | | |
| abnormalities | | | | | | | |

# NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

206898

# 9. REFERENCES

Dube MP, Stein JH, Aberg JA, Fichtenbaum CJ, Gerber JG, Tashima KT et al. Guidelines for the evaluation and management of dyslipidemia in human immunodeficiency virus (HIV)-infected adults receiving antiretroviral therapy: recommendations of the HIV Medical Association of the Infectious Disease Society of America and the Adult AIDS Clinical Trials Group. Clin Infect Dis 2003; 37(5):613-27.

GlaxoSmithKline Document Number 2016N293702\_00 (Original – 20-JUL-2017): An Open Label, Phase 1 Study to Evaluate the PK, Safety, Tolerability and Acceptability of Long Acting Injections of the HIV Integrase Inhibitor, Cabotegravir (CAB; GSK1265744) in HIV Uninfected Chinese Men (20-JUL-2017)

Levey AS, Stevens LA, Schmid CH, Zhang YL, Castro AF, Feldman HI, et.al. A new equation to estimate glomerular filtration rate. Ann Int Med. 2009; 150: 604-12.

206898

# 10. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 4 | : Analysis Populations |
| Section 10.1 | Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population |
| RAP Section 5 | : General Considerations for Data Analyses & Data Handling Conventions |
| Section 10.2 | Appendix 2: Time and Events |
| Section 10.3 | Appendix 3: Assessment Windows |
| Section 10.4 | Appendix 4: Treatment States & Phases |
| Section 10.5 | Appendix 5: Data Display Standards & Handling Conventions |
| | Study Treatment & Sub-group Display Descriptors |
| | Baseline Definitions & Derivations |
| | Reporting Process & Standards |
| Section 10.6 | Appendix 6: Derived and Transformed Data |
| | General, Study Population & Safety |
| Section 10.7 | Appendix 7: Premature Withdrawals & Handling of Missing Data |
| | Premature Withdrawals |
| | Handling of Missing Data |
| Section 10.8 | Appendix 8: Values of Potential Clinical Importance |
| Section 10.9 | Appendix 9: Multicentre Studies |
| Section 10.10 | Appendix 10: Examination of Covariates and Subgroups & Other Strata |
| Section 10.11 | Appendix 11: Multiple Comparisons and Multiplicity |
| Section 10.12 | Appendix 12: Model Checking and Diagnostics for Statistical Analyses |
| Other RAP App | endices |
| Section 10.13 | Appendix 13: Abbreviations & Trade Marks |
| Section 10.14 | Appendix 14: List of Data Displays |

206898

# 10.1. Appendix 1: Protocol Deviation Management and Definitions for Per Protocol Population

Protocol waivers or exemptions are not allowed with the exception of immediate safety concerns that may arise after the oral administration of CAB.

Deviations from inclusion and exclusion criteria are not allowed because they can potentially jeopardize the scientific integrity of the study, regulatory acceptability or participant safety. Therefore, adherence to the criteria as specified in the protocol is essential

# 10.1.1. Exclusions from Per Protocol Population

Not applicable. Per protocol population is not defined in this study.

206898

# 10.2. Appendix 2: Time & Events

# 10.2.1. Protocol Defined Time & Events

# Table 21 Schedule of Activities<sup>q</sup>

| Clinical Assessments | Screeninga | Oral P | hase <sup>m</sup> | Injection | on P | hase | | | | | | | | | | | | Follow-<br>& Final | up Phase<br>Visit |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Day 1 | Day 28 (Week 4) | Day 35 (Week 5)<br>Injection 1 | Day 42 (Week 6) | Week 9<br>Injection 2 | Week 10 | Week 17 | Week 18 | Week 25 | Injection 4 | Week 26 | Week 33 | Injection 5 | Week 34 | Week 37 | Week 41 | Week 53, 65, 77 | Week 89 |
| Written informed consent | Χ | | | | | | | | | | | | | | | | | | |
| Inclusion/Exclusion criteria <sup>b</sup> | Х | | | | | | | | | | | | | | | | | | |
| Demographic information | Χ | | | | | | | | | | | | | | | | | | |
| Full physical exam/medical history <sup>C</sup> | X | | | | | | | | | | | | | | | | | | X |
| Brief physical exam | | Χ | Χ | Χ | Х | Χ | Х | Х | Х | Χ | | Χ | Χ | ) | Χ | | Χ | | |
| Height/weight/BMI <sup>d</sup> | Χ | | | | | | | | | | | | | | | | | | X |
| Medication/drug/alcohol history | Χ | | | | | | | | | | | | | | | | | | |
| HIV counseling | Χ | Χ | Χ | Χ | | Χ | Χ | Χ | Х | Χ | | Χ | Χ | ) | Χ | Χ | Χ | Χ | Х |
| Offer condoms and lubricant | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | | Χ | X | ) | X | Χ | Χ | Χ | Χ |
| Dispense oral study medication (with counseling) <sup>e</sup> | | X | | | | | | | | | | | | | | | | | |
| Drug accountability (pill counts) | | Χ | Χ | | | | | | | | | | | | | | | | |

206898

| Clinical Assessments | Screening <sup>a</sup> | Oral<br>Phas | e <sup>m</sup> | Injection | Phase | e | | | | | | | | | | Follov<br>Phase<br>& Fina<br>Visit | е . |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Day 1 | Day 28 (Week 4) | Day 35 (Week 5)<br>Injection 1 | Day 42 (Week 6) | Week 9<br>Injection 2 | Week 10 | Week 17<br>Injection 3 | Week 18 | Week 25<br>Injection 4 | Week 26 | Week 33<br>Injection 5 | Week 34 | Week 37 | Week 41 | Week 53, 65, 77 | Week 89 |
| CAB LA Injection (with counseling) | | | | Х | | X | | X | | Χ | | X | | | | | |
| HIV-PrevTSQc <sup>f</sup> | | | | | | | Χ | | | | | | | | | | |
| ISR AE Diary <sup>g</sup> | | | | X | | Х | | Х | | Χ | | Х | | | | | |
| AE | | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Χ | Х | Χ | Χ | Χ | Χ | Χ |
| SAE review (SAE will be collected from the signing of ICF) | X | X | X | Х | Х | Х | Χ | X | X | X | X | Х | X | X | X | | X |
| Concomitant medication check | | Χ | Χ | X | Χ | Х | Χ | Х | Χ | X | Χ | X | Χ | Χ | Χ | Χ | Χ |
| Vital signs <sup>h</sup> | Χ | Χ | | X | Χ | Х | Χ | Х | Χ | X | Χ | X | Χ | Χ | Χ | Χ | Χ |
| Qualitative HIV RNA by NAAT <sup>i</sup> | Χ | | | | | | | | | | | | | | | | |
| HIV PoC test <sup>j</sup> | Χ | Χ | | Χ | | Χ | | Χ | | Χ | | Χ | | | Χ | Χ | Χ |
| ECG <sup>k</sup> | Χ | | | | | | | | | | | | | | | | |
| HbsAg and HbsAb, HCV Antibody | Х | | | | | | | | | | | | | | | | |
| Hematology/Chemistry testing | Χ | Χ | Χ | X | Χ | X | | X | | X | | X | | | Χ | | Χ |
| Urinalysis | Χ | | | | | | | | | | | | | | Χ | | |
| Urine screen for Chlamydia and gonorrhea | X | | | | | | | | | | | | | | | | |
| Liver Chemistry Tests <sup>I</sup> | | | | | | | | _ | | | | | | | | Χ | |

206898

| Clinical Assessments | Screening <sup>a</sup> | Oral In<br>Phase <sup>m</sup> | | Injection | njection Phase | | | | | | | | | | | Follow- up<br>Phase<br>& Final<br>Visit | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Day 1 | Day 28 (Week 4) | Day 35 (Week 5)<br>Injection 1 | Day 42 (Week 6) | Week 9<br>Injection 2 | Week 10 | Week 17<br>Injection 3 | Week 18 | Week 25<br>Injection 4 | Week 26 | Week 33<br>Injection 5 | Week 34 | Week 37 | Week 41 | Week 53, 65, 77 | Week 89 |
| Fasting lipid profile | | Χ | | | | | | | | | | | | | X | | |
| Coagulation testing | Χ | | | | | | | | | | | | | | Χ | | |
| TRUST for Syphilis screen | Χ | | | | | | | | | | | | | | | | |
| Plasma for CAB concentration <sup>m,n,o</sup> | | | Χm | X | Χ | Х | Х | X | Χ | X | X | X | Х | X | Χ | Х | Х |
| Plasma storage sample <sup>p</sup> | Χ | Χ | Χ | Х | Χ | Χ | Χ | Х | Χ | X | Χ | X | X | Χ | Χ | Χ | Χ |

AE: Adverse events, BMI: Body mass index, CAB: Cabotegravir, CAB LA: Cabotegravir long-acting, ECG: Electrocardiogram, HbsAg: Hepatitis B surface antigen, HIV: Human Immunodeficiency Virus, HCV: Hepatitis C Virus, ISR: Injection site reactions, SAE: Serious adverse event, HIV-PrevTSQc: HIV-Prevention Treatment Satisfaction Questionnaire (change): TRUST: Toluidine Red Unheated Serum Test, RNA: Ribonucleic acid.

- a. Screening (including drug screen) is to be performed within 30 days of the first dose in the Oral Phase of the study. See Appendix 2 from the study protocol
- b. Inclusion/exclusion criteria will be fully assessed at the Screening visit. Changes between the screening visit and the Day 1 visit should be assessed to ensure eligibility, including additional assessments performed at Day 1.
- c. A full physical exam will be performed at Week 89.
- d. Weight will be collected at Screening and at Week 89. Height and BMI will be collected at Screening only.
- e. Oral phase consists of 28 days with a 7 day washout period between Day 28 (last oral dose) and Day 35 (first injection visit).
- f. HIV-PrevTSQc: HIV-Prevention Treatment Satisfaction Questionnaire (change) will be given at Week 10 only (after 2<sup>nd</sup> injection).
- g. ISR AE 7 Day Post Injection Diary will be distributed at the injection visit at Week 5, 9, 17, 25 and 33 and returned to the clinic at weeks 6, 10, 18, 26, and 34. For participants having ISR on the last day of week 5, 9, 17, 25 and 33, additional ISR AE Weeks 2 12 Post Injection Diary will be distributed at weeks 6,10, 18, and 26,34. Participants will be asked to bring the diary to each clinic visit.
- h. Vital sign measurements will be performed following 5 minutes of rest.
- i. Qualitative HIV Nucleic Acid Amplification Testing (NAAT) will be performed at Screening. See Appendix 9 from the study protocol for the HIV testing algorithm at screening, Day 1 and during the course of the study.

206898

- j. HIV PoC (Point of care) test will be performed at each time point during the course of the study and must be reviewed prior to IM dosing. See Appendix 9 from the study protocol for the HIV testing algorithm at screening, Day 1 and during the course of the study.
- k. ECGs will be performed following 5 minutes of rest in a semi-supine position.
- I. Liver Chemistry Tests include Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), Bilirubin total and direct.
- m. Oral Pharmacokinetic (PK) sampling at trough will be collected for all subjects prior to dose within 20 to 28 hours following oral administration the day prior. Intensive oral PK sampling will be collected from approximately16 participants as shown in Table 20.
- n. PK sampling for Injection phase: All PK samples will be collected prior to CAB LA injections at Week 5, 9, 17, 25, and 33 with the exception of 1-week post injection samples at Weeks 6, 10, 18, 26, 34, 37 (2-week post injection sample) and Week 41
- o. Long-term follow up PK samples: PK sampling during follow up will occur at, Week 53, 65, 77, and 89.
- p. Additional testing is required for participants who have a reactive or positive HIV test after enrolment. Stored plasma from the visit previous to the positive test should be tested for HIV using the 4th generation HIV test to best estimate time of infection. HIV acquisition must be confirmed by either western blot, HIV ½ Multispot or the Geenius HIV Confirmation ½ Assay, and HIV RNA.
- q. Visit may occur in a window ±3 Day

Table 22 Schedule of Intensive Oral PK (Approximately 16 Participants) a,b

| | Day 25 | Day 26 | Day 27 | | | | | | | Day 28 | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | Check-<br>in | Oral dose<br>administered<br>(e.g. 8AM) | dose (e.g. | administered<br>(e.g. 8AM) | hour post<br>dose (e.g. | post dose<br>(e.g. | post dose<br>(e.g. | post dose<br>(e.g.<br>12AM) | hour<br>post | hour post<br>dose (e.g. | Oral dose<br>administered<br>(e.g. after 8<br>AM) |
| Plasma for<br>CAB<br>concentration | | | X | | X | X | X | X | X | X | |

- a. PK sampling may occur ±15min
- b. Central lab tests for the intensive oral PK subjects refer to Table 21.

206898

# 10.3. Appendix 3: Assessment Windows

# 10.3.1. Assessment Windows

The nominal visit information collected on CRF will be used in the analysis. Analysis visit based on the time window will not be defined in this study.

206898

# 10.4. Appendix 4: Study Phase and State

# 10.4.1. Treatment Phases

Assessments and events will be classified according to the time of occurrence relative to the start date of study treatment.

| Treatment Phase | Definition |
|---|---|
| Screening Phase | Date < Date of first Oral CAB |
| Oral Phase | Date of First Oral CAB <= Date <= Date of First CAB LA Injection -1 day; for subjects who discontinued before receiving CAB LA Injection, the end date of the oral phase is the date of last study visit. |
| Injection Phase | Date of First CAB LA Injection <= Date <= 8 weeks after Last CAB LA Injection |
| Follow-up Phase | Date > 8 weeks after Last CAB LA Injection |

#### 10.4.2. Treatment States

Assessments and events will be classified according to time of occurrence relative to the start date of the study treatment.

# 10.4.2.1. Treatment States for AE Data

| Treatment State | Definition |
|---|---|
| Screening Phase | AE Start Date < Date of First Oral CAB |
| On-Oral CAB-<br>Treatment | Day 1 ≤ AE Start Date ≤ Date of First CAB LA Injection – 1;<br>for subjects who withdraw from oral CAB treatment, Day 1 ≤ AE Start Date ≤<br>Withdrawal date + 7 days |
| On-CAB LA-<br>treatment | Date of First CAB LA Injection ≤ AE Start Date ≤ Date of Week 41 Visit; for subjects who withdraw from CAB LA injection, Date of First CAB LA Injection ≤ AE Start Date ≤ Date of Last CAB LA Injection + 8 Weeks |
| Post-Treatment | AE Start Date > Date of Last CAB LA Injection + 8 weeks |
| Onset Time Since<br>1st Dose (Days) | If Date of First Oral CAB (or CAB LA injection) >AE Onset Date, duration = AE Onset Date - Treatment Start Date |
| | If Date of First Oral CAB (or CAB LA injection) ≤ AE Onset Date, duration = AE Onset Date - Treatment Start Date +1 Missing otherwise. |
| AE Duration<br>(Days) | AE Resolution Date – AE Onset Date + 1 |
| Drug-related | If relationship is marked 'YES' on CRF OR value is missing |

206898

# 10.5. Appendix 5: Data Display Standards & Handling Conventions

# 10.5.1. Study Treatment & Sub-group Display Descriptors

| | Treatment Group Descriptions | | |
|---|---|---|---|
| | Study Group Data Displays for Reporting | | |
| Code | Description | Description | Order [1] |
| Α | CAB PO 30 mg QD | CAB 30 mg | 1 |
| В | CAB LA IM 600 mg Q8W | CAB LA 600 mg | 2 |

#### NOTES:

#### 10.5.2. Baseline Definition & Derivations

#### 10.5.2.1. Baseline Definitions

The baseline or pre-dose assessment is the last available assessment prior to the time of the first dose unless it is specified otherwise.

#### 10.5.2.2. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|---|---|
| Change from Baseline | = Post-Dose Visit Value – Baseline |
| % Change from Baseline | = 100 x [(Post-Dose Visit Value – Baseline) / Baseline] |
| Maximum Change from Baseline | = Calculate the change from baseline at each given timepoint and determine the maximum change |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 10.5.2.1 Baseline Definitions will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.
- The baseline definition will be footnoted on all change from baseline displays.

#### 10.5.3. Reporting Process & Standards

# Software The currently supported versions of SAS software 9.2 or higher and Phoenix WinNonlin will be used.

#### **Analysis Datasets**

- Analysis datasets will be created according to CDISC standards SDTMIG v3.2 & ADaMIG v1.0
- For creation of ADaM datasets (ADCM/ADAE), the same version of dictionary datasets will be implemented for conversion from SI to SDTM.

<sup>1.</sup> Order represents treatments being presented in TFL, as appropriate.

206898

# **Reporting Process**

#### **Generation of RTF Files**

RTF files will be generated for the TLFs. But only compiled PDF file will be used in the delivery.

#### **Reporting Standards**

#### General

- The current GSK Integrated Data Standards Library (IDSL) will be applied for reporting, unless otherwise stated:
  - 4.03 to 4.23: General Principles
  - o 5.01 to 5.08: Principles Related to Data Listings
  - o 6.01 to 6.11: Principles Related to Summary Tables
  - 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the actual treatment the subject received unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places (DP's) will be adopted for reporting of data based on the raw data collected.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's

#### **Planned and Actual Time**

- Reporting for tables, figures and formal statistical analyses:
  - Nominal visits collected on the eCRF will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in Pharmacokinetic listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.
  - Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings but omitted from figures, summaries and statistical analyses.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables.
- Unscheduled visits will not be included in figures.
- All unscheduled visits will be included in listings.

| All unscrieduled | All unscriedated visits will be included in listings. |
|---|---|
| Descriptive Summary Statistics | |
| Continuous Data Refer to IDSL Statistical Principle 6.06.1 | |
| Categorical Data | N, n, frequency, % |
| Reporting of Pharm | Reporting of Pharmacokinetic Concentration Data |
| Descriptive | Refer to IDSL Statistical Principle 6.06.1 |
| Summary Statistics | Assign zero to NQ values (Refer to GUI_51487 for further details) |

206898

| Reporting Standard | s |
|---|---|
| Reporting of Pharmacokinetic Parameters | |
| Reporting for PK tables, figures and listings: | |
| <ul> <li>Planned time relative to dosing will be used in mean concentration-time figures and<br/>summaries, and actual times will be used for individual concentration-time figures.</li> </ul> | |
| <ul> <li>The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate</li> <li>Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in all PK figures, summaries and listings.</li> </ul> | |
| Descriptive<br>Summary Statistics<br>(Log Transformed) | N, n, geometric mean, 95% CI of geometric mean, standard deviation (SD) of logged data and [between and or within] geometric coefficient of variation (CV <sub>b</sub> (%)) will be reported. $ \text{CV}_b \text{ (%)} = \sqrt{\left(\text{exp}(\text{SD}^2) - 1\right) * 100} $ (SD = SD of log transformed data) |
| Parameters Not<br>Being Log<br>Transformed | tmax, first point, last point, and number of points used in the determination of $\lambda z$ . |
| Summary Tables | The following PK parameters will not be summarised: first point, last point, and number of points used in the determination of $\lambda z$ |
| Listings | Additionally, include the first point, last point and number of points used in the determination of lambda_z for listings. |
| <b>Graphical Displays</b> | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |
206898

# 10.6. Appendix 6: Derived and Transformed Data

### 10.6.1. General

### **Multiple Measurements at One Time Point**

- If there are two values within a time window the value closest to the target day for that window will be used. If values are the same distance from the target then the mean will be taken.
- Subjects having both High and Low values for Normal Ranges at any post-baseline visits for safety parameters will be counted in both the High and Low categories of "Any visit postbaseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

### **Study Day**

- Calculated as the number of days from Day 1 Visit:
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < Date of Day 1 Visit → Study Day = Ref Date -Date of Day 1 Visit</li>
  - Ref Date ≥ Date of Day 1 Visit → Study Day = Ref Date –Date of Day 1 Visit + 1

### 10.6.2. Study Population

### **Demographics**

#### Age

- As the month and date of birth will not be collected in the study, the age will be calculated as Year of ICF – Year of Birth;
- Birth date will be presented in listings as 'YYYY'.

#### **Body Mass Index (BMI)**

Calculated as Weight (kg) / [Height (m)<sup>2</sup>]

#### **Extent of Exposure**

- Duration of exposure to study drug will be calculated based on the formula:
  - The duration of exposure for oral phase is defined as the number of days starting from the first oral dose to the last oral dose.
  - Duration of exposure for injection phase is defined as the number of injections (1, 2, 3, 4 or 5)
  - Overall exposure to CAB is defined as number of days from the first oral dose to 8 weeks
    following the participant's last injection. If a participant does not enter the injection phase,
    the overall CAB exposure for the study will be defined as the number of days from the first
    oral dose to the last oral dose.
  - Overall exposure to the study (for safety evaluation) is defined as number of days from the first dose to last visit (including unscheduled visit) in days.
- The cumulative dose will be based on the formula:
  - Cumulative dose in oral phase is defined as (number of tablets dispensed number of tablets returned) \* 30 mg
  - Cumulative dose in injection phase is defined as number of injections \* 600 mg

206898

### 10.6.3. Safety

### **Adverse Events**

### **Adverse Events of Special Interest**

- Diarrhea
- Hypertriglyceridemia/ Hypercholesterolemia
- Decline in Renal Function
- Proximal Renal Tubule Dysfunctions
- Proteinuria

### **Laboratory Parameters**

- HIV-1 RNA: For summaries and analyses which use HIV-1 RNA level as a continuous measure, the logarithm to base 10 of the value will be used.
- If a laboratory value which is expected to have a numeric value for summary purposes, has a non-detectable level reported in the database, where the numeric value is missing, but typically a character value starting with '<x' or '>x' (or indicated as less than x or greater than x in the comment field) is present, the number of significant digits in the observed values will be used to determine how much to add or subtract in order to impute the corresponding numeric value.
  - Example 1: 2 Significant Digits = '< x' becomes x 0.01</li>
  - Example 2: 1 Significant Digit = '> x' becomes x + 0.1
  - Example 3: 0 Significant Digits = '< x' becomes x 1

206898

# 10.7. Appendix 7: Premature Withdrawals & Handling of Missing Data

## 10.7.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | Subject study completion (i.e. as specified in the protocol) was defined as completing all phases of the study including week 89. |
| | <ul> <li>If participants prematurely discontinue the oral phase of the study, additional<br/>replacement participants may be recruited at the discretion of the Sponsor.<br/>Participants who enter the injection phase of the study will not be replaced</li> </ul> |
| | <ul> <li>All available data from subjects who were withdrawn from the study will be listed<br/>and all available planned data will be included in summary tables and figures,<br/>unless otherwise specified.</li> </ul> |

# 10.7.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument: These data will be indicated using a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table. |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to<br/>be missing data and should be displayed as such.</li> </ul> |
| | Missing endpoints which are not covered in the following rule will not be imputed, unless otherwise specified. |
| Outliers | Any subjects excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

# 10.7.2.1. Handling of Missing Dates

| Reporting Detail |
|---|
| Partial dates will be displayed as captured in subject listing displays. |
| <ul> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> <li>Partial missing start or end dates will be imputed using the convention specified in Section 10.7.2.2 Handling of Partial Dates</li> </ul> |

206898

# 10.7.2.2. Handling of Partial Dates

| Element | Reporting Detail |
|---|---|
| Concomitant<br>Medications | <ul> <li>Partial dates for any concomitant medications recorded in the CRF will be imputed using the following convention: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |
| Adverse<br>Events | <ul> <li>Any partial dates for adverse events will be raised to data management. If the full date cannot be ascertained, the following assumptions will be made: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month.</li> <li>However, if these results in a date prior to Week 1 Day 1 and the event could possibly have occurred during treatment from the partial information, then the Week 1 Day 1 date will be assumed to be the start date. The AE will then be considered to start on-treatment (worst case).</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

# 10.7.2.3. Handling of Missing Data for Statistical Analysis

| Element | Reporting Detail |
|---------|-----------------------------------------------------------------|
| N/A | No statistical analysis is planned, unless otherwise specified. |

206898

# 10.8. Appendix 8: Values of Potential Clinical Importance

# 10.8.1. Laboratory Values

| Haematology | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| | | Male | | 0.54 |
| Hematocrit | Ratio of 1 | Female | | 0.54 |
| | | $\Delta$ from BL | ↓0.075 | |
| | // | Male | | 180 |
| Hemoglobin | g/L | Female | | 180 |
| | | $\Delta$ from BL | ↓25 | |
| Lymphocytes | x10 <sup>9</sup> / L | | 8.0 | |
| Neutrophil Count | x109/ L | | 1.5 | |
| Platelet Count | x109/ L | | 100 | 550 |
| While Blood Cell Count (WBC) | x109/ L | | 3 | 20 |

| Clinical Chemistry | | | | |
|---|---|---|---|---|
| Laboratory Parameter | Units | Category | Clinical Concern Range | |
| | | | Low Flag (< x) | High Flag (>x) |
| Albumin | g/L | | 30 | |
| Calcium | mmol/L | | 2 | 2.75 |
| Creatinine | umol/L | $\Delta$ from BL | | <b>↑ 44.2</b> |
| Glucose | mmol/L | | 3 | 9 |
| Phosphorus | mmol/L | | 0.8 | 1.6 |
| Potassium | mmol/L | | 3 | 5.5 |
| Sodium | mmol/L | | 130 | 150 |
| Total CO2 | mmol/L | | 18 | 32 |

| Liver Function | | | |
|--------------------|--------|----------|------------------------|
| Test Analyte | Units | Category | Clinical Concern Range |
| ALT/SGPT | U/L | High | ≥ 2x ULN |
| AST/SGOT | U/L | High | ≥ 2x ULN |
| AlkPhos | U/L | High | ≥ 2x ULN |
| T Bilirubin | μmol/L | High | ≥ 1.5xULN |
| | μmol/L | | 1.5xULN T. Bilirubin |
| T. Bilirubin + ALT | | High | + |
| | U/L | | ≥ 2x ULN ALT |

206898

### 10.8.2. ECG

| ECG Parameter | Units | Clinical Cor | cern Range |
|----------------------------|-------|--------------|----------------------|
| | | Lower | Upper |
| Absolute | | | |
| | | > 450 [1] | |
| Abaalista OTa Intanial | | > 450 [1] | ≤ 479 <sup>[1]</sup> |
| Absolute QTc Interval | msec | ≥ 480 [1] | ≤ 499 <sup>[1]</sup> |
| | | ≥ 500 [1] | |
| Absolute PR Interval | msec | < 110 [1] | > 220 [1] |
| Absolute QRS Interval | msec | < 75 [1] | > 110 [1] |
| Change from Baseline | | | |
| | msec | > 60 [1] | |
| Increase from Baseline QTc | msec | > 30 [1] | ≤ 59 <sup>[1]</sup> |
| | msec | ≥ 60 [1] | |

**NOTES:** [Remove footnotes for RAP development]

- 1. Represent standard ECG values of PCI for HV studies
- 2. Represent further subdivisions of ECG values for analysis whereby the RAP team needs to decide whether these need to be generated in addition to standard ECG values being flagged. IF not required, then delete.

### 10.8.3. Vital Signs

| Vital Sign Parameter | Units | Clinical Concern Range | |
|--------------------------|-------|------------------------|-------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |

| Vital Sign Parameter | Units | Clinical Concern Range | | | |
|---|---|---|---|---|---|
| (Change from Baseline) | | Decrease | | Increase | |
| | | Lower | Upper | Lower | Upper |
| Systolic Blood Pressure | mmHg | ≥ 20 | ≥ 40 | ≥ 20 | ≥ 40 |
| Diastolic Blood Pressure | mmHg | ≥ 10 | ≥ 20 | ≥ 10 | ≥ 20 |
| Heart Rate | bpm | ≥ 15 | ≥ 30 | ≥ 15 | ≥ 30 |

**NOTES:** [Remove footnotes for RAP development]

Represent further subdivisions of BP & HR for analysis whereby the RAP team needs to decide whether these need to be generated in addition to standard absolute BP & HR values being flagged. IF not required, then delete.

206898

# 10.9. Appendix 9: Multicenter Studies

# 10.9.1. Methods for Handling Centres

• In this multicentre study, enrolment will be presented by investigative site.

206898

# 10.10. Appendix 10: Examination of Covariates, Subgroups & Other Strata

## 10.10.1. Handling of Covariates, Subgroups & Other Strata

- Demographic covariates that may be used in descriptive summaries and statistical analyses, some of which may also be used for subgroup analyses.
- Additional covariates of clinical interest may also be considered.

206898

# 10.11. Appendix 11: Multiple Comparisons & Multiplicity

# 10.11.1. Handling of Multiple Comparisons & Multiplicity

Not applicable.

206898

# 10.12. Appendix 12: Model Checking and Diagnostics for Statistical Analyses

## 10.12.1. Statistical Analysis Assumptions

| Endpoint(s) | • | PK endpoint $C_{\tau}$ |
|-------------|---|------------------------|
| Analysis | • | ANOVA (primary) |

- Model assumptions will be applied, but appropriate adjustments maybe made based on the data
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.

206898

# 10.13. Appendix 13 – Abbreviations & Trade Marks

# 10.13.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AUC(0-τ) | Area under the concentration-time curve (AUC) over the dosing interval |
| Сτ | The observed concentration at the end of the dosing interval |
| CAB | Cabotegravir |
| CAB LA | Cabotegravir Long Acting |
| CDISC | Clinical Data Interchange Standards Consortium |
| CI | Confidence Interval |
| CL/F | The apparent clearance (adjusted for bioavailability, F) |
| Cmax | Maximum observed concentration |
| CSR | Clinical Study Report |
| CTMS | Clinical Trial Management System |
| $CV_b$ | Coefficient of Variation (Between) |
| DOB | Date of Birth |
| DP | Decimal Places |
| eCRF | Electronic Case Record Form |
| GSK | GlaxoSmithKline |
| HIV | Human Immunodeficiency Virus |
| ICH | International Conference on Harmonisation |
| IDSL | Integrated Data Standards Library |
| IM | Intramuscular |
| IP | Investigational Product |
| MedDRA | Medical Dictionary for Regulatory Activities |
| mg | Milligrams |
| PCI | Potential Clinical Importance |
| PK | Pharmacokinetic |
| PrEP | Pre-exposure prophylaxis |
| QC | Quality Control |
| RAP | Reporting & Analysis Plan |
| SAC | Statistical Analysis Complete |
| SAS | Statistical Analysis Software |
| SD | Standard deviation |
| SDTM | Study Data Tabulation Model |
| SOP | Standard Operation Procedure |
| t½ | Terminal phase half-life |
| tmax | Time to first occurrence of Cmax |
| TFL | Tables, Figures & Listings |
| Vz/F | The volume of distribution associated with the terminal phase (adjusted |
| | for bioavailability, F) |
| λz | Terminal-phase rate constant |

206898

### 10.13.2. Trademarks

Trademarks of the GlaxoSmithKline Group of Companies

NONE

Trademarks not owned by the GlaxoSmithKline Group of Companies

SAS

Phoenix WinNonlin

206898

# 10.14. Appendix 14: List of Data Displays

### 10.14.1. Data Display Numbering

The following numbering will be applied for RAP generated display according to ICH standards:

| Section | Tables | Figures |
|------------------|-------------|---------|
| Study Population | 1.1 to 1.10 | NA |
| Safety | 2.1 to 2.32 | NA |
| Pharmacokinetic | 3.1 to 3.11 | 3.1-3.8 |
| Section | Listings | |
| ICH Listings | 1-51 | |

## 10.14.2. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated and if required an example mock-up displays provided in Appendix 15: Example Mock Shells for Data Displays.

| Section | Figure | Table | Listing |
|------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |

#### NOTES:

Non-Standard displays are indicated in the 'IDSL / TST ID / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

### 10.14.3. Deliverable [Priority]

| Delivery [Priority] [1] | Description |
|-------------------------|--------------------------------------------------|
| W41 SAC [1] | Primary Statistical Analysis Complete at Week 41 |
| SAC [1] | Final Statistical Analysis Complete at Week 89 |

### NOTES:

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort.

206898

# 10.14.4. Study Population Tables

| Study Pop | oulation Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| Study Po | pulation, Dispos | ition and Demographic | es | | |
| 1.1 | Screened | SP1 | Summary of Study Population | | W41 SAC [1],<br>SAC [1] |
| 1.2 | Screened | ES6 | Summary of Screen Status and Reasons for Screen Failures | | W41 SAC [1],<br>SAC [1] |
| 1.3 | Screened | ES1 | Summary of Subject Disposition for the Subject Conclusion Record | | W41 SAC [1], SAC [1] |
| 1.4 | Safety | SD1 | Summary of Treatment Status and Reasons for Discontinuation of Study Treatment | | W41 SAC [1], SAC [1] |
| 1.5 | Safety | DM1 | Summary of Demographic Characteristics | | W41 SAC [1], SAC [1] |
| Medical H | History and Cond | omitant Medications | | | |
| 1.6 | Safety | MH4 | Summary of Medical Conditions | | W41 SAC [1], SAC [1] |
| 1.7 | Safety | CM1 | Summary of Prior Medications | | W41 SAC [1], SAC [1] |
| 1.8 | Safety | CM1 | Summary of Concomitant Medications | | W41 SAC [1], SAC [1] |
| Protocol | Deviations | | | | |
| 1.9 | Safety | IE1 | Summary of Inclusion/Exclusion Criteria Deviations | | W41 SAC [1], SAC [1] |
| 1.10 | Safety | DV1A | Summary of Important Protocol Deviations | | W41 SAC [1], SAC [1] |

206898

# 10.14.5. Safety Tables

| | | | Safety: Tables | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| Exposure | | | | | |
| 2.1 | Safety | EX1 | Summary of Extent of Exposure | | W41 SAC [1],<br>SAC [1] |
| Injection S | Site Reactions | | | | |
| 2.2 | Safety<br>Injection | | Summary of Injection Site Reaction | | W41 SAC [1],<br>SAC [1] |
| Adverse E | vents | | | | |
| 2.3 | Safety | AE1 | Summary of All Adverse Events by System Organ Class and Preferred Term | | W41 SAC [1], SAC [1] |
| 2.4 | Safety | AE5B | Summary of All Adverse Events by Maximum Grade by<br>System Organ Class and Preferred Term | | W41 SAC [1], SAC [1] |
| 2.5 | Safety | AE3 | Summary of All Grade 2 or Higher Adverse Events by<br>Overall Frequency | | W41 SAC [1], SAC [1] |
| 2.6 | Safety | AE3 | Summary of Serious Adverse Events | | W41 SAC [1], SAC [1] |
| 2.7 | Safety | AE16 | Summary of Serious Adverse Events by System Organ<br>Class and Preferred Term (Number of Subjects and<br>Occurrences) | | W41 SAC [1], SAC [1] |
| 2.8 | Safety | AE3 | Summary of Adverse Events Leading to Permanent Discontinuation of Study Drug or Withdrawal from Study | | W41 SAC [1], SAC [1] |
| 2.9 | Safety | AE1 | Summary of Drug-Related Adverse Events | | W41 SAC [1], SAC [1] |
| 2.10 | Safety | AE1 | Summary of Drug-Related Serious Adverse Events | | W41 SAC [1], SAC [1] |

| | | | Safety: Tables | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| 2.11 | Safety | AE3 | Summary of Drug-related Grade 2 or Higher Adverse<br>Events by Overall Frequency | | W41 SAC [1], SAC [1] |
| 2.12 | Safety | AE3 | Summary of Common (>=5%) Adverse Events by Overall Frequency | | W41 SAC [1], SAC [1] |
| 2.13 | Safety | AE15 | Summary of Common (>=5%) Non-Serious Adverse<br>Events by System Organ Class and Preferred Term<br>(Number of Subjects and Occurrences) | | W41 SAC [1], SAC [1] |
| 2.14 | Safety | AE3 | Summary of Common (>=5%) Grade 2-4 Adverse Events by Overall Frequency | | W41 SAC [1], SAC [1] |
| 2.15 | Safety | AE3 | Summary of Common (>=5%) Drug-Related Grade 2-4<br>Adverse Events by Overall Frequency | | W41 SAC [1], SAC [1] |
| Laboratory | Tests | | | | |
| 2.16 | Safety | | Summary of Grade 2 or Higher Laboratory Tests | | W41 SAC [1], SAC [1] |
| 2.17 | Safety | ES11 | Summary of Characteristics of Adverse Events of Special Interest | | W41 SAC [1], SAC [1] |
| 2.18 | Safety | LB1 | Summary of Change from Baseline in Hematology and Coagulation Data | | W41 SAC [1], SAC [1] |
| 2.19 | Safety | LB1 | Summary of Change from Baseline in Fasting Chemistry Data and Lipid Profile | | W41 SAC [1], SAC [1] |
| 2.20 | Safety | UR3 | Summary of Urinalysis and Urine Chemistry Results | | W41 SAC [1], SAC [1] |
| 2.21 | Safety | LB18 | Summary of Hematology and Coagulation Grade Shifts from Baseline Grade | | W41 SAC [1], SAC [1] |
| 2.22 | Safety | LB18 | Summary of Fasting Chemistry and Lipid Profile Grade Shifts from Baseline Grade | | W41 SAC [1], SAC [1] |

| | | | Safety: Tables | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable [Priority] |
| 2.23 | Safety | LB18 | Summary of Urinalysis Grade Shifts from Baseline Grade | | W41 SAC [1], SAC [1] |
| Vital Signs | | | | | |
| 2.24 | Safety | VS1 | Summary of Change from Baseline in Vital Signs | | W41 SAC [1], SAC [1] |
| 2.25 | Safety | VS8 | Summary of Vital Sign Shifts from Baseline with Respect to Clinical Concern Range | | W41 SAC [1], SAC [1] |
| Liver Event | S | | | | |
| 2.26 | Safety | LIVER1 | Summary of Liver Events Reporting | | W41 SAC [1], SAC [1] |
| 2.27 | Safety | LIVER10 | Summary of Hepatobiliary Laboratory Abnormalities | | W41 SAC [1], SAC [1] |

206898

# 10.14.6. Tolerability Tables

| | | | Tolerability: Tables | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Tolerability | Tolerability of CAB Injection | | | | |
| 2.28 | Safety<br>Injection | | Summary of HIV-Prevention Treatment Satisfaction Scores | | W41 SAC [1],<br>SAC [1] |

206898

# 10.14.7. Acceptability Tables

| | Acceptability: Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| | Acceptability of the CAB Injection | | | | |
| 2.29 | Safety | | Summary of Acceptability of the CAB LA | | W41 SAC [1],<br>SAC [1] |

206898

## 10.14.8. Pharmacokinetic Tables

| Pharma | Pharmacokinetic : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Oral Ph | ase | | | | |
| 3.1 | Oral PK | PKCT1 | Summary of CAB Plasma Pharmacokinetic Concentration-<br>Time Data – Oral Phase | | SAC [1] |
| 3.2 | Oral PK | PKPT4 | Summary of Derived CAB Plasma Pharmacokinetic Parameters (Non-Transformed) – Oral Phase | Parameters with units | SAC [1] |
| 3.3 | Oral PK | PKPT4 | Summary of Derived CAB Plasma Pharmacokinetic Parameters (Log-Transformed) – Oral Phase | Parameters with units | SAC [1] |
| Injection | n Phase (up to Week | 41) | | | |
| 3.4 | Injection<br>(Week 41) PK | PKCT1 | Summary of CAB Plasma Pharmacokinetic Concentration-<br>Time Data – Injection Phase (up to Week 41) | | W41 SAC [1],<br>SAC [1] |
| 3.5 | Injection<br>(Week 41) PK | PKPT4 | Summary of Derived CAB Plasma Pharmacokinetic<br>Parameters (Non-Transformed) – Injection Phase (up to<br>Week 41) | Parameters with units | W41 SAC [1],<br>SAC [1] |
| 3.6 | Injection<br>(Week 41) PK | PKPT4 | Summary of Derived CAB Plasma Pharmacokinetic<br>Parameters (Log-Transformed) – Injection Phase (up to<br>Week 41) | Parameters with units | W41 SAC [1]<br>SAC [1] |
| 3.7 | Injection<br>(Week 41) PK | PKPT3 | Statistical Analysis of CAB Plasma Accumulation – Injection Phase (up to Week 41) | Cτ only for Injection<br>Phase at Week 41. | W41 SAC [1],<br>SAC [1] |
| 3.8 | Injection<br>(Week 41) PK | PKPT3 | Statistical Analysis of CAB Plasma Steady-state Pre-dose Concentrations – Injection Phase (up to Week 41) | Cτ only for Injection<br>Phase at Week 41. | W41 SAC [1],<br>SAC [1] |

| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
|---|---|---|---|---|---|
| Injection | n Phase (up to Week | 89) | | | |
| 3.9 | Injection<br>(Week 89) PK | PKCT1 | Summary of CAB Plasma Pharmacokinetic Concentration-<br>Time Data – Injection Phase (up to Week 89) | | SAC [1] |
| 3.10 | Injection<br>(Week 89) PK | PKPT4 | Summary of Derived CAB Plasma Pharmacokinetic<br>Parameters (Non-Transformed) – Injection Phase (up to<br>Week 89) | Parameters with units | SAC [1] |
| 3.11 | Injection<br>(Week 89) PK | PKPT4 | Summary of Derived CAB Plasma Pharmacokinetic<br>Parameters (Log-Transformed) – Injection Phase (up to<br>Week 89) | Parameters with units | SAC [1] |

206898

# 10.14.9. Pharmacokinetic Figures

| Pharm | Pharmacokinetic : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming<br>Notes | Deliverable<br>[Priority] |
| Oral Pl | Oral Phase | | | | |
| 3.1 | Oral PK | PKCF1P | Individual CAB Plasma Concentration-Time Plots (Linear and Semi-Logarithmic) – Oral Phase | | SAC [1] |
| 3.2 | Oral PK | PKCF4 | Mean (±SD) CAB Plasma Concentration-Time Plots (Linear and Semi-Logarithmic) – Oral Phase | | SAC [1] |
| Injection | on Phase (up to Wee | k 41) | | | |
| 3.3 | Injection<br>(Week 41) PK | PKCF1P | Individual CAB Plasma Concentration-Time Plots (Linear and Semi-Logarithmic) – Injection Phase (up to Week 41) | | W41 SAC [1],<br>SAC [1] |
| 3.4 | Injection<br>(Week 41) PK | PKCF4 | Mean (±SD) CAB Plasma Concentration-Time Plots (Linear and Semi-Logarithmic) – Injection Phase (up to Week 41) | | W41 SAC [1],<br>SAC [1] |
| 3.5 | Injection<br>(Week 41) PK | PK26 | Individual CAB Plasma Pre-dose Concentration versus Week (Linear and Semi-Logarithmic) – Injection Phase (up to Week 41) | | W41 SAC [1],<br>SAC [1] |
| 3.6 | Injection<br>(Week 41) PK | PK27 | Median (range) CAB Plasma Pre-dose Concentration versus Week (Linear and Semi log) – Injection Phase (up to Week 41) | | W41 SAC [1],<br>SAC [1] |
| Injection | Injection Phase (up to Week 89) | | | | |
| 3.7 | Injection<br>(Week 89) PK | PKCF1P | Individual CAB Plasma Concentration-Time Plots (Linear and Semi-Logarithmic) – Injection Phase (up to Week 89) | | SAC [1] |
| 3.8 | Injection<br>(Week 89) PK | PKCF4 | Mean (±SD) CAB Plasma Concentration-Time Plots (Linear and Semi-Logarithmic) – Injection Phase (up to Week 89) | | SAC [1] |

206898

# 10.14.10. ICH Listings

| ICH: Listi | ngs | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Study Po | opulation, Dispositi | on and Demogra | phics | | <u> </u> |
| 1 | Screened | SP3 | Listing of Subjects Excluded from Any Population | | W41 SAC [1], SAC [1] |
| 2 | Screened | ES7 | Listing of Reasons for Screen Failure | | W41 SAC [1], SAC [1] |
| 3 | Safety | ES2 | Listing of Reasons for Withdrawal | | W41 SAC [1], SAC [1] |
| 4 | Safety | SD2 | Listing of Study Drug Discontinuation Record | | W41 SAC [1], SAC [1] |
| 5 | Safety | DM2 | Listing of Demographic Characteristics | | W41 SAC [1], SAC [1] |
| 6 | Safety | EX3 | Listing of Exposure Data – Oral Dose | | W41 SAC [1], SAC [1] |
| 7 | Safety | | Listing of Exposure Data – Injection | | W41 SAC [1], SAC [1] |
| Medical | History and Conco | mitant Medication | on | | |
| 8 | Safety | MH2 | Listing of Medical Conditions | | W41 SAC [1], SAC [1] |
| 9 | Safety | CM5 | Listing of Prior Medications | | W41 SAC [1], SAC [1] |
| 10 | Safety | CM5 | Listing of Concomitant Medications | | W41 SAC [1], SAC [1] |

| ICH: List | ings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Protoco | l Deviations | | | | · |
| 11 | Safety | IE3 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | W41 SAC [1], SAC [1] |
| 12 | Safety | DV2 | Listing of Important Protocol Deviations | | W41 SAC [1], SAC [1] |
| Injection | Site Reaction | | | | |
| 13 | Safety Injection | | Listing of Injection Site Reaction –<br>Daily Diary Card 1 | | W41 SAC [1],<br>SAC [1] |
| 14 | Safety Injection | | Listing of Injection Site Reaction –<br>Daily Diary Card 2 | | W41 SAC [1],<br>SAC [1] |
| Adverse | Events | | | | <u> </u> |
| 15 | Safety | AE7 | Listing of Subject Numbers for Individual Adverse Events | | W41 SAC [1],<br>SAC [1] |
| 16 | Safety | AE8 | Listing of All Adverse Events | | W41 SAC [1], SAC [1] |
| 17 | Safety | AE8CPA | Listing of Serious Adverse Events (Fatal and Non-Fatal) | | W41 SAC [1], SAC [1] |
| 18 | Safety | AE8 | Listing of Grader 2 or Higher Adverse Events | | W41 SAC [1], SAC [1] |
| 19 | Safety | AE8 | Listing of All Adverse Events Leading to Premature Discontinuation of Study Drug or Withdrawal from Study | | W41 SAC [1], SAC [1] |
| 20 | Safety | AE8 | Listing of Adverse Events of Special Interest | | W41 SAC [1], SAC [1] |

| ICH: List | ings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| 21 | Safety | | Listing of Possible Suicidality-Rated Adverse Events | | W41 SAC [1], SAC [1] |
| 22 | Safety | AE2 | Listing of Relationship Between<br>System Organ Classes and Verbatim<br>Text | | W41 SAC [1], SAC [1] |
| 23 | Safety | AE14 | Listing of Reasons for Considering as a Serious Adverse Event | | W41 SAC [1], SAC [1] |
| Deaths | <u> </u> | | | | |
| 24 | Safety | | Listing of Death | | W41 SAC [1], SAC [1] |
| Laborato | ory Tests | | | | <u> </u> |
| 25 | Safety | LB5 | Listing of Chemistry Data and Fasting Lipid Profile | | W41 SAC [1], SAC [1] |
| 26 | Safety | LB5 | Listing of Hematology and Coagulation Data | | W41 SAC [1], SAC [1] |
| 27 | Safety | UR2a | Listing of Urinalysis and Urine<br>Chemistry Data | | W41 SAC [1], SAC [1] |
| 28 | Safety | LB5 | Listing of Laboratory Data for Subjects with Grade 2 or Higher Abnormalities | | W41 SAC [1], SAC [1] |
| 29 | Safety | LB14 | Listing of HIV Tests | | W41 SAC [1], SAC [1] |
| 30 | Safety | LB5 | Listing of Local Lab Data | | W41 SAC [1], SAC [1] |

| ICH: Listings | CH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Vital Sign | rital Sign | | | | |
| 31 | Safety | VS4 | Listing of Vital Signs | | W41 SAC [1], SAC [1] |
| 32 | Safety | VS4 | Listing of Vital Signs for Subjects with<br>Any Value of Potential Clinical<br>Importance | | W41 SAC [1], SAC [1] |
| ECG's | | | | | |
| 33 | Safety | | Listing of ECG Results | | W41 SAC [1], SAC [1] |
| Social Harm | | | | | |
| 34 | Safety | | Listing of Social Harm | | W41 SAC [1], SAC [1] |
| Cardiovascul | ar Event | | | | |
| 35 | Safety | | Listing of Cardiovascular Event | | W41 SAC [1], SAC [1] |
| Liver Event | | | | | |
| 36 | Safety | | Listing of Liver Event | | W41 SAC [1], SAC [1] |
| Tolerability o | Tolerability of CAB Injection | | | | |
| 37 | Safety Injection | | Listing of HIV-Prevention Treatment Satisfaction Questionnaire | | W41 SAC [1], SAC [1] |

| ICH: Listi | ICH: Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST<br>ID / Example<br>Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Acceptab | oility of the CAB Inject | ion | | | |
| 38 | Safety | | Listing of Acceptability of the CAB LA | | W41 SAC [1],<br>SAC [1] |
| Pharmac | okinetic | | | | |
| 39 | Oral PK | PKCL1P | Listing of CAB Plasma Pharmacokinetic Concentration-Time Data – Oral Phase | Please list all the concentration data including unscheduled. | SAC [1] |
| 40 | Oral PK | PKPL1P | Listing of Derived CAB Plasma Pharmacokinetic Parameters – Oral Phase | | SAC [1] |
| 41 | Injection<br>(Week 41) PK | PKCL1P | Listing of CAB Plasma Pharmacokinetic Concentration-Time Data – Injection Phase (up to Week 41) | Please list all the concentration data including unscheduled. | W41 SAC [1],<br>SAC [1] |
| 42 | Injection<br>(Week 41) PK | PKPL1P | Listing of Derived CAB Plasma<br>Pharmacokinetic Parameters –<br>Injection Phase (up to Week 41) | | W41 SAC [1],<br>SAC [1] |
| 43 | Injection<br>(Week 89) PK | PKCL1P | Listing of CAB Plasma Pharmacokinetic Concentration-Time Data – Injection Phase (up to Week 89) | Please list all the concentration data including unscheduled. | SAC [1] |
| 44 | Injection<br>(Week 89) PK | PKPL1P | Listing of Derived CAB Plasma<br>Pharmacokinetic Parameters –<br>Injection Phase (up to Week 89) | | SAC [1] |

206898

# 10.14.11. Non-ICH Listings

| Non-ICH: Listings | |
|-------------------|---------------------------|
| | Deliverable<br>[Priority] |

206898

# 10.15. Appendix 15: Example Mock Shells for Data Displays

Data Display Specification will be made available on Request